

Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## **SPONSOR:**

# **BioMed Valley Discoveries**

## PROTOCOL NUMBER:

BVD-523-HCQ

# STATISTICAL ANALYSIS PLAN

| Author: | Julien Lucas |
|----------|--------------|
| Version: | 2.0 |
| Date: | 02-Sep-2024 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 1 Cover and signature pages

| Sponsor: | BioMed Valley Discoveries |
|---|---|
| Protocol Number: | BVD-523-HCQ |
| Study Title: | A phase 2 basket trial of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring MAPK pathway mutations (BVD-523-HCQ) |
| Document Version No | 1.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorise its approval.

#### Statistician

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|---|---|---|---|
| | Biostat III | | Signed by: Julium (Mas Signer Name: Julien Lucas Signing Reason: I approve this document Signing Time: 09-Sep-2024 11:19 BST 1805EF259FF0471980A64D0037F8D5D3 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## **Client Representative**

| Title Name [text box when using eSignatures]: | | Date | Signature |
|---|---|---|---|
| | Senior Scientist | | Signed by: Chank Chance Signer Name: Anna Groover Signing Reason: I approve this document Signing Time: 03-Sep-2024 08:40 CDT 71380BDD08BC4D289E63FA3831CD4243 |
| | President | | Signed by: Brent Kreides Signer Name: Brent Kreider Signing Reason: I approve this document Signing Time: 04-Sep-2024 08:58 PDT 9FC8BD6421864A9788CCD264914F8A6C |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 2 Table of Contents

| 1 | | Cove | er and signature pages | 2 |
|---|---|---|---|---|
| 2 | | Tabl | e of Contents | 4 |
| 3 | | List ( | of Abbreviations | 6 |
| 4 | | Intro | oduction | 8 |
| 5 | | Stud | ly Objectives | 8 |
| 6 | | Stud | ly Design | 9 |
| | 6. | 1 | STUDY DESIGN AND POPULATION | 9 |
| | 6. | 2 | STUDY TREATMENTS AND ASSESSMENTS | 11 |
| | 6. | 3 | RANDOMIZATION AND BLINDING | 12 |
| | 6.4 | 4 | SAMPLE SIZE JUSTIFICATION | 12 |
| 7 | | Stati | istical Considerations | 13 |
| | 7. | 1 | STUDY TREATMENT | L3 |
| | 7. | 2 | PLANNING OF ANALYSES | |
| | 7. | 3 | STUDY AND ANALYSIS PERIODS | L <b>4</b> |
| | 7. | 4 | SOFTWARE | <u> 4</u> |
| | 7. | 5 | MISSING DATA HANDLING | <b>L</b> 4 |
| | 7. | 6 | PARTIAL DATE IMPUTATION | <u> 4</u> |
| | 7. | 7 | VISIT WINDOWING | ۱6 |
| | 7. | 8 | REPORTING GUIDELINES | 16 |
| 8 | | Anal | lysis Sets1 | ١9 |
| 9 | | Met | hods of Analyses and Presentations | |
| | 9. | 1 | PATIENT DISPOSITION | |
| | 9. | 2 | PROTOCOL DEVIATIONS AND/OR VIOLATIONS | 1 |
| | 9. | 3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 1 |
| | 9. | 4 | MEDICAL HISTORY AND CONCOMITANT DISEASES | |
| | 9. | 5 | PRIOR THERAPIES | 23 |
| | 9. | 6 | STUDY DRUG EXPOSURE AND/OR COMPLIANCE | |
| | 9. | 7 | PHARMACOKINETIC/ PHARMACODYNAMIC ENDPOINTS AND ANALYSES | |
| | | 9.7.1 | | |
| | | 9.7.2 | | |
| | 9. | 8 | EFFICACY DATA ENDPOINTS AND ANALYSES | |
| | | 9.8.1 | | |
| | | 9.8.2 | | |
| | | 9.8.3 | . , , | |
| | 9. | _ | SAFETY DATA ENDPOINTS AND ANALYSES | |
| | | 9.9.1 | · , | |
| | | 9.9.2 | | |
| | | 9.9.3 | | |
| 10 | | | rim Analyses | |
| 1: | 1 | Char | nges to Planned Analyses | 34 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| 12 | Doc | ument History | 35 |
|----|-----|-------------------------------------------|----|
| | | erences | |
| | | endices | |
| | | Schedule of events | |
| 14 | 4.2 | Schedule of Correlative Sample Collection | 40 |
| 14 | 1.3 | CTCAE v5.0 Grading for Laboratory Values | 41 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 3 List of Abbreviations

AE Adverse Event

ATC Anatomical Therapeutic Chemical Classification

BOR Best Overall Response

BRAF V-raf murine sarcoma viral oncogene homolog B1

BVD BioMed Valley Discoveries

CI Confidence interval

CM Concomitant medications

CR Complete Response

CRA Clinical Research Associates

CRC Colorectal cancer

CRO Clinical Research Organization

DBP Diastolic blood pressure

DOR Duration of response

EAS Evaluable Analysis Set

EC Ethics Committee

eCRF Electronic Case Report Form

ERK Extracellular signal-regulated kinase

FAS Full Analysis Set

ICF Informed consent form

ICH International Conference on Harmonization

IRB Institutional Review Boards

IxRS Interactive Voice/Web Response System

MedDRA Medical Dictionary for Regulatory Activities

MEK Mitogen-activated protein kinase/extracellular signal-related kinase

mRNA Messenger ribonucleic acid

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

ORR Overall Response Rate

OS Overall survival
PD Pharmacodynamic

PDCF Protocol Deviation Criteria Form



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

PFS Progression Free Survival

PK Pharmacokinetic

PP Per-protocol analysis set

PR Partial Response
PT Preferred Term

SAE Serious adverse event
SAP Statistical analysis plan
SBP Systolic blood pressure

SMC Safety Monitoring Committee

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

TFLs Tables, listings and figures
WHO World Health Organization



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 4 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in the analysis of the Phase II study titled "A phase 2 basket trial of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring MAPK pathway mutations (BVD-523-HCQ)". This is an open-label, prospective phase two basket trial assessing the efficacy of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies. All patients enrolled must have a MAPK activating mutation to be deemed eligible for trial participation. Each disease-based basket will open to enrollment in two-stages. The opening of stage two will be dependent on the observed responses in the patients enrolled in the first stage.

This statistical analysis plan (SAP) covers the final analysis for the study. The list of tables, figures and listings (TFLs) to be developed for each analysis, as well as the shells for each TFL, are described in a separate document.

The preparation of this SAP is based on study Protocol version 2.0 from 02May2023, the most up to date electronic Case Report Form (eCRF) version and on the International Conference on Harmonization (ICH) E3 and E9 Guidelines.

## 5 Study Objectives

The primary, secondary, and exploratory objectives along with the associated endpoints as per the study protocol are presented as follows:

### Primary Objective

- To assess the safety and tolerability of ulixertinib and hydroxychloroquine in patients with advanced, RAS, non-V600 BRAF, MEK1/2, or ERK1/2 mutated gastrointestinal (GI) malignancies.
- To assess the efficacy of ulixertinib and hydroxychloroquine in patients with advanced, RAS, non-V600 BRAF, ERK1/2, or MEK1/2 mutated gastrointestinal malignancies.

#### Primary Endpoint

- The incidence and frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the national Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 5.0), seriousness, duration, and relationship to study treatment.
- Overall response rate as defined by the proportion of patients achieving a confirmed PR and CR (defined by RECIST 1.1) as evaluated by the local treating investigator.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

### Secondary Objective

 To assess the duration of efficacy of ulixertinib and hydroxychloroquine in patients with advanced RAS, non-V600 BRAF, MEK1/2 or ERK1/2 mutated gastrointestinal malignancies.

### Secondary Endpoint

 Progression-free survival (PFS) as defined as the time from study drug initiation to the time of documented disease progression (as assessed by RECIST 1.1) or death from any cause.

#### **Exploratory Objective**

 To evaluate the bioactivity of ulixertinib and hydroxychloroquine against ERK1/2, autophagy pathways, and pharmacodynamic biomarkers.

## **Exploratory Endpoint**

- Pharmacokinetics (PK) of ulixertinib and hydroxychloroguine.
- Blood and/or tissue samples used to assess biomarkers (RPPA, Nanostring, circulation tumor (ctDNA) examples of assays planned but not limited to only these).

## 6 Study Design

### 6.1 STUDY DESIGN AND POPULATION

This is an open-label, multicenter, phase II basket study of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring RAS, non-V600 BRAF, MEK1/2, or ERK1/2 mutations. The trial will have five baskets based on primary disease as listed below:

- Basket 1: Cholangiocarcinoma including intrahepatic cholangiocarcinoma, perihilar cholangiocarcinoma, or extrahepatic cholangiocarcinoma.
- Basket 2: Pancreatic adenocarcinoma.
- Basket 3: Colorectal adenocarcinoma.
- Basket 4: Esophageal adenocarcinoma, esophageal squamous cell carcinoma, or GEJ adenocarcinoma.
- Basket 5: Gastric adenocarcinoma.

To assess eligibility, cancer mutational status must be confirmed through patient medical records by treating physician. Once deemed eligible, ulixertinib and hydroxychloroquine will be orally administered twice daily on 28-day cycles. Safety will be assessed regularly through the



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

monitoring of adverse events, laboratory values, physical exams, vital signs, echocardiogram, eye exams, and ECGs. Disease assessments will be performed regularly as well to assess treatment efficacy. Upon disease progression, patients will be followed for safety for 60 days ± 7 days.

While the overall trial is a basket design, each basket will operate as a Simon two-stage design and therefore, will open to enrollment in two-stages.

An overview of the study design is presented in Figure 1 below.

Figure 1. Study Design



The first stage in each basket will open to enrollment and remain open until 13 patients are declared evaluable for response, at which time enrollment will be placed on hold for the evaluation of efficacy. To be evaluable for this Stage 1 efficacy analysis, a patient must have completed at least one cycle of therapy and must have at least 75% of the prescribed doses of ulixertinib and hydroxychloroquine during Cycle 1. Non-evaluable patients may remain on study therapy if deemed to be clinically benefiting by the treating Investigator.

The Stage 1 efficacy analysis will occur when all evaluable patients have had at least one post-treatment disease evaluation or have discontinued study therapy due to clinical progressive disease or drug-related adverse events. Patients who have discontinued study therapy due to clinical progressive disease or drug-related adverse events prior to the first efficacy evaluation will be considered non-responders. If a patient in the first 13 evaluable patients has an unconfirmed partial or complete response but has not yet had a confirmatory scan at the time



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

of the Stage 1 efficacy analysis, that patient may be counted as a responder for the purposes of the Stage 1 evaluation. If ≥ 4 of the first 13 evaluable patients in Stage 1 have a complete or partial response, with permission of the SMC the sponsor may open enrollment to Stage 2 for that basket. Stage 2 will expand enrollment of each basket until a total of 43 patients, including those enrolled during Stage 1, have been enrolled. Any patient deemed non-evaluable for the primary efficacy endpoint may be replaced.

An internal SMC will be charged with assuring risk/benefit balance for patients involved in the study. They will make study conduct recommendations based on emerging safety and efficacy data. Stage 2 of enrollment on each basket will not open until data review and approval from the SMC.

#### 6.2 STUDY TREATMENTS AND ASSESSMENTS

Ulixertinib and hydroxychloroquine will be administered twice-daily on a 28-day cycle starting with Cycle One Day One. Ulixertinib and hydroxychloroquine will be administered orally twice daily (every 12 hours ± 2 hours) together with food, at approximately the same time every day. Patients will be provided the study drug for a full cycle to self-administer at home.

Dose interruptions for study treatment-related AEs are allowed as per the dose modification recommendations (Table 1).

Table 1. Ulixertinib and Hydroxychloroquine Dose Levels

| Dose Level | Ulixertinib |
|---------------|--------------------|
| Dose Level 0 | 450 mg twice daily |
| Dose Level -1 | 300 mg twice daily |
| Dose Level -2 | 150 mg twice daily |

| Dose Level | Hydroxychloroquine |
|---------------|--------------------|
| Dose Level 0 | 600 mg twice daily |
| Dose Level -1 | 800 mg daily |

Doses of any investigational product that were not administered due to toxicity will not be replaced within the same cycle. In addition to dose interruption, the need for a dose reduction at the time of treatment resumption should also be considered based on the dose modifications recommendations. If toxicities require dose hold, both study drugs should be held and resumed concurrently. If a toxicity-related dose delay lasts for > 21 days, treatment will be discontinued permanently, and the patient should be removed from study treatment. If a patient requires a dose hold for > 21 days for a non-treatment related adverse event or situation (i.e. radiation therapy) the patient may continue on study only after approval and discussion with the Sponsor and Medical Monitor.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 6.3 RANDOMIZATION AND BLINDING

Not applicable.

#### 6.4 SAMPLE SIZE JUSTIFICATION

Under Simon's optimal two-stage design with a 5% significance level and 80% power, assuming a null hypothesis for ORR ≤ 20% versus the alternate hypothesis of ORR ≥ 40%, a total of 43 evaluable patients are required for the evaluation of the primary endpoint; 13 in Stage 1 and an additional 30 in Stage 2, for each basket.

In the first stage, if there are 3 or fewer patients achieving a response in the 13 patients, the study will be stopped for this basket. Otherwise, 30 additional patients will be accrued for a total of 43.

Then, if there are 12 or fewer responses in the 43 patients, the null hypothesis will not be rejected and any further investigation of the study medication in this basket will not be warranted. However, should at least 13 of the 43 evaluable patients achieve a response then the null hypothesis will be rejected, and it will be concluded that the study medication demonstrates activity for this basket to allow further investigation.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 7 Statistical Considerations

### 7.1 STUDY TREATMENT

The study drugs are ulixertinib (BVD-523) and hydroxychloroquine. The study treatment refers to treatment with ulixertinib (BVD-523) and hydroxychloroquine.

#### 7.2 PLANNING OF ANALYSES

This SAP covers the final analysis for the study. The planned timing of analysis for this study is after the last patient completes 8 cycles.

As per the Protocol a Safety Monitoring Committee (SMC) will occur for bi-annual or ad-hoc reviews as needed. The Tables, Figures and Listings (TFLs) planned in this SAP may also be used for SMC meetings as applicable. The TFLs shells table of contents will flag which outputs will be prepared for SMC purposes.

Given that the study was early terminated during Stage 1, an abbreviated CSR focusing on safety will be prepared. Therefore not all Tables, Listings and Figures planned in SAP version 1 will be required. The Shells table of contents will have an additional column to indicate which outputs will be delivered for the final analysis of Stage 1.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 7.3 STUDY AND ANALYSIS PERIODS

Study periods are summarized in <u>Table 1</u> below. Analysis periods will mirror these periods and are summarized in <u>Table 2</u> below.

**Table 1. Study periods** 

| Period | Visit | Planned days |
|---|---|---|
| SCREENING Screening (up to 4 weeks before Baseline) | | Day -28 to Day -1 |
| TREATMENT | Cycle 1 | Baseline |
| | | Day 8 ± 2 |
| | | Day 15 ± 2 |
| Cycle 2 | | Day 1 ± 2 |
| | | Day 15 ± 2 |
| | Cycle 3 – Cycle n | Day 1 ± 2 |
| POST TREATMENT | End of Treatment (EOT) Visit | +7 days after last dose |
| | Safety Follow-Up | 60 ± 7 days after last dose |
| Follow-Up | | Every 8 months (± 7 days) until death, disease progression or initiation of subsequent anticancer therapy. |

Table 2. Analysis periods

| Period | Definition |
|---|---|
| PRE-TREATMENT | From informed consent form (ICF) signature to the day before first dose of study treatment. |
| ON-TREATMENT | From the day of first dose of study treatment to 28 days after last dose of study treatment, or the earliest date of subsequent anti-cancer drug therapy – 1 day, whichever occurs first. |
| FOLLOW-UP | Follow-up period will be from the end of the on-treatment period until end of study. |

## 7.4 SOFTWARE

The SAS Viya version 3.5 or higher, will be used for all analysis, unless otherwise specified.

#### 7.5 MISSING DATA HANDLING

No imputation for missing data will be carried out other than to complete partial dates using standard imputation techniques as described below in <u>Section 7.6</u>.

## 7.6 PARTIAL DATE IMPUTATION

Detailed rules for partial date imputation are described below.

A permanent new date variable should be created if there is a requirement to be used in



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

determining flags (such as on-treatment flags), sort orders and other derived variables needed for a table, listing, or figure. Imputed date variable names will be defined in the derived dataset specifications.

Original (raw) date variables must not be overwritten. Imputed dates will not be displayed in the listings.

## General rules for Adverse events (AE) and prior and concomitant medications (CM)

In case of partial dates with missing day:

For AE and CM, any partial start date during the month of first dosing will be imputed to be the date of first dose, taking the worst-case scenario.

For any AE and CM starting after the month of first dosing, the start date will be imputed to be the first day of the month.

For any AE and CM starting before the month of first dosing, the start date will be imputed to be the last day of the month.

Partial AE and CM end dates will be imputed to be the last day of the month or at the date of study discontinuation/completion, whichever occurs first.

In case of partial dates with missing day and missing month:

For AE and CM, any partial start date during the year of first dosing will be imputed to be the date of first dose, taking the worst-case scenario.

For any AE and CM starting after the year of first dosing, the start date will be imputed to be the first day of the year (i.e. 01 January).

For any AE and CM started before the year of first dosing, the start date will be imputed to be the last day of the year (i.e. 31 December).

Partial AE and CM end dates will be imputed to be the last day of year (i.e. 31 December) or at the date of study discontinuation/completion, whichever occurs first.

Some examples are given below (DDMMMYYYY).

In most cases, start dates are imputed as first day of the month or first of January.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 3: Examples of missing dates imputation

| Data Type | Start<br>Date | Imputed<br>Start Date | First Dose<br>date | End Date | Imputed End<br>Date |
|---|---|---|---|---|---|
| Adverse Event, Prior/Concomitant Meds | JAN2017 | 31JAN2017 | 11NOV2017 | MAR2017 | 31MAR2017 |
| Adverse Event,<br>Prior/Concomitant Meds | MAR2017 | 01MAR2017 | 27JAN2017 | MAR2017 | 31MAR2017 |
| Adverse Event,<br>Prior/Concomitant Meds | 2017 | 27JAN2017 | 27JAN2017 | 2017 | 16MAR2017 <sup>£</sup> |
| Adverse Event,<br>Prior/Concomitant Meds | MAR2017 | 01MAR2017 | 27JAN2017 | MAR2017 | 01MAR2017* |
| Adverse Event,<br>Prior/Concomitant Meds | JAN2017 | 31JAN2017 | 27FEB2017 | 2017 | 31DEC2017 |

<sup>£</sup> Patient discontinued on 16MAR2017; \* Patient discontinued on 01MAR2017.

### Rules for other partial dates

Partial dates are not expected for death. However, should a partial date be present for death, the date will be imputed to be the day after the last visit/assessment date when the patient was known to be alive, if there is at least one visit/assessment during the month of the corresponding partial death date. If there is no visit/assessment performed during the month of the corresponding partial death date, then the partial death date would be imputed as the first day of the month. A similar approach will be followed for partial date for death in which only year is known.

If partial date is present for dates related to disease history, the same rules as for AE and CM will be applied.

## 7.7 VISIT WINDOWING

Planned assessments will not be re-assigned to any planned visits using statistical programming based on assessment date. All the data will be analysed according to the planned visit as collected in the eCRF. Data obtained at unscheduled and repeat assessments will be considered for the derivation of baseline, worst on-treatment result for safety analyses (clinical safety laboratory evaluation, other safety data), and time to event analyses.

#### 7.8 REPORTING GUIDELINES

#### Visit labels

The visit labels displayed in <u>Table 4</u> will be used to display results in the TFLs. Following Cycle 2, any subsequent Cycle will consider Day 1 as start of Cycle and not the days since first study dose as for Cycle 2.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### Table 4. Visit Labels

| Period | Visit | TFLs Label |
|---|---|---|
| Screening: Day -28 to Day -1 | Screening Day -28 to Day -1 | Screening |
| Cycle 1 | Cycle 1 Day 1 | Baseline |
| | Cycle 1 Day 8 | C1D8 |
| | Cycle 1 Day 15 | C1D15 |
| Cycle 2 | Cycle 2 Day 29 | C2D29 |
| | Cycle 2 Day 36 | C2D36 |
| | Cycle 2 Day 43 | C2D43 |
| Cycle 3 | Cycle 3 Day 1 | C3D1 |
| Cycle n | Cycle n Day 1 | CnD1 |
| End of Treatment: +7 days after last dose of study treatment. | End of Treatment Visit | ЕОТ |
| Safety Follow-Up: 60 ± 7 days after last dose of study treatment. | Safety Follow-Up | SFU |
| Follow-Up: every eight months (± 7 days) until death, disease progression or initiation of subsequent anticancer therapy whichever comes first. | Follow-Up | FUn |

### Summaries of baseline and change from baseline

Baseline and change from baseline will be calculated for all assessments, including additional assessments (if applicable), as follows:

- Baseline is defined as the last available assessment prior to first dose of both study treatment, including additional assessments (where applicable). Assessments that occurred on the same day as first dose, when time of assessment is not available, will be assumed to be prior to first dose (unless the assessment is planned after first dose in the protocol).
- Change from baseline will be calculated as the difference between the post-baseline assessment value and the baseline value.

Whenever applicable, percent change from baseline will be calculated as the difference between the post-baseline assessment value and baseline value divided by the baseline value multiplied by 100. Percent change will only be calculated when possible (e.g. if baseline value is 0 or the data has negative values as a possible occurrence percent change will not be calculated).

## Unscheduled visit / Repeat assessments

Data obtained at unscheduled and repeat assessments will be considered for the derivation of baseline, worst on-treatment result for safety analyses (clinical safety laboratory evaluation and vital signs), and time to event analyses.

All other data from unscheduled or repeat assessments will not be included in summaries and will only be presented in data listings, if not otherwise specified.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### N

N will be the number of patients in the specified population and group.

## Summary presentation

All outputs will be presented by basket as defined in SAP section 6.1 and overall if not otherwise specified.

#### Continuous data

Continuous data will be summarized using number of patients (n), mean, standard deviation, median, first and third quartiles (Q1 and Q3), minimum value, and maximum value.

#### Categorical data

Categorical data will be summarized using n and percentage.

- All categories will be presented, even if no patients are counted in a particular category, unless otherwise stated.
- A missing category will be displayed in all tables for categories where at least one missing value exists, unless otherwise specified.
- Counts of zero in any category will be presented without percentage.
- All summary percentages will be calculated using N, unless otherwise stated in a footnote.
- For AEs, medical history, prior and concomitant medications, the counts are based on single counts of patients with multiple events/treatments under the same category, while the percentages are calculated using N. Counts will be displayed by descending order of frequency for the overall group by dictionary hierarchy.

#### Precision of summary statistics

- Integer Sample size (n, N) and number of missing data (if displayed).
- One additional decimal place than reported/collected Mean, median, other percentile, confidence interval.
- Two additional decimal places than reported/collected Standard deviation.
- Same number of decimal places as reported/collected Minimum, maximum.
- Percentages One decimal place.

#### Study day

Study day will be calculated as (assessment date – date of first study treatment dose) for prebaseline assessments and [(assessment date – date of first study treatment dose) + 1] for postbaseline assessments, i.e. there will be no study day 0 and study day 1 will correspond to the first study treatment dose.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

### Ordering

Data will be presented in listings in order of group, patient ID, visit, assessment date/time, and assessment type/parameters chronological order unless otherwise specified. In case of clinical laboratory results, the listings will be presented in order of group, patient ID, parameter, assessment date/time, visit.

#### Date format

Dates will be presented in format DDMMMYYYY.

#### Dictionaries

Latest version of Medical Dictionary for Regulatory Activities (MedDRA) will be used for the relevant outputs.

Latest version of World Health Organization (WHO) Drug Global B3 will be used for the relevant outputs.

NCI-CTCAE v5.0 will be used for the relevant outputs.

The version will be documented in the footnote of the corresponding TFLs.

### File naming

Each TFL output file will be named with a t, l, or f added before the TFL number to denote the output type and then according to its table numbering in the following way: Table 14.2-1.1 would be t14\_2\_1\_1, Table 14.2-11 would be t14\_2\_11, Listing 16.2.7-1.1 would be l16\_2\_7\_1\_1, and Figure 14.2-2.1 would be f14\_2\_1.

#### Reporting guidelines

- Page Orientation: Landscape.
- Tables and listings: will be created in .rtf.
- · Figures: will be generated directly in .rtf.
- Font: Courier New font with minimum of 8-point font size.
- . Margins: Left: 3.8 cm, Right: 2 cm, Top: 3 cm, Bottom: 2 cm, on A4 paper.
- Columns header will be left aligned for listings.

## 8 Analysis Sets

#### All Patients Analysis Set



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

of whether they received the study drug or not.

### Full Analysis Set

The full analysis set (FAS) will consist of all patients who received at least one dose of both study medications. This analysis set will be used for all safety and efficacy analyses.

#### Stage 1 Analysis Set

The Stage 1 analysis set (S1AS) will consist of the first 13 patients who have completed at least one cycle of therapy and who have received a minimum of 75% of prescribed study therapy during Cycle 1. This analysis set will be used only for the purpose of the Stage 1 efficacy analysis.

#### **Evaluable Analysis Set**

The evaluable analysis set (EAS) will consist of all patients who received at least one dose of study drug and have at least one post-treatment study evaluation or who have discontinued therapy prior to the first post-treatment study evaluation due to clinical progressive disease or drug-related adverse events. This analysis set will be used for the evaluation of the primary efficacy endpoint, i.e., ORR, and all the secondary efficacy endpoints.

#### PK Analysis Set

The PK analysis set will consist of all patients who have received at least one dose of study medication and have at least one post dose PK measurement. This analysis set will be used for PK analyses.

Given that the study was early terminated and an abbreviated CSR focusing mostly on safety data will be prepared, S1AS, EAS and PK will not be used in any analysis.

## 9 Methods of Analyses and Presentations

#### 9.1 PATIENT DISPOSITION

The patient disposition data will be presented by basket and overall, on the All Patients Analysis Set. The number and percentage of patients belonging to the following disposition modalities will be presented along with the reason for discontinuation: patients enrolled, patients eligible for inclusion in the study, patients completed/discontinued screening, patients rescreened, patients treated, patients completed/discontinued treatment, patients completed/discontinued study.

The number and percentage of patients in each analysis set will also be presented.

A consort diagram with disposition information will also be provided.

In addition, information on analysis sets, study completion and discontinuation, informed consent



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

and failed inclusion and exclusion criteria will be included in the listings.

## 9.2 PROTOCOL DEVIATIONS AND/OR VIOLATIONS

ICH E3 Q&A R1 defines a protocol deviation as "any change, divergence, or departure from the study design or procedures defined in the protocol", and important protocol deviations as "a subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a patient's rights, safety, or well-being". The non-compliance may be either on the part of the patient, the investigator, or the study site staff. The list of potential protocol deviations, including classification (Important/Non-important) for each protocol deviation, will be pre-defined in the Protocol Deviation Criteria Form (PDCF).

Protocol deviations identified during the trial by the Clinical Research Associates (CRAs), Medical Monitors, or Data Managers will be tracked throughout the study using a protocol deviation tracker and classified as Important/Non-important. All protocol deviations will be read into SAS® prior to reporting.

Prior to data lock for the primary and final analyses, a review classification meeting will be held to review protocol deviations and classifications, and to agree on the final analysis sets.

Important protocol deviations will be summarized (frequencies and percentages) by deviation category and summary term on the FAS.

A listing of all protocol deviations will be provided for all patients.

#### 9.3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

The following demographic and baseline characteristics will be summarized using descriptive statistics and presented by basket and overall on the FAS:

- Age at baseline (years), as derived in the eCRF continuous and categorical using EudraCT categorization (18-64, 65-84, ≥ 85)
- Sex at Birth
- Childbearing/Reproductive potential
- Ethnicity
- Race
- Height at baseline (cm)
- Weight at baseline (kg)
- ECOG performance status at baseline
- Smoking history
- Gene/Codon/Amino acid change as reported in the eCRF



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

The following disease history characteristics will be summarized using descriptive statistics and presented by basket and overall on the FAS:

- Cancer Diagnosis (only reported diagnosis will be displayed, not all categories displayed in the CRF)
- Time since initial diagnosis (in months)
- Disease stage at initial diagnosis (from 1 to 4)
- Disease stage at enrollment (from 1 to 4)
- Prior Radiation Therapies (Yes/No)

Time since initial diagnosis will be calculated as [(date of first dose of study treatment - date of diagnosis) / 30.4375].

In addition, listings of the above data will be produced for all patients.

A by-patient, detailed listing of smoking history will be also presented.

#### 9.4 MEDICAL HISTORY AND CONCOMITANT DISEASES

Medical history and concomitant diseases will be coded using MedDRA.

Medical histories are defined as events reported on the Medical History and Disease History eCRF pages, which started before the first study treatment date and were not ongoing at the first study treatment date.

Concomitant diseases are defined as diseases which started before the first study treatment date but were ongoing at the first study treatment date.

The number and percentage of patients with a medical history will be tabulated by basket and overall, by system organ class (SOC) and preferred term (PT) on the FAS. A by-patient listing will be produced.

The number and percentage of patients with a concomitant disease will be tabulated by basket and overall, for each SOC and PT using the FAS. A by-patient listing will be produced.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 9.5 PRIOR THERAPIES

The following summaries will be created by basket and overall, on the FAS:

#### Prior radiotherapy:

- Received at least one prior radiotherapy
- Number of prior radiotherapy courses
- Site of prior radiotherapies (only reported sites will be displayed, not all categories displayed in the eCRF)
- Most recent therapy received before study treatment start: duration of therapy (months)
  and site

For prior radiotherapy, duration in months will be calculated as [(end date of therapy – start date of therapy) + 1] / 30.4375.

#### Prior Systemic Anti-Cancer Therapies:

- Received at least one prior anti-cancer therapy
- Lines of prior anti-cancer therapies
- Most recent therapy received before study treatment start: regimen name, BOR, duration
  of therapy (months), time since BOR, time since relapse/progression, and reason for
  discontinuation.

For prior anti-cancer therapies, duration in months will be calculated as [(end date of therapy - start date of therapy) + 1] / 30.4375.

Time since BOR (months) will be calculated as [(date of first study treatment - date of BOR) + 1] / 30.4375.

Time since relapse/progression (months) will be calculated as [(date of first study treatment - date of Relapse/Progression) + 1] / 30.4375.

#### Prior and Concomitant Medication:

Medications other than the study treatment will be coded using the WHO Drug Global dictionary. The version of the dictionary will be provided in the corresponding TFLs footnotes.

#### Medications will be defined as follows:

- Prior Medication: any medications whose end date is before the first study treatment date.
- Concomitant Medication: any medications whose start or end date is either the same or after the first dose of study treatment and up to the end of the on-treatment period.
  - Any medication with a missing medication end date will be assumed to be concomitant medication.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 9.5 PRIOR THERAPIES

The following summaries will be created by basket and overall, on the FAS:

## Prior radiotherapy:

- Received at least one prior radiotherapy
- Number of prior radiotherapy courses
- Site of prior radiotherapies (only reported sites will be displayed, not all categories displayed in the eCRF)
- Most recent therapy received before study treatment start: duration of therapy (months)
  and site

For prior radiotherapy, duration in months will be calculated as [(end date of therapy – start date of therapy) + 1] / 30.4375.

#### Prior Systemic Anti-Cancer Therapies:

- Received at least one prior anti-cancer therapy
- Lines of prior anti-cancer therapies
- Most recent therapy received before study treatment start: regimen name, BOR, duration
  of therapy (months), time since BOR, time since relapse/progression, and reason for
  discontinuation.

For prior anti-cancer therapies, duration in months will be calculated as [(end date of therapy - start date of therapy) + 1] / 30.4375.

Time since BOR (months) will be calculated as [(date of first study treatment - date of BOR) + 1] / 30.4375.

Time since relapse/progression (months) will be calculated as [(date of first study treatment - date of Relapse/Progression) + 1] / 30.4375.

## Prior and Concomitant Medication:

Medications other than the study treatment will be coded using the WHO Drug Global dictionary. The version of the dictionary will be provided in the corresponding TFLs footnotes.

#### Medications will be defined as follows:

- Prior Medication: any medications whose end date is before the first study treatment date.
- Concomitant Medication: any medications whose start or end date is either the same or after the first dose of study treatment and up to the end of the on-treatment period.
  - Any medication with a missing medication end date will be assumed to be concomitant medication.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Ongoing medications are considered as concomitant medications.

The number and percentage of patients with prior and concomitant medications will be tabulated by basket and overall, by Anatomical Therapeutic Chemical Classification (ATC) and preferred term (PT) on the FAS. A by-patient listing will be produced for prior and concomitant medications as well as for all prior therapies.

On treatment Radiation, Surgery and Medical Procedures, and Blood Transfusions:

On treatment Radiation, Surgery and Medical Procedures, and Blood Transfusions will be listed on the FAS.

## 9.6 STUDY DRUG EXPOSURE AND/OR COMPLIANCE

Duration on treatment and cumulative dose received will be calculated for both ulixertinib and hydroychloroquine as defined below with the same tables and listings.

- Number of cycles received =
   Number of cycles where the patient received at least one dose.
- Duration of exposure (months) =
  [(Date of last known treatment dosing with study treatment date of initial dosing with ulixertinib) + 1] / 30.4375
- Planned cumulative dose (mg) =
   Number of cycles received x number of doses per day x mg prescribed per dose.
- Actual cumulative dose received (mg) =
   For each time period reported in the eCRF:
   (Stop date Start date + 1)\*Dose
   Sum all available periods where dose was given.
- Relative dose intensity =

100 x Actual dose intensity / Planned dose intensity, with:

- Actual dose intensity (mg/day) = Actual cumulative dose received (mg) / Duration of exposure (days).
- Planned dose intensity (mg/day) = Planned cumulative dose (mg) / Duration of exposure (days).

Summary statistics will be presented for the number of cycles received, duration of exposure, actual cumulative dose, and relative dose intensity, by basket and overall on the FAS.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

The number and percentage of patients having at least one dosing interruption or adjustment will be tabulated with the corresponding reason by basket and overall on the FAS. A by-patient listing will be produced.

## 9.7 PHARMACOKINETIC/ PHARMACODYNAMIC ENDPOINTS AND ANALYSES

#### 9.7.1 Pharmacokinetic Data

For patients enrolled in stage 1 of each basket, PK concentrations of ulixertinib and hydroxychloroquine will be determined pre-dose and post-dose in plasma at cycle 1 day 15. Summary parameters such as AUC, Cmax, Cmin, t1/2, tmax will be calculated.

PK parameters in plasma will be tabulated and summarized, by basket, using descriptive statistics (e.g., sample size, arithmetic and geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum).

For patients enrolled in stage 2 of each basket, PK concentration of ulixertinib will be measured on cycle 1 day 15. This will be a single timepoint collection prior to taking study drug on this day.

PK values will be presented in by-patient listings.

PK analysis will be conducted on the PK analysis set.

#### 9.7.2 Pharmacodynamic Data

Not applicable.

#### 9.8 EFFICACY DATA ENDPOINTS AND ANALYSES

## 9.8.1 Primary Efficacy

## 9.8.1.1 Overall Response Rate (ORR)

Tumor response will be assessed by the Investigator using RECIST 1.1 criteria1.

Disease assessments must include all known or suspected sites of disease; therefore, the decision for body areas to be scanned will depend on the extent of disease. The minimum recommended body areas to be scanned is chest, abdomen, and pelvis.

Disease assessments will be evaluated radiologically and conducted at baseline (within 28 days prior to the first dose of study treatment) and then every 8 weeks thereafter  $\leq$  7 days prior to the start of the following cycle (e.g., prior to cycle 3 day one, cycle 5 day 1, cycle 7 day 1, etc.). If a response is observed (CR or PR), confirmation of response is required  $\geq$  4 weeks from the first documentation of response. Disease assessments will continue until disease progression, the



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

initiation of subsequent anti-cancer therapy, or death. In addition, radiological tumor assessments will be conducted whenever disease progression is suspected (e.g., symptomatic deterioration) or when clinically indicated. The schedule of tumor assessments should be fixed according to the calendar, starting with cycle one day one, regardless of treatment delays or interruptions due to toxicity.

Brain CT or MRI scans are required at baseline for all patients with stable brain lesions and for those for whom Central Nervous System (CNS) involvement is suspected. If stable brain metastases are present at baseline, brain imaging should be repeated at each tumor assessment. Otherwise, brain imaging will be conducted post-baseline only when clinically indicated.

The table below provides a summary of the overall response status determination at each time point.

Table 5. Evaluation of Overall Response

| Target lesions | get lesions Non-target lesions | | Overall response |
|---|---|---|---|
| CR | CR (or no non-target lesions) | No | CR |
| No target lesion a | CR | No | CR |
| CR | NE b | No | PR |
| CR | Non-CR/non-PD | No | PR |
| PR | Non-PD and NE (or no non-target lesions) b | No | PR |
| SD | Non-PD and NE (or no non-target lesions) b | No | SD |
| Not all evaluated | Non-PD | No | NE |
| No target lesion a | Not all evaluated | No | NE |
| No target lesion a | Non-CR/non-PD | No | Non-CR/non-PD |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |
| No target lesion a | Unequivocal PD | Yes or No | PD |
| No target lesion a | Any | Yes PD | |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, and NE = not evaluable

The ORR is defined as the number of patients having a confirmed response of either CR or PR divided by the total number of patients in the FAS/EAS. ORR will be calculated with the 95% confidence intervals (CIs), by basket and overall on the FAS and EAS. The 95% CIs will be estimated using the Clopper-Pearson method.

Complete and partial response must be confirmed by a repeat assessment performed ≥ 4 weeks after the criteria for response are first met. Date of confirmed CR/PR will be the date of the first CR/PR that qualifies for confirmation. Additionally, patients with no post-baseline efficacy measurement due to reasons accountable for disease progression, will be assessed as non-evaluable and will count in the denominator of the ORR.

Defined as no target lesion at baseline.

<sup>&</sup>lt;sup>b</sup> Not evaluable is defined as when either no or only a subset of lesion measurements is made at an assessment.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BOR will be assessed based on the tumor response at different evaluation time points from baseline until the first documented disease progression for RECIST or the last response assessment if there is no documented disease progression at the time of the analysis. The order used to determine BOR is CR>PR>SD>PD, ignoring visits with missing tumor assessments. For SD to qualify for BOR, the SD assessment should be at least 6 weeks after first ulixertinib dose. BOR date in this case will be the date of the first SD/PR/CR documented after 6 weeks.

The following table, based on Table 3 from the RECIST 1.1 guidelines<sup>1</sup>, summarizes the algorithm describing how confirmed response and BOR are determined from the overall tumor assessments.

Table 6. Evaluation of Confirmed BOR

| | Overall | Overall response | |
|---|---|---|---|
| | response | subsequent | |
| Case | first timepoint | timepoint | Confirmed response/BOR |
| 1 | CR | CR | CR (if assessments at least 28 days apart). (note: sequence of CR – |
| | | | NE – CR would be considered as confirmed CR) |
| 2 | CR | PR | SD, PD, or PR |
| | | | <ul> <li>If CR truly met at first timepoint, any subsequent assessment</li> </ul> |
| | | | of PR should make the disease PD at that point. That is, |
| | | | neither a PR nor SD may follow CR. |
| | | | <ul> <li>Therefore, SD, if CR assessment &gt;=6 weeks (42 days after date</li> </ul> |
| | | | of first treatment), otherwise PD. |
| | | | However, BOR may be PR if subsequent scans suggest small |
| | | | lesions were still present at first assessment (in which case |
| | | | first assessment of CR should be changed to PR) |
| 3 | CR | SD | SD or PD |
| | | | SD, if CR or SD assessment >=6 weeks (42 days) after date of |
| | | | first treatment, |
| | | | otherwise PD |
| 4 | CR | PD | SD or PD |
| | | | SD, if CR assessment >=6 weeks (42 days after date of first |
| | | | treatment), |
| <u> </u> | | | otherwise PD |
| 5 | CR | NE | SD or NE |
| | | | SD, if CR assessment >=6 weeks (42 days after date of first |
| | | | treatment |
| _ | nn. | CD. | otherwise NE |
| 7 | PR | CR | PR (if assessments at least 28 days apart). |
| <b>'</b> | PR | PR | PR (if assessments at least 28 days apart). (note: sequence of PR – NE – PR would be considered as confirmed PR) |
| | | | Where there are cases of more than one SD assessment between |
| | | | two PR assessments, then this should be discussed. |
| 8 | PR | SD | SD SD |
| 9 | PR | PD | SD or PD |
| , | FN | 10 | SD, if PR assessment >=6 weeks (42 days after date of first) |
| | | | treatment), |
| | | | otherwise PD |
| | | | other wise 10 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| | Overall response | Overall response<br>subsequent | |
|---|---|---|---|
| Case | first timepoint | timepoint | Confirmed response/BOR |
| 10 | PR | NE | SD or NE SD, if PR assessment >= 6 weeks (42 days after date of first treatment), otherwise NE |
| 11 | SD | SD, PR, CR | SD |
| 12 | SD | PD | SD or PD SD, if SD assessment >=6 weeks (42 days after date of first treatment), otherwise PD |
| 13 | SD | NE | SD or NE SD, if SD assessment >= 6 weeks (42 days after date of first treatment), otherwise NE |
| 14 | NE, - | SD | SD |
| 15 | CR, PR, SD | - | SD or NE SD, if assessment >=6 weeks (42 days after date of first treatment) and does not qualify for CR or PR, otherwise NE. |
| 16 | PD | | PD. Ignore all assessments after initial overall response of PD. |
| 17 | NE | NE | NE<br>Where all assessments are Not evaluable |

For changes in target tumor size, spider and waterfall plots will be presented. For all response assessments, swimmer plots will be presented. Target and Non-Target Lesions response assessments and incidence of new lesions will be summarized by visit and listed. All response assessments will be listed.

## 9.8.2 Secondary Efficacy

## **9.8.2.1** Progression-free Survival (PFS)

The PFS (in months) is defined as the time from the first ulixertinib dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

PFS = [(Date of first PD/death - Date of first study treatment) + 1] / 30.4375

Patients with no documented progression or death will be censored at the last available tumor assessment (last assessment that is CR, PR or SD):

PFS = [(Date of last assessment where patient is PD free – Date of first study treatment) + 1] / 30.4375



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

For patients with no post baseline tumor assessment a censored PFS at day 1 will be considered.

PFS = (Date of first study treatment - Date of first study treatment) + 1

The analysis of PFS will be performed with a Kaplan-Meier method (product-limit estimates) and a summary of associated statistics will be presented including corresponding two-sided 95% CI. The CI for the median will be calculated according to Brookmeyer and Crowley and CI for the survival function estimates at Month 3, 6, 9, 12, and 18 will be derived using the log-log transformation (SAS PROC LIFETEST CONFTYPE=LOGLOG). However, the final choice of timepoints may be updated dependent upon the data.

## 9.8.3 Exploratory Efficacy

## 9.8.3.1 Duration of Response (DOR)

The DOR (in months) is defined as the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause. Only patients with BOR of CR or PR (i.e. responders) will be included in the analysis of DOR.

DOR = [(Date of first PD/death - Date of first recorded confirmed CR/PR) + 1] / 30.4375

Patients with no documented progression or death after CR or PR will be censored at the last available tumor assessment (last assessment that is CR, PR, or SD):

DOR = [(Date of last assessment where patient is PD free – Date of first recorded CR/PR) + 1] / 30.4375

The analysis of DOR will be performed with a Kaplan-Meier method (product-limit estimates) and a summary of associated statistics will be presented including corresponding two-sided 95% CI. The CI for the median will be calculated according to Brookmeyer and Crowley and CI for the survival function estimates at Month 3, 6, 9, 12, and 18 will be derived using the log-log transformation (SAS PROC LIFETEST CONFTYPE=LOGLOG), only if there are sufficient data for responders. However, the final choice of timepoints may be updated dependent upon the data.

## 9.8.3.2 Overall Survival (OS)

The OS (in months) is defined as the time from first treatment to death. Patients who did not die during the study will be censored at the last known alive date.

OS = [(Date of death – Date of first study treatment) + 1] / 30.4375

For censored patients:



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

OS = [(Last known alive date - Date of first study treatment) + 1] / 30.4375

The last known alive date will be determined among study treatment administrations, any visits where at least one assessment has been completed, or any follow-up assessment where the patient has been confirmed to be alive.

OS will be analyzed using the same Kaplan-Meier method used to analyze the DOR.

#### 9.9 SAFETY DATA ENDPOINTS AND ANALYSES

All safety analyses will be performed by basket and overall on the FAS, using descriptive statistics.

## 9.9.1 Adverse Events (AEs)

The following definitions will be used:

- Treatment-emergent AEs (TEAEs): Treatment-emergent adverse event (TEAE) is defined
  as any AE that emerges during on-treatment period.
- Related AEs: AEs suspected by the Investigator and/or Sponsor to have a relationship to study treatment (as recorded on the AE eCRF page, Causality = Related, Possibly Related, or missing), including ulixertinib or hydroxychloroquine or both.
- Serious Adverse Events (SAE): serious AEs (as recorded on the AE eCRF page, Does AE Meet the Definition of an SAE = Yes).
- AEs leading to treatment discontinuation: AEs leading to permanent discontinuation of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Drug withdrawn).
- AEs leading to dose reduction: AEs leading to dose reduction of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Dose Reduced).
- AEs leading to treatment interruption: AEs leading to treatment interruption of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Drug Interrupted).
- AEs leading to Death: adverse event leading to death (as recorded on the AE eCRF page, Results in death, or Outcome = Fatal, or Grade = 5).

An overview summary table will present the number and percentage of patients with a TEAE, all treatment-related adverse events will be indicated as Ulixertinib-related or Hydroxychloroquine-related or both, including:

- TEAEs / TEAEs related to study treatment
- SAEs / SAEs related to study treatment
- TEAEs leading to treatment discontinuation / TEAEs related to study treatment leading to treatment discontinuation



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

- TEAEs leading to treatment discontinuation within 1 cycle / TEAEs related to study treatment leading to treatment discontinuation within 1 cycle
- TEAEs leading to treatment discontinuation following 1 cycle / TEAEs related to study treatment leading to treatment discontinuation following 1 cycle
- TEAEs leading to treatment interruption / TEAEs related to study treatment leading to treatment interruption
- TEAEs leading to treatment interruption within 1 cycle / TEAEs related to study treatment leading to treatment interruption within 1 cycle
- TEAEs leading to treatment interruption following 1 cycle / TEAEs related to study treatment leading to treatment interruption following 1 cycle
- TEAEs leading to dose reduction / TEAEs related to study treatment leading to dose reduction
- TEAEs leading to dose reduction within 1 cycle / TEAEs related to study treatment leading to dose reduction within cycle 1
- TEAEs leading to dose reduction following 1 cycle / TEAEs related to study treatment leading to dose reduction following cycle 1
- TEAEs leading to death / TEAEs related to study treatment leading to death
- TEAEs with grade ≥ 3 / TEAEs related to study treatment with grade ≥ 3

In addition, the following tables will be produced by SOC and PT:

- TEAEs / TEAEs related to study treatment
- Serious TEAEs / Serious TEAEs related to study treatment
- TEAEs and maximum CTCAE grade / TEAEs related to study treatment and maximum CTCAE grade
- TEAEs leading to treatment discontinuation within/following cycle 1 / TEAEs related to study treatment leading to treatment discontinuation within/following cycle 1
- TEAEs leading to treatment interruption within/following cycle 1 / TEAEs related to study treatment leading to treatment interruption within/following cycle 1
- TEAEs leading to dose reduction within/following cycle 1 / TEAEs related to study treatment leading to dose reduction within/following cycle 1
- TEAEs leading to death / TEAEs related to study treatment leading to death

The following tables will be produced by PT:

- TEAEs / TEAEs related to study treatment
- Serious TEAEs / Serious TEAEs related to study treatment

A patient with multiple occurrences of an AE will be counted only once in the AE category. SOCs will be sorted by descending order of frequency for the overall group, PTs will be sorted by descending order of frequency for the overall group within each SOC.

All deaths will be summarized and listed with the corresponding reasons, split by overall deaths, and deaths occurring after the first dose of ulixertinib.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

The following listings will be provided:

- All AEs (All Patient Set)
- TEAEs (FAS)
- SAEs (FAS)
- Deaths (FAS)

## 9.9.2 Clinical Safety Laboratory Evaluation

All haematology, biochemistry, coagulation and urinalysis laboratory tests collected will be reported.

The numerical measurements and change from baseline of all haematology, biochemistry, and urinalysis laboratory tests will be summarized using descriptive summary statistics for each visit.

For laboratory tests covered by the NCI-CTCAE (version 5), laboratory data will be graded accordingly. 'Normal' will be assigned for all non-missing values not graded as 1 or higher. For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classifications based on laboratory normal ranges as collected in the CRF. Separate tables will be created for Gradable and Non-gradable laboratory values.

Haematology and biochemistry laboratory tests will be summarized by:

- Tables (Gradable and Non-gradable) to describe the worst on-treatment value by cycle.
- Shift tables (Gradable and Non-gradable) to compare baseline to the worst on-treatment value.

Listings of all laboratory data with values flagged to show the corresponding NCI-CTCAE grades and the classifications relative to the laboratory normal ranges will also be provided. Also results of serum pregnancy tests and tumor markers will be listed.

## 9.9.3 Other Safety data

#### 9.9.3.1 Vital signs

Vital signs include the following parameters: systolic blood pressure (SBP) (mmHg), diastolic blood pressure (DBP) (mmHg), pulse (beats/min), respiratory rate (breaths/min), pulse oximetry (%) and temperature (°C).

The numerical measurements and change from baseline of all vital signs parameters will be summarized using descriptive summary statistics for each visit.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Shift tables of baseline to worst on-treatment result (low, normal, high, very high) will be presented.

Table 7. Thresholds for classification of vital signs test results

| Vital Sign | Criteria | Flag |
|------------------|-------------------|-----------|
| Temperature | < 36.4°C | Low |
| | 36.4°C – 37.7°C | Normal |
| | > 37.7°C | High |
| Pulse | < 55 bpm | Low |
| | 55-100 bpm | Normal |
| | 101-150 bpm | High |
| | > 150 bpm | Very High |
| Respiratory rate | <12 breaths/min | Low |
| | 12-16 breaths/min | Normal |
| | >16 breaths/min | High |
| Pulse oximetry | <90 % | Very Low |
| | 90-95 % | Low |
| | ≥95 % | Normal |
| Systolic Blood | < 90 mmHg | Low |
| Pressure | 90-130 mmHg | Normal |
| | 131-160 mmHg | High |
| | ≥161 mmHg | Very High |
| Diastolic Blood | < 60 mmHg | Low |
| Pressure | 60-85 mmHg | Normal |
| | 86-100 mmHg | High |
| | ≥ 101 mmHg | Very High |

All Vital Signs will be Listed.

## 9.9.3.2 Electrocardiogram (ECG)

ECG includes the following parameters: Heart Rate (beats/min), PR Interval (msec), QRS Duration (msec), RR Interval (msec), QT Interval (msec), and QT interval corrected for heart rate by the Fridericia's formula (QTcF) Interval (msec).

The numerical measurements and change from baseline of all ECG parameters will be summarized using descriptive summary statistics for each visit.

A listing of ECG evaluations will be created.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 9.9.3.3 ECHO

ECHO assessments at baseline will be summarized using descriptive summary statistics.

A listing of ECHO evaluations will be created.

### 9.9.3.4 Physical Examination

Physical Examination includes the following parameters: HEENT, Thorax, Abdomen, Skin and Mucosae, Neurological, Extremities, Urogenital, General Appearance, Heart, Back, and Lymph Nodes.

All physical examination assessments at baseline will be summarized using descriptive summary statistics.

A listing of physical examination evaluations will be created.

## 9.9.3.5 Ophthalmology exam

A listing of ophthalmological examination assessments will be created.

## 9.9.3.6 ECOG Performance status

The number and percentages of patients will be tabulated for ECOG performance score categories at each visit.

A listing of all ECOG Performance status at all visits will be presented.

## 10 Interim Analyses

No interim analysis is planned.

## 11 Changes to Planned Analyses

No major changes to analyses planned in the protocol are expected.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 12 Document History

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 17Jul2023 | 1.0 | David Manteigas | First SAP Version. |
| 20-Aug-2024 | 1.1 | Julien Lucas | Updated version to include required changes after the study was terminated early. |
| 02-Sep-2024 | 2.0 | Julien Lucas | Second SAP version. |

## 13 References

 Eisenhauer EA, Therasse P, Bogaerts J, et al. (2009), New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer; 45:228-47.


Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# 14 Appendices

## 14.1 Schedule of events

| | | | On-Treatment Period | | | = 28 days | | Post-Treatment Period | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | :le 2 | Cycle 3+ | EOT" | Safety<br>Follow-<br>Up <sup>™</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1 <sup>tv</sup> | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| Informed Consent | Х | | | | | | | | | |
| Demographics | Х | | | | | | | | | |
| Cancer History <sup>v</sup> | Х | | | | | | | | | |
| Medical History | Х | | | | | | | | | |
| Eligibility Criteria | Х | | | | | | | | | |
| Clinical Assessments | | | | | | | | | | |
| Vital Signs <sup>vl</sup> | Х | X | X | X | X | X | X | X | X | |
| Physical Exam <sup>vII</sup> | х | X | X | x | X | x | x | X | Х | |
| ECOG Score | х | X | X | x | X | х | x | X | х | |
| ECG | х | | X | x | x | | | X | | |
| Echocardiogram | × | | ACI | | | | | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

| | | | On-Trea | tment Period | : One Cycle | = 28 days | | Pos | t-Treatment P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | :le 2 | Cycle 3+ | EOTII | Safety<br>Follow-<br>Up <sup>™</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1 <sup>lv</sup> | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| Ophthalmologic Exam <sup>vill</sup> | Х | | | | X | | X | | | |
| Adverse event collection | Х | | x | | | | | | | |
| Concomitant medications | Х | | X | | | | | | | |
| Laboratory Studies <sup>lx</sup> | | | | | | | | | | |
| Hematology | Х | Х | х | X | х | х | X | X | X | |
| Chemistry | Х | Х | X | X | X | X | X | X | X | |
| Creatine kinase <sup>x</sup> | Х | | | A | CI | | | | | |
| LDH and Phosphorus | Х | Х | X | X | X | A | CI | | | |
| Coagulation | Х | | | A | CI | | | | | |
| Urinalysis | Х | | | А | CI | | | | | |
| Tumor Marker <sup>xl</sup> | | Х | | | X | | X | X | | |
| Pregnancy Test <sup>xll</sup> | Х | | ACI | | | | | | | |
| Disease Assessments | | | | | | | | | | |
| CT Scans or MRIXII | X | | | | | | X | X | | Xxiv |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| | | | On-Trea | tment Period | : One Cycle | = 28 days | | Post-Treatment Period | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | ile 2 | Cycle 3+ | EOT" | Safety<br>Follow-<br>Up <sup>™</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1₩ | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| RECIST 1.1 Assessment | Х | | | | | | Х | Х | | X |
| Treatment Compliance ar | nd Distribution | | | | | | | | | |
| Hydroxychloroquine | | X | | | X | | х | | | |
| Ulixertinib | | X | | | X | | х | | | |
| Treatment administration on site | | | | X <sup>15</sup> | | | x | | | |
| Meal provided by site | | | | Х | | | X16 | | | |

Abbreviations: ACI = as clinically indicated; LDH = lactate dehydrogenase; CT = computed tomography; MRI = magnetic resonance imaging; ECG = electrocardiogram; EOT = end of treatment



Protocol: BVD-523-HCQ Statistical Analysis Plan:

- ¹ Screening procedures must be completed ≤ 28 days prior to C1D1 unless noted otherwise.
- <sup>2</sup> The end of treatment visit should occur when the decision to discontinue treatment is made. If this visit overlaps with a regularly scheduled visit, only the procedures listed in the calendar for the EOT visit will be performed. All end of treatment procedures should be completed within 7 days after the decision to discontinue treatment has been made.
- 3 Patients will have a safety follow-up visit 60 days (± 7 days) after last dose of study drug.
- 4 C1D1 procedures do not need to be repeated if screening procedures were performed ≤ 7 days of the start of treatment.
- Oncologic history of the malignancy under study including prior regimens (duration of therapy, best response on therapy, date of discontinuation, and reason for discontinuation), surgery, and radiation therapy.
- <sup>6</sup> Vital signs include systolic/diastolic blood pressure, heart rate, respiration rate, pulse oximetry, weight, and body temperature. Height will be captured at screening only.
- 7 If necessary to facilitate scheduling, the physical exam may occur one day prior to study treatment.
- <sup>8</sup> A standard ophthalmologic exam must be completed at screening, C2D1, and every 3 cycles thereafter (i.e. C5D1, C8D1, etc.) and as clinically indicated to assess for retinopathies. All assessments must be conducted up to 7 days prior to the clinic visit to enable timely results review.
- <sup>9</sup> Labs may be performed ≤ 3 days prior to a scheduled day one visit except for C1D1 labs which may be completed ≤ 7 days prior to C1D1.
- 10 After screening, creatine kinase should only be drawn if creatinine is elevated.
- <sup>11</sup> Tumor marker should be drawn on day one of each cycle. Tumor markers will be disease specific: pancreatic adenocarcinoma only CA 19-9; colorectal carcinoma only CEA; cholangiocarcinoma only CEA and CA 19-9. Tumor markers are not required for patients with esophageal or stomach cancers.
- <sup>12</sup> Pregnancy test (serum or urine) must be obtained at screening ≤ 7 days prior to C1D1 for all women of childbearing potential and as clinically indicated while on treatment.
- <sup>13</sup> Disease assessment will be repeated every 8 weeks (± 7 days) regardless of dose holds or delays. Patients who discontinue treatment for reasons other than progression will have computed tomography (CT) scans at the EOT visit (unless their previous restaging was performed within 6 weeks).
- 14 Patients that discontinue study treatment for any reason other than disease progression, must continue to have disease assessments every 8 weeks (± 7 days) until disease progression or initiation of subsequent anticancer therapy.
- 15 Patient should be instructed to not take their study treatment before arriving at clinic. Study treatment and meal should be provided after the pre-dose PK draw.
- 16 Meal is only required to be given at C3D1, i.e., at the time of drug administration for ctDNA and tumor biopsy for stage 1.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

## 14.2 Schedule of Correlative Sample Collection

| 0 | | | | | | C11 | D15 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Correlative<br>Test | | | Pre-<br>Dose | | | ı | Post-D | ose | | | C3D1 | EOT |
| Time Point<br>(hour) | Screening | C1D1 | | 0.5 | 1 | 2 | 4 | 6 | 8 | 12 | ± 7 | |
| Window (min) | | | ≤ 60 | ±2 | ±3 | ±6 | ±12 | ±18 | ±24 | ±36 | days | |
| | | | | STA | GE 1 | | | | | | | |
| PK Blood <sup>1</sup> | | | Х | X | Х | Х | Х | Х | Х | X | | |
| ctDNA | | X | | | | | | | | | X <sup>2</sup> | X <sup>3</sup> |
| Biopsy | X | | | | | | | | | | X | X |
| | STAGE 2 | | | | | | · | | | | | |
| PK Blood <sup>4</sup> | | | Х | | | | | | | | | |

Abbreviations: C = cycle; ctDNA = circulating tumor DNA; D = day; EOT = end of treatment; PK = pharmacokinetics.

<sup>&</sup>lt;sup>1</sup>To accommodate PK blood draws, patients should be instructed not to take their morning doses of both medications until told to do so in the clinic. A meal should be provided by the site when taking the medications in the clinic. Pre-dose PK sample should be collected prior to the administration of study drugs. Post-dose PK samples should be collected at the appropriate time points following administration of study drugs. PK samples should be drawn while patients are at steady state, which is 5 days, or 10 consecutive doses.

<sup>&</sup>lt;sup>2</sup>To be drawn at the time of the tumor biopsy.

<sup>&</sup>lt;sup>3</sup>Required blood draw at EOT. If optional biopsy is collected at EOT, ctDNA should be drawn at the time of the tumor biopsy.

<sup>&</sup>lt;sup>4</sup>Biopsies at screening and C3D1 (± 7 days) are required. When blood is being drawn at D3D1, site will provide a meal when study drugs are taken. An optional biopsy will be offered at the time when the decision to discontinue treatment is made (+ 7 days).



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

## 14.3 CTCAE v5.0 Grading for Laboratory Values

Table 8. Hematology Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Hematocrit | No | | |
| Hemoglobin | Yes | Blood and lymphatic<br>system disorders | Anemia |
| | | Investigations | Hemoglobin increased |
| Platelets | Yes | Investigations | Platelet count decreased |
| White blood cells | Yes | Investigations | White blood cell decreased |
| | | Blood and lymphatic system disorders | Leukocytosis |
| Neutrophils absolute | Yes | Investigations | Neutrophil count decreased |
| Lymphocytes absolute | Yes | Investigations | Lymphocyte count decreased |
| | | | Lymphocyte count increased |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 9. Coagulation Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|-----------|-----------------|----------------|-----------------|
| PT | No | | |
| INR | Yes | Investigations | INR increased |
| PTT | No | | |

<sup>†</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 10. Serum Chemistry Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Albumin | Yes | Metabolism and<br>nutrition disorders | Hypoalbuminemia |
| Alkaline phosphatase | Yes | Investigations | Alkaline phosphatase increased |
| ALT | Yes | Investigations | Alanine aminotransferase increased |
| AST | Yes | Investigations | Aspartate aminotransferase increased |
| Blood urea nitrogen | No | | |
| Uric acid | No | | |
| Chloride | No | | |
| Calcium | Yes | Metabolism and | Hypocalcemia |
| | | nutrition disorders | Hypocalcemia |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Creatinine | Yes | Investigations | Creatinine increased |
| Lactate Dehydrogenase | Yes | Investigations | Lactate Dehydrogenase increased |
| Glucose | Yes | Metabolism and | Hyperglycemia |
| | | nutrition disorders | Hypoglycemia |
| Potassium | Yes | Metabolism and | Hyperkalemia |
| | | nutrition disorders | Hypokalemia |
| Sodium | Yes | Metabolism and | Hypernatremia |
| | | nutrition disorders | Hyponatremia |
| Inorganic Phosphorus | No | | |
| Total bilirubin | Yes | Investigations | Blood bilirubin increased |
| Direct bilirubin | No | | |
| Total protein | No | | |
| Urea Nitrogen | No | | |
| Carbon Dioxide | No | | |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 11. Urinalysis Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Dipstick Evaluation Of<br>Bilirubin | No | | |
| Dipstick Evaluation Of<br>Blood | No | | |
| Dipstick Evaluation Of<br>Glucose | No | | |
| Dipstick Evaluation Of<br>Ketones | No | | |
| Dipstick Evaluation Of<br>Leukocytes | No | | |
| Dipstick Evaluation Of<br>Protein | No | | |
| Microscopic<br>Examination Of Casts | No | | |
| Microscopic<br>Examination Of Rbc | No | | |
| Microscopic<br>Examination Of Wbc | No | | |
| pH | No | | |
| Specific Gravity | No | | |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# **SPONSOR:**

# **BioMed Valley Discoveries**

## PROTOCOL NUMBER:

BVD-523-HCQ

# STATISTICAL ANALYSIS PLAN TFL SHELLS

| Author: | Julien Lucas |
|----------|--------------|
| Version: | 2.0 |
| Date: | 02-Sep-2024 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 1 Cover and signature pages

| Sponsor: | BioMed Valley Discoveries |
|---|---|
| Protocol Number: | BVD-523-HCQ |
| Study Title: | A phase 2 basket trial of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring MAPK pathway mutations (BVD-523-HCQ) |
| Document Version No | 1.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorize its approval.

#### Statistician

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|---|---|---|---|
| | Biostat III | | Signed by: Julium (mas Signer Name: Julien Lucas Signing Reason: I approve this document Signing Time: 09-Sep-2024 11:20 BST 1805EF259FF0471980A64D0037F8D5D3 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

### **Client Representative**

| Name | Title [text box when using eSignatures]: | Date | Signature |
|---|---|---|---|
| | Senior Scientist | | Signed by: Signer Name: Anna Groover Signing Reason: I approve this document Signing Time: 03-Sep-2024 08:40 CDT 71380BDD08BC4D289E63FA3831CD4243 |
| | President | | Signed by: Breat Kreider Signer Name: Brent Kreider Signing Reason: I approve this document Signing Time: 04-Sep-2024 08:58 PDT 9FC8BD6421864A9788CCD264914F8A6C |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# 2 Document History

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 27Jul2023 | 1.0 | David Manteigas | First SAP version |
| 20Aug2024 | 1.1 | Julien Lucas | Updated version to include required changes after the study was early terminated. |
| 02Sep2024 | 2.0 | Julien Lucas | Second SAP version. |

# 3 List of Tables, Figures and Listings

| TFL<br>Type | TFL<br>Number | Title Population | | SMC* | Included<br>in Final<br>Analysis |
|---|---|---|---|---|---|
| 14.1 | | Demographic Data | | | |
| Table | 14.1-1.1 | Patient Disposition | All Patients Set | Y | Y |
| Table | 14.1-1.2 | Number of Patients in the Analysis Sets | All Patients Set | | Υ |
| Table | 14.1-1.3 | Summary of Important Protocol Deviations | Full Analysis Set | | Υ |
| Table | 14.1-2.1 | Demographics and Baseline Characteristics | Full Analysis Set | Υ | Y |
| Table | 14.1-2.2 | Disease History | Full Analysis Set | Υ | Υ |
| Table | 14.1-2.3 | Summary of Medical History | Full Analysis Set | | Υ |
| Table | 14.1-2.4 | Summary of Concomitant Diseases | Full Analysis Set | | Y |
| Table | 14.1-3.1 | Prior Systemic Anti-Cancer Therapies | Full Analysis Set | Y | Υ |
| Table | 14.1-3.2 | Prior Radiotherapy Courses | Full Analysis Set | Y | Υ |
| Table | 14.1-3.3 | Prior Medications | Full Analysis Set | | Υ |
| Table | 14.1-3.4 | Concomitant Medications | Full Analysis Set | | Υ |
| Table | 14.1-4.1.1 | Treatment Exposure (Ulixertinib) | Full Analysis Set | Υ | Υ |
| Table | 14.1-4.1.2 | Treatment Exposure (Hydroxychloroquine) | Full Analysis Set | Υ | Υ |
| Table | 14.1-4.2.1 | Dosing Interruptions and Adjustments (Ulixertinib) | Full Analysis Set | Υ | Υ |
| Table | 14.1-4.2.2 | Dosing Interruptions and Adjustments | Full Analysis Set | Υ | Υ |
| | | (Hydroxychloroquine) | | | |
| 14.2 | | Efficacy Data | | | |
| Table | 14.2-1.1.1 | Best Overall Response and Overall Response Rate | Full Analysis Set | | Υ |
| Table | 14.2-1.1.2 | Best Overall Response and Overall Response Rate | Evaluable Analysis Set | | |
| Table | 14.2-1.2.1 | Overall, Target and Non-Target Lesion Response | Full Analysis Set | | Υ |
| Table | 14.2-1.2.2 | Overall, Target and Non-Target Lesion Response | Evaluable Analysis Set | | |
| Table | 14.2-1.3.1 | Incidence of New Lesions | Full Analysis Set | | Υ |
| Table | 14.2-1.3.2 | Incidence of New Lesions | Evaluable Analysis Set | | |
| Table | 14.2-1.4.1 | Progression-free Survival (PFS) | Full Analysis Set | | Υ |
| Table | 14.2-1.4.2 | Progression-free Survival (PFS) | Evaluable Analysis Set | | |
| Table | 14.2-1.5.1 | Overall Survival (OS) | Full Analysis Set | | Υ |
| Table | 14.2-1.5.2 | Overall Survival (OS) | Evaluable Analysis Set | | |
| Table | 14.2-1.6.1 | Duration of Response (DOR) | Full Analysis Set | | |
| 14.3 | | Safety Data | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

| Table | 14.3-1.1 | Overview Summary of Treatment-Emergent Adverse Events | Full Analysis Set | Y | Y |
|---|---|---|---|---|---|
| Table | 14.3-1.2 | Summary of Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term | Full Analysis Set | Υ | Υ |
| Table | 14.3-1.3 | Summary of Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | Full Analysis Set | Υ | Υ |
| Table | 14.3-1.4 | Summary of Serious Treatment-Emergent Adverse<br>Events by System Organ Class and Preferred Term | Full Analysis Set | Y | Υ |
| Table | 14.3-1.5 | Summary of Related Serious Treatment-Emergent<br>Adverse Events by System Organ Class and Preferred<br>Term | Full Analysis Set | Y | Υ |
| Table | 14.3-1.6 | Summary of Treatment-Emergent Adverse Events by<br>Preferred Term | Full Analysis Set | | |
| Table | <u>14.3-1.7</u> | Summary of Related Treatment-emergent Adverse<br>Events by Preferred Term | Full Analysis Set | | |
| Table | 14.3-1.8 | Summary of Serious Treatment-emergent Adverse<br>Events by Preferred Term | Full Analysis Set | | |
| Table | 14.3-1.9 | Summary of Related Serious Treatment-emergent<br>Adverse Events by Preferred Term | Full Analysis Set | | |
| Table | 14.3-1.10 | Summary of Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term for Maximum<br>CTCAE grade | Full Analysis Set | | Y |
| Table | 14.3-1.11 | Summary of Related Treatment-Emergent Adverse<br>Events by System Organ Class and Preferred Term for<br>Maximum CTCAE grade | Full Analysis Set | Y | Y |
| Table | 14.3-1.12 | Summary of Treatment-emergent Adverse Leading to<br>Treatment Discontinuation Events by System Organ<br>Class and Preferred Term | Full Analysis Set | Y | Y |
| Table | 14.3-1.13 | Summary of Related Treatment-emergent Adverse Events Leading to Treatment Discontinuation by System Organ Class and Preferred Term | Full Analysis Set | Y | Y |
| Table | 14.3-1.14 | Summary of Treatment-emergent Adverse Events Leading to Treatment Discontinuation within Cycle 1 by System Organ Class and Preferred Term | Full Analysis Set | Y | Y |
| Table | 14.3-1.15 | Summary of Related Treatment-emergent Adverse Events Leading to Treatment Discontinuation within Cycle 1 by System Organ Class and Preferred Term | Full Analysis Set | Y | Υ |
| Table | 14.3-1.16 | Summary of Treatment-emergent Adverse Events Leading to Treatment Discontinuation following Cycle 1 by System Organ Class and Preferred Term | Full Analysis Set | Y | Υ |
| Table | 14.3-1.17 | Summary of Related Treatment-emergent Adverse Events Leading to Treatment Discontinuation following Cycle 1 by System Organ Class and Preferred Term | Full Analysis Set | Y | Y |
| Table | 14.3-1.18 | Summary of Treatment-emergent Adverse Events Leading to Treatment Interruption by System Organ Class and Preferred Term | Full Analysis Set | | Y |
| Table | 14.3-1.19 | Summary of Related Treatment-emergent Adverse<br>Events Leading to Treatment Interruption by System<br>Organ Class and Preferred Term | Full Analysis Set | | Y |
| Table | 14.3-1.20 | Summary of Treatment-emergent Adverse Events Leading to Treatment Interruption within Cycle 1 by System Organ Class and Preferred Term | Full Analysis Set | Y | Y |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

| Table | 14.3-1.21 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | Y | Y |
|---|---|---|---|---|---|
| | | Events Leading to Treatment Interruption within Cycle | | | |
| | | 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.22 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Treatment Interruption following Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.23 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Treatment Interruption following | | | |
| | | Cycle 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.24 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | | Υ |
| | | Leading to Dose Reduction by System Organ Class and | | | |
| | | Preferred Term | | | |
| Table | 14.3-1.25 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Dose Reduction by System Organ | | | |
| | | Class and Preferred Term | | | |
| Table | 14.3-1.26 | Summary of Treatment-Emergent Adverse Events | Full Analysis Set | Υ | Υ |
| | | Leading to Dose Reduction within Cycle 1 by System | | | |
| | | Organ Class and Preferred Term | | | |
| Table | 14.3-1.27 | Summary of Related Treatment-Emergent Adverse | Full Analysis Set | γ | Y |
| | | Events Leading to Dose Reduction within Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.28 | Summary of Treatment-Emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Dose Reduction following Cycle 1 by System | | | ' |
| | | Organ Class and Preferred Term | | | |
| Table | 14.3-1.29 | Summary of Related Treatment-Emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Dose Reduction following Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.30 | Summary of Treatment-emergent Adverse Events by | Full Analysis Set | | Y |
| , abic | 11.0 1.00 | System Organ Class and Preferred Term Leading to | T dill 7 illuly 515 oct | | 1. |
| | | Death | | | |
| Table | 14.3-1.31 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| Tubic | 14.0 1.01 | Events by System Organ Class and Preferred Term | Tuli Allulysis occ | | 1. |
| | | Leading to Death | | | |
| Table | 14.3-1.32 | Summary of Deaths | All Patients Set | Y | Y |
| Table | 14.3-2.1 | Summary and Change from Baseline in Hematology | Full Analysis Set | - ' | Y |
| Table | 14.5-2.1 | Laboratory Results by Visit | ruii Anaiysis set | | ' |
| Table | 142221 | Gradable Hematology Laboratory Results – Worst On- | Full Analysis Set | _ | |
| Table | 14.3-2.2.1 | | ruii Anaiysis set | | |
| Table | 142222 | treatment Value by Cycle | Full Applysis Cot | | |
| Table | 14.3-2.2.2 | Non-gradable Hematology Laboratory Results – Worst | Full Analysis Set | | |
| Table | 142221 | On-treatment Value by Cycle | Full Application Code | v | v |
| Table | 14.3-2.3.1 | Shift Table of Gradable Hematology Laboratory Results | Full Analysis Set | Y | Y |
| | | Baseline vs Worst On-treatment Value | | _ | |
| Table | 14.3-2.3.2 | Shift Table of Non-gradable Hematology Laboratory | Full Analysis Set | | Y |
| | | Results – Baseline vs Worst On-treatment Value | | | |
| Table | 14.3-2.4 | Summary and Change from Baseline in Biochemistry | Full Analysis Set | | Y |
| | | Laboratory Results by Visit | | | |
| Table | 14.3-2.5.1 | Gradable Biochemistry Laboratory Results – Worst On- | Full Analysis Set | | |
| | | treatment Value by Cycle | | | |
| Table | 14.3-2.5.2 | Non-gradable Biochemistry Laboratory Results – | Full Analysis Set | | |
| | | Worst On-treatment Value by Cycle | | | |
| Table | 14.3-2.6.1 | Shift Table of Gradable Biochemistry Laboratory | Full Analysis Set | Υ | Y |
| | | Results – Baseline vs Worst On-treatment Value | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

| | | | <u> </u> | T |
|---|---|---|---|---|
| 14.3-2.6.2 | Shift Table of Non-gradable Biochemistry Laboratory<br>Results — Baseline vs Worst On-treatment Value | Full Analysis Set | | Y |
| 14.3-2.7 | Summary at Baseline in Coagulation Laboratory<br>Results by Visit | Full Analysis Set | | Y |
| 14.3-2.8 | Summary at Baseline in Urinalysis Laboratory Results by Visit | Full Analysis Set | | |
| 14.3-3.1 | Summary and Change from Baseline in Vital Signs by | Full Analysis Set | | Υ |
| 14.3-3.2 | Shift table of Vital Signs – Baseline vs worst on-<br>treatment value | Full Analysis Set | | Y |
| 14.3-3.3 | Summary and Change from Baseline in ECG parameters by Visit | Full Analysis Set | Υ | Υ |
| 14.3-3.4 | Summary of ECHO at Baseline | Full Analysis Set | | |
| 14.3-3.5 | Summary of Physical Examination at Baseline | Full Analysis Set | | |
| | | • | Υ | |
| | Pharmacokinetic Data | | | |
| 14.5-1.1 | Pharmacokinetic Concentration Data | PK Analysis Set | | Υ |
| | | <del>'</del> | | Υ |
| 21.5 2.2 | | | | <u> </u> |
| 14 2-1 1 | | Full Analysis Set | γ | Υ |
| 14.2-1.2.1 | Spider plot of Percentage Change from Baseline in | Full Analysis Set | | Y |
| 14.2-1.2.2 | Spider plot of Percentage Change from Baseline in | Evaluable Analysis Set | | |
| 14.2-1.3.1 | Waterfall plot of Maximum Percentage Change from<br>Baseline in Sum of Longest Diameter | Full Analysis Set | | Y |
| 14.2-1.3.2 | Waterfall plot of Maximum Percentage Change from<br>Baseline in Sum of Longest Diameter | Evaluable Analysis Set | | |
| 14.2-1.4.1 | Swimmer Plot of Response Assessments | Full Analysis Set | | Υ |
| 14.2-1.4.2 | Swimmer Plot of Response Assessments | Evaluable Analysis Set | | |
| 14.2-1.5.1 | Kaplan-Meier Estimate for Progression-free Survival (PFS) | Full Analysis Set | | Υ |
| 14.2-1.5.2 | Kaplan-Meier Estimate for Progression-free Survival (PFS) | Evaluable Analysis Set | | |
| 14.2-1.6.1 | Kaplan-Meier Estimate for Overall Survival (OS) | Full Analysis Set | | Υ |
| 14.2-1.6.2 | Kaplan-Meier Estimate for Overall Survival (OS) | Evaluable Analysis Set | | |
| 14.2-1.7.1 | Kaplan-Meier Estimate for Duration of Response<br>(DOR) | Full Analysis Set | | |
| | Patient Data Listings | | | |
| | Patient Disposition | | | |
| 16.2.1-1 | Patient Informed Consent | All Patients Set | | Υ |
| 16.2.1-2 | Failed Inclusion and Exclusion Criteria | All Patients Set | | Υ |
| 16.2.1-3 | Patient Disposition | All Patients Set | | Υ |
| | Analysis Sets | | | |
| 16.2.2-1 | Analysis Sets | All Patients Set | | |
| | Protocol Deviations | | | |
| | Destacel Deviations | Full Applysis Cot | | Υ |
| 16.2.3-1 | Protocol Deviations | ruli Alialysis set | | |
| <u>16.2.3-1</u> | | ruii Ariaiysis set | | ' |
| 16.2.4-1 | Demographic Data Demographics and Baseline Characteristics | Full Analysis Set | | Y |
| | 14.3-2.8 14.3-3.1 14.3-3.2 14.3-3.3 14.3-3.4 14.3-3.5 14.3-3.6 14.5-1.1 14.5-1.2 14.2-1.2.1 14.2-1.2.1 14.2-1.3.1 14.2-1.3.2 14.2-1.5.1 14.2-1.5.1 14.2-1.5.1 14.2-1.5.2 14.2-1.5.1 14.2-1.5.2 | Results – Baseline vs Worst On-treatment Value 14.3-2.7 Summary at Baseline in Coagulation Laboratory Results by Visit 14.3-2.8 Summary at Baseline in Urinalysis Laboratory Results by Visit 14.3-3.1 Summary and Change from Baseline in Vital Signs by Visit 14.3-3.2 Shift table of Vital Signs – Baseline vs worst on- treatment value 14.3-3.3 Summary and Change from Baseline in ECG parameters by Visit 14.3-3.4 Summary of ECHO at Baseline 14.3-3.5 Summary of Physical Examination at Baseline 14.3-3.6 Summary of ECOG Performance Status by Visit Other Efficacy Data Pharmacokinetic Data 14.5-1.1 Pharmacokinetic Concentration Data 14.5-1.2 Pharmacokinetic Parameters Data Figures 14.2-1.1 Consort Diagram 14.2-1.2.1 Spider plot of Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.3.1 Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.3.2 Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.4.1 Swimmer Plot of Response Assessments 14.2-1.4.2 Swimmer Plot of Response Assessments 14.2-1.5.1 Kaplan-Meier Estimate for Progression-free Survival (PFS) 14.2-1.5.2 Kaplan-Meier Estimate for Progression-free Survival (PFS) 14.2-1.6.1 Kaplan-Meier Estimate for Overall Survival (OS) 14.2-1.6.2 Kaplan-Meier Estimate for Overall Survival (OS) 14.2-1.6.3 Failed Inclusion and Exclusion Criteria 16.2.1-1 Patient Informed Consent 16.2.1-1 Patient Disposition | Results – Baseline vs Worst On-treatment Value 14.3-2.7 Summary at Baseline in Coagulation Laboratory Results by Visit 14.3-2.8 Summary at Baseline in Urinalysis Laboratory Results by Visit 14.3-3.1 Summary and Change from Baseline in Vital Signs by Visit 14.3-3.2 Shift table of Vital Signs – Baseline vs worst on- treatment value 14.3-3.3 Summary and Change from Baseline in ECG parameters by Visit 14.3-3.4 Summary of ECHO at Baseline 14.3-3.4 Summary of ECHO at Baseline 14.3-3.5 Summary of Physical Examination at Baseline 14.3-3.6 Summary of ECHO at Baseline Pharmacokinetic Data Other Efficacy Data Pharmacokinetic Concentration Data Pharmacokinetic Parameters Data 14.5-1.1 Pharmacokinetic Parameters Data Data Data Data Data Data Data Dat | Results - Baseline vs Worst On-treatment Value 14.3-2.7 Summary at Baseline in Coagulation Laboratory Results by Visit 14.3-2.8 Summary at Baseline in Urinalysis Laboratory Results by Visit 14.3-3.1 Summary and Change from Baseline in Vital Signs by Visit 14.3-3.2 Shift table of Vital Signs - Baseline vs worst on- treatment value 14.3-3.3 Summary and Change from Baseline in ECG parameters by Visit 14.3-3.4 Summary and Change from Baseline in ECG parameters by Visit 14.3-3.5 Summary of ECHO at Baseline 14.3-3.5 Summary of ECOG performance Status by Visit 14.3-3.6 Summary of ECOG Performance Status by Visit 14.3-3.6 Summary of ECOG Performance Status by Visit 14.3-3.6 Summary of ECOG Performance Status by Visit 14.3-3.6 Other Efficacy Data Pharmacokinetic Data Pharmacokinetic Data 14.5-1.1 Pharmacokinetic Concentration Data Pharmacokinetic Concentration Data Pharmacokinetic Concentration Data Pharmacokinetic Concentration Data Pharmacokinetic Concentration Data PK Analysis Set Figures 14.2-1.2 Spider plot of Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.3.1 Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.3.2 Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter 14.2-1.4 Swimmer Plot of Response Assessments Paseline in Sum of Longest Diameter 14.2-1.4.1 Swimmer Plot of Response Assessments Full Analysis Set 14.2-1.5 (Raplan-Meier Estimate for Progression-free Survival Full Analysis Set 14.2-1.5 (Raplan-Meier Estimate for Overall Survival (OS) Patient Disposition Patient Data Listings Patient Disposition All Patients Set Protocol Deviations |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

| Listing | 16.2.4-3 | Disease History | Full Analysis Set | Y |
|---|---|---|---|---|
| Listing | 16.2.4-4 | Medical History and Concomitant Diseases | Full Analysis Set | Υ |
| Listing | 16.2.4-5 | Prior Systemic Anti-Cancer Therapies | Full Analysis Set | Υ |
| Listing | 16.2.4-6 | Prior Radiotherapy Courses | Full Analysis Set | Υ |
| Listing | 16.2.4-7 | Prior and Concomitant Medications | Full Analysis Set | Υ |
| Listing | 16.2.4-8 | On Treatment Radiation | Full Analysis Set | |
| Listing | 16.2.4-9 | On Treatment Surgery and Medical Procedures | Full Analysis Set | |
| Listing | 16.2.4-10 | On Treatment Blood Transfusions | Full Analysis Set | |
| Listing | 16.2.4-11 | NGS Data | Full Analysis Set | Y |
| 16.2.5 | | Compliance and/or Drug Concentration Data | | |
| Listing | 16.2.5-1 | Ulixertinib In-clinic Administration | Full Analysis Set | |
| Listing | 16.2.5-2 | Hydroxychloroquine In-clinic Administration | Full Analysis Set | |
| Listing | 16.2.5-3 | Ulixertinib Interruptions and Adjustments | Full Analysis Set | Y |
| Listing | 16.2.5-4 | Hydroxychloroquine Interruptions and Adjustments | Full Analysis Set | Y |
| Listing | 16.2.5-5 | Ulixertinib Exposure | Full Analysis Set | Y |
| Listing | 16.2.5-6 | Hydroxychloroquine Exposure | Full Analysis Set | Y |
| Listing | 16.2.5-7 | Ulixertinib Dispensed | Full Analysis Set | |
| Listing | 16.2.5-8 | Hydroxychloroquine Dispensed | Full Analysis Set | |
| Listing | 16.2.5-9 | Ulixertinib Returned | Full Analysis Set | |
| Listing | 16.2.5-10 | Hydroxychloroquine Returned | Full Analysis Set | |
| 16.2.6 | | Individual Efficacy Response data | | |
| Listing | 16.2.6-1 | Target Lesions | Full Analysis Set | Υ |
| Listing | 16.2.6-2 | Non-Target Lesions | Full Analysis Set | Υ |
| Listing | 16.2.6-3 | New Lesions | Full Analysis Set | Υ |
| Listing | 16.2.6-4 | Overall Response | Full Analysis Set | Y |
| Listing | 16.2.6-5 | Progression-Free Survival (PFS | Full Analysis Set | Υ |
| Listing | 16.2.6-6 | Survival Status | Full Analysis Set | Υ |
| Listing | 16.2.6-7 | Duration of Response (DOR) | Full Analysis Set | |
| 16.2.7 | | Adverse Events | Full Analysis Set | |
| Listing | 16.2.7-1 | Adverse Events | All Patients Set | Y |
| Listing | 16.2.7-2 | Treatment Emergent Adverse Events | Full Analysis Set | Y |
| Listing | 16.2.7-3 | Serious Adverse Events | Full Analysis Set | Y |
| Listing | 16.2.7-4 | Deaths | All Patients Set | Y |
| 16.2.8 | | Laboratory Data | | |
| Listing | 16.2.8-1 | Hematology | Full Analysis Set | Y |
| Listing | 16.2.8-2 | Biochemistry | Full Analysis Set | Y |
| Listing | 16.2.8-3 | Coagulation | Full Analysis Set | Y |
| Listing | 16.2.8-4 | Urinalysis | Full Analysis Set | Y |
| Listing | 16.2.8-5 | Tumor Markers | Full Analysis Set | |
| Listing | 16.2.8-6 | Pregnancy | Full Analysis Set | |
| 16.2.9 | | Other Safety Data | | |
| Listing | 16.2.9-1 | Vital Signs | Full Analysis Set | Y |
| Listing | <u>16.2.9-2</u> | Electrocardiogram | Full Analysis Set | Υ |
| Listing | <u>16.2.9-3</u> | ECHO/MUGA | Full Analysis Set | Y |
| Listing | 16.2.9-4 | Physical Examination | Full Analysis Set | Υ |
| Listing | 16.2.9-5 | Ophthalmology exam | Full Analysis Set | Υ |
| Listing | 16.2.9-6 | ECOG Performance Status | Full Analysis Set | Υ |
| 16.2.11 | | Pharmacokinetic Data | | |
| Listing | 16.2.11-1 | Pharmacokinetic Concentration Data | PK Analysis Set | Y |
| Listing | 16.2.11-2 | Pharmacokinetic Parameters Data | PK Analysis Set | Υ |
| Listing | | Pharmacokinetic Concentration Data | , | |

<sup>\*</sup>Table, Figure or Listing that will be used for SMC purposes. Y=Yes



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 4 General programming notes

All tables will be reported by treatment Basket.

An 'Overall' column will be included in all tables.

| Column headers | | | | | |
|----------------|----------|----------|----------|----------|---------|
| Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |

For tables reporting data on All Patients Set, a screening failures column will be added.

The full-page header to be included for each delivery is indicated in the table below:

| Delivery | Туре | Page Header |
|----------------|---------|-------------|
| Dry run | Dry run | Dry-run |
| SMC N* | Final | Final |
| Final analysis | Draft | Draft |
| | Final | Final |

<sup>\*</sup>N references to the SMC chronological number

For the listings, all cases where 'Other' is present, please present the respective 'Other' specification.

All Listings will be sorted by Basket and patient ID. A programming note will be added to each Listing when another variable is needed to make the sorting meaningful (e.g., assessment date).



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.1 - Patient Disposition
All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients enrolled [a] | xx | XX | XX | XX | XX | XX | XX |
| Patients completed screening [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued from screening [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary reason for discontinuation [c] | | | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Screen Failure | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Technical Problems | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients rescreened [b] | | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients eligible for inclusion in the study [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Patients treated with study drug [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

<sup>[</sup>a] Patients who signed the informed consent.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


Template Author: Andra Rusu Version 5.0 25Jun2020 

<sup>[</sup>b] Percentages are calculated from the number of patients enrolled.

<sup>[</sup>c] Percentages are calculated from the number of patients who discontinued from screening.

<sup>[</sup>d] Percentages are calculated from the number of patients who were treated with study drug.

<sup>[</sup>e] Percentages are calculated from the number of patients who discontinued from treatment.

<sup>[</sup>f] Percentages are calculated from the number of patients who discontinued from study.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-1.1 - Patient Disposition All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients completed treatment [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Discontinued from treatment [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Primary reason for discontinuation [e] | | | | | | | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

<sup>[</sup>a] Patients who signed the informed consent.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>[</sup>b] Percentages are calculated from the number of patients enrolled.

<sup>[</sup>c] Percentages are calculated from the number of patients who discontinued from screening.

<sup>[</sup>d] Percentages are calculated from the number of patients who were treated with study drug.

<sup>[</sup>e] Percentages are calculated from the number of patients who discontinued from treatment.

<sup>[</sup>f] Percentages are calculated from the number of patients who discontinued from study.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.1 - Patient Disposition
All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients completed study [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Primary reason for completion [f] | | | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Sponsor Request | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol-Specified Withdrawal Criterion Met | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

- [a] Patients who signed the informed consent.
- [b] Percentages are calculated from the number of patients enrolled.
- [c] Percentages are calculated from the number of patients who discontinued from screening.
- [d] Percentages are calculated from the number of patients who were treated with study drug.
- [e] Percentages are calculated from the number of patients who discontinued from treatment.
- [f] Percentages are calculated from the number of patients who completed the study.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


#### PROGRAMMING NOTES:

• Display all possible reasons, either reported for at least one patient or not.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.2 - Number of Patients in the Analysis Sets
All Patients Set


| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| All Patients Set [a] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Full Analysis Set [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Stage 1 Analysis Set [c] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Evaluable Analysis Set [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| PK Analysis Set [e] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

- [a] Patients who were enrolled regardless of whether they received the study drug or not.
- [b] Patients who received at least 1 dose of the study drug.
- [c] First 13 patients who have completed at least one cycle of therapy and who have received a minimum of 75% of prescribed study therapy during Cycle 1
- [d] Patients who received at least one dose of study drug and have at least one post-treatment study evaluation or who have discontinued therapy prior to the first post-treatment study evaluation due to clinical progressive disease or drug-related adverse events.
- [e] Patients who received at least one dose of study medication and have at least one post dose PK measurement.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.3 - Summary of Important Protocol Deviations Full Analysis Set Page 1 of Y

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Number of patients with at least one important protocol deviation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Deviation category 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *************************************** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Deviation category 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: A patient with multiple occurences of a protocol deviation is counted only once in this deviation category/summary term.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Categories / Summary terms to match the PDCF.
- Present only important protocol deviations with at least one occurrence (where classification=Important).




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Age (Years) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XXX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| Age category (Years) n (%) | | | | | | |
| 18 - 64 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 65 - 84 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| >=85 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Gender - n (%) | | | | | | |
| Female<br>Childbearing potential n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Male | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reproductive potential n (%) Yes | VU /VU V\ | VV /VV V\ | עט עטן טט | 00 /00 01 | 00 (00 0) | יט יטט טו |
| No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


BMSOP111/F2


<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set Page 2 of Y

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Race - n (%) | | | | | | |
| American Indian or | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Alaska Native | | | | | | |
| Asian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pacific Islander | | | | | | |
| White | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Ethnicity - n (%) | | | | | | |
| Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Weight (kg) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set Page 3 of Y

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Height (cm) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| ECOG performance at Baseline (%) [b] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Smoking History - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Current | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Former | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


<sup>[</sup>b] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Gene/Codon/Amino acid change<br>HRAS/G469/Alanine A | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) |
| KRAS/G469/Arginine R | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) |
| NRAS/G469/Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.doc)


BMSOP111/F2


<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.2 - Disease History Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| ancer Diagnosis - n (%) | | | | | | |
| Intrahepatic cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Perihilar cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Extrahepatic cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pancreatic adenocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ime since initial diagnosis<br>onths) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.XX (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| isease stage at enrollment - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | | | - | | |

[a] Calculated as (date of first dose of study treatment - date of diagnosis) / 30.4375.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Table 14.1-2.2 - Disease History Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Disease stage at initial | | | | | | |
| diagnosis - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Method of diagnosis - n (%) | | | | | | |
| Cytological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Histological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Prior Radiation Therapies - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | | | | | | |

[a] Calculated as (date of first dose of study treatment - date of diagnosis) / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-2.3 - Summary of Medical History Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any relevant medical history | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ********** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>.

If there is more than one medical history within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one medical history within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within primary SOC.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.4 - Summary of Concomitant Diseases Full Analysis Set Page 1 of Y

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any relevant concomitant disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ********** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ************ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>.

If there is more than one concomitant disease within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one concomitant disease within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within primary SOC.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

able 14 1-3 1 - Drior Systemic Anti-Cancer Theranies

Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Received at least one systemic prior anti-cancer Therapy - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lines of systemic prior anti-cancer therapies - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mean (SD) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Most recent therapy before study treatment start Regimen name - n (%) | | | | | | |
| xxxxxxx | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXXXXXX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| xxxxxxx | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies
Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Best Response - n (%) | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Duration of therapy (months) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Time since Best Overall Response | | | | | | |
| (months) [b] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.


Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)

<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Time since Relapse/Progression | | | | | | |
| (months) [c] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Reason for discontinuation - n (%) | | | | | | |
| Intolerance | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lack of Efficacy (incl. PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed Therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-3.2 - Prior Radiotherapy Courses Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Received at least one prior<br>radiotherapy - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total number of prior radiotherapy courses - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Site of prior radiotherapy - n (%) [a] | | | | | | |
| Abdominal Cavity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adrenal Gland | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Most recent prior radiotherapy before study | | | | | | |
| treatment start | | | | | | |
| Site of prior radiotherapy - n (%) | | | | | | |
| Abdominal Cavity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Duration of therapy (months) [b] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | (XX.XX) | (XX.XX) | (XX.XX) | (XX.XX) | (XX.XX) | (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

<sup>[</sup>a] Patients can have more than 1 site of prior radiotherapy if they had multiple prior radiotherapies.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-3.3 - Prior Medications Full Analysis Set

| ATC Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any Prior Medications | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: WHOHD-B3 <vx.x>. ATC=Anatomical Therapeutic Chemical.

If there is more than one medication within an ATC class, the patient is counted only once under that ATC class. If there is more than one medication within an ATC class and preferred term (PT), the patient is counted only once in that ATC class and PT.

ATC classes are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within ATC class.

Prior medication is defined as any medications whose end date is before the first study treatment date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.1-3.4 - Concomitant Medications Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.1-3.3
- Present concomitant medications.
- Replace footnote 'Prior medication is defined as...' with the following footnote:
   (Concomitant medication is defined as any medication ongoing at first day of study drug or started after first day of study drug up to the end of the ontreatment period.'




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.1.1 - Treatment exposure (Ulixertinib) Full Analysis Set

| | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Number of cycles received | | | | | | |
| [a] - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | , | | , | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| Duration of exposure to | | | | | | |
| ulixertinib (months) [b] - n | | | | | | |
| (%) | | | | | | |
| < 1 month | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1-2 months | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2-3 months | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

<sup>[</sup>a] Number of cycles received = Number of cycles where the patient received at least one dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


BMSOP111/F2


<sup>[</sup>b] Duration of exposure (months) = [(Date of last known treatment dosing with drug - date of initial dosing with drug) + 1] / 30.4375.

<sup>[</sup>c] Actual cumulative dose received (mg) = Sum of [(Stop date - Start date for each time period reported in the dairy) x Dose].

<sup>[</sup>d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days). Filename: (Specify file name.rtf)


Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.1.1 - Treatment exposure (Ulixertinib) Full Analysis Set


| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Actual cumulative dose on | | | | | | |
| llixertinib (mg) [c] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| Relative dose intensity [d] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

<sup>[</sup>a] Number of cycles received = Number of cycles where the patient received at least one dose.

BMSOP111/F2

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


<sup>[</sup>b] Duration of exposure (months) = [(Date of last known treatment dosing with drug - date of initial dosing with drug) + 1] / 30.4375.

<sup>[</sup>c] Actual cumulative dose received (mg) = Sum of [(Stop date - Start date for each time period reported in the dairy) x Dose].

<sup>[</sup>d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days). Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.1-4.1.2 - Treatment exposure (Hydroxychloroquine) Full Analysis Set

# PROGRAMMING NOTES:

• Repeat Table 14.1-4.1.1



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.2.1 - Dosing Interruptions and Adjustments (Ulixertinib) Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| At least one dose adjustment - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason dose changed - n (%) [a] Adverse event Parental/Guardian decision | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Consent withdrawal | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Other | | | , | • | • | |
| Dose changed to - n (%) [b]<br>150mg<br>300mg | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 450mg | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| At least one dose interruption - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason dose interrupted [a] | | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dispensing Error | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Investigator Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Consent Withdrawal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patient Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] A patient can be counted under several reasons if they had multiple different dose changes/interruptions.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


<sup>[</sup>b] A patient can be counted under more than one dose level if they had multiple different dose changes.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.1-4.2.2 - Dosing Interruptions and Adjustments (Hydroxychloroquine) Full Analysis Set

# PROGRAMMING NOTES:

• Repeat Table 14.1-4.2.1




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.2-1.1.1 - Best Overall Response and Overall Response Rate Full Analysis Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Best overall response - n (%) [a] | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| overall response rate (CR+PR) - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 95 % CI for Overall response rate | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Disease control rate (CR+PR+SD) - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 95 % CI for Disease Control rate | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Non-responders (SD+PD+NE) - n (%) [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable , CI=Confidence Interval.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


<sup>95%</sup> CI is estimated using the Clopper-Pearson method.

<sup>[</sup>a] Confirmed Best overall response as per RECIST 1.1

<sup>[</sup>b] Non responders: Patients without a confirmed response or a missing baseline/screening tumor assessment will be considered non-responders



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.2-1.1.2 - Best Overall Response and Overall Response Rate
Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.2-1.1.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.2-1.2.1 - Overall, Target and Non-Target Lesion Response Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| C3D1 | | | | | | |
| Target Lesion Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Target Lesion Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Complete Response/Non | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | | | | | | |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Applicable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Overall Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Programming Note: Repeat for all | | | | | | |
| available assessments | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.2-1.2.2 - Overall, Target and Non-Target Lesion Response
Evaluable Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.2-1.2.1
- Present data on Evaluable AnalysisSet.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.2-1.3.1 - Incidence of New Lesions Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3D1 | | | | | | |
| New Lesions - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of New Lesions - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.3.2 - Incidence of New Lesions Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.3.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.2-1.4.1 - Progression-Free Survival (PFS)
Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with events - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PFS (months) [a] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| KM probability estimates for PFS (95% | | | | | | |
| CI) [b] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |

Note: CI=Confidence Interval.

Progression-Free Survival (PFS) is the time from the first ulixertinib dose dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

- [a] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [b] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)

<sup>\*</sup> Censored observation at maximum value.



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.4.2 - Progression-Free Survival (PFS) Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.4.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Table 14.2-1.5.1 - Overall Survival (OS) Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with events - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| OS (months) [a] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| OM probability estimates for PFS (95% | | | | | | |
| (I) [b] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |

Note: CI=Confidence Interval.

Overall Survival is defined as the time from first treatment to death.

- [a] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [b] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


<sup>\*</sup> Censored observation at maximum value.



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.5.2 - Overall Survival (OS) Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.4.1
- Present data on Evaluable Analysis Set.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.2-1.6.1 - Duration of Response Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with response (CR+PR) | XX | XX | XX | XX | XX | XX |
| Patients with events - n (%) [a] Patients censored - n (%) [a] | XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| DOR (months) [b] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| KM probability estimates for PFS (95% CI) [c] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |

Note: CI=Confidence Interval, CR=Complete Response, PR=Partial Response.

Duration of response is the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause. +1

- [a] Percentage calculated on patients with response. Events are death or disease progression.
- [b] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [c] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>\*</sup> Censored observation at maximum value.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.1 - Overview Summary of Treatment-Emergent Adverse Events Full Analysis Set Page 1 of Y

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0) |
| Number of patients with: | | | | | | |
| Any TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to Both | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to Uli. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to HCQ. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any SAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related SAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation within 1 cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation within 1 cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation following 1 cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| following 1 cycle | | | | | | |
| Any TEAE leading to treatment interruption | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment interruption | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment interruption within 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| cycle | | | | | | |
| Any Related TEAE leading to treatment interruption within 1 cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment interruption following l cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment interruption following 1 cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: SAE=Serious Adverse Events, TEAE=Treatment-Emergent Adverse Events

Note 2: Any related TEAE includes TEAEs that are considered related to either hydroxychloroquine or ulixertinib.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


# Table 14.3-1.1 - Overview Summary of Treatment-Emergent Adverse Events

## Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Number of patients with: | | | | | | |
| Any TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any related TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to dose reduction within | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 1 | | | | | | |
| Any Related TEAE leading to dose reduction within Cycle 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to dose reduction following Cycle 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to dose reduction following Cycle 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE with Grade >= 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE with Grade >= 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: SAE=Serious Adverse Events, TEAE=Treatment-Emergent Adverse Events

Note 2: Any related TEAE includes TEAEs that are considered related to either hydroxychloroquine or ulixertinib.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

# Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

"Related TEAE to Both", "Related TEAE to Uli." and "Related TEAE to HCQ." will be presented for all treatment-related adverse events [...]" in the above table.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.2 - Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *************************************** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within each SOC.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.3 - Summary of Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term
Full Analysis Set


| System<br>Organ<br>Class<br>Preferred<br>Term | | Basket 1<br>N=XX<br>n (%) | | | Basket 2<br>N=XX<br>n (%) | ! | | Basket 3<br>N=XX<br>n (%) | | | Basket 4<br>N=XX<br>n (%) | | | Basket 5<br>N=XX<br>n (%) | | | Overall<br>N=XX<br>n (%) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ |
| Any<br>related<br>TEAE | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) | XX<br>(XX.X) |
| System<br>organ<br>class 1 | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) |
| Preferred<br>term 1 | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) |
| Preferred<br>term 2 | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

Note 2: Both = TEAE related to both treatments, Uli = TEAE related to ulixertinib, HCQ = TEAE related to Hydroxychloriquine.

Related TEAE: TEAEs with causality=Related, Possibly Related or missing.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within each SOC.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.4 - Summary of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.2
- Present Serious TEAE: TEAEs with SAE =" Yes".
- Add footnote:

"Serious TEAE: TEAEs with SAE =" Yes"."

Table 14.3-1.5 - Summary of Related Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Present Related Serious TEAE: SAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"SAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Table 14.3-1.6 - Summary of Treatment-Emergent Adverse Events by Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1<br>Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a preferred term (PT), the patient is counted only once in that PT.

PTs are sorted in descending order of frequency for the overall Basket.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.3-1.7 - Summary of Related Treatment-emergent Adverse Events by Preferred Term Full Analysis Set

| Preferred<br>Term | | Basket 1<br>N=XX<br>n (%) | | | Basket 2<br>N=XX<br>n (%) | ! | | Basket 3<br>N=XX<br>n (%) | | | Basket 4<br>N=XX<br>n (%) | ı | | Basket 5<br>N=XX<br>n (%) | | | Overall<br>N=XX<br>n (%) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ |
| Any<br>related<br>TEAE | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) |
| Preferred<br>term 1 | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) |
| Preferred<br>term 2 | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

Note 2: Both = TEAE related to both treatments, Uli = TEAE related to ulixertinib, HCQ = TEAE related to Hydroxychloriquine.

Related TEAE: TEAEs with causality=Related, Possibly Related or missing.

If there is more than one TEAE within a preferred term (PT), the patient is counted only once in that PT.

PTs are sorted in descending order of frequency for the overall Basket.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.8 - Summary of Serious Treatment-emergent Adverse Events by Preferred Term Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.6
- Present Serious TEAE: TEAEs with SAE =" Yes".
- Add footnote:

"Serious TEAE: TEAEs with SAE =" Yes"."

Table 14.3-1.9 - Summary of Related Serious Treatment-emergent Adverse Events by Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.7
- Present Related Serious TEAE: SAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"SAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.10 - Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term for Maximum CTCAE Grade Full Analysis Set

Basket: Basket X

| System Organ Class<br>Preferred Term | Any CTC Grade<br>n (%) [Events] | CTC Grade 1<br>n (%) | CTC Grade 2<br>n (%) | CTC Grade 3<br>n (%) | CTC Grade 4<br>n (%) | CTC Grade 5<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *************************************** | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>; CTCAE v5.0. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC and maximum severity. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC, PT and maximum severity. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

[Events] presents the number of TEAEs reported overall, by primary SOC and PT regardless of severity.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

Present for each Basket and overall.


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.11 - Summary of Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term for Maximum CTCAE Grade

Full Analysis Set


Basket: Basket X, Related to both study treatments

| System Organ Class<br>Preferred Term | Any CTC Grade<br>n (%) [Events] | CTC Grade 1<br>n (%) | CTC Grade 2<br>n (%) | CTC Grade 3<br>n (%) | CTC Grade 4<br>n (%) | CTC Grade S<br>n (%) |
|---|---|---|---|---|---|---|
| Any related TEAE | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | [XX] (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ********** | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | [XX] (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>; CTCAE v5.0. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC and maximum severity. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC, PT and maximum severity. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

[Events] presents the number of TEAEs reported overall, by primary SOC and PT regardless of severity.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- Present for each Basket and overall. For each Basket and Overall present TEAEs that are Related to both study treatments, related to ulixertinib and related to hydroxychloriquine
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Template Author: Andra Rusu  BMSOP111/F2

Version 5.0 25Jun2020



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.3-1.12 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket l<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE leading to treatment discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE leading to treatment discontinuation within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE leading to treatment discontinuation within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.13 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation by System Organ Class and
Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Table 14.3-1.14 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Within Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn within the first 28 days of study."

Table 14.3-1.15 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Within Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation within cycle 1'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:


"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn within the first 28 days of study."

Template Author: Andra Rusu  BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.16 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn after the first 28 days of study." 
"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Table 14.3-1.17 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Following Cycle 1 by

System Organ Class and Preferred Term

Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation following cycle 1'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn after the first 28 days of study." "Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Template Author: Andra Rusu  BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.18 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption by System Organ Class and Preferred
Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- · Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption.'
- Add footnote:
- "Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted'.

Table 14.3-1.19 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption by System Organ Class and
Preferred Term
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted'.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.20 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption Within Cycle 1 by System Organ Class and Preferred Term

Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption within Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' within the first 28 days of study.

Table 14.3-1.21 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption Within Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption within Cycle 1.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' within the first 28 days of study.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.22 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption Following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption following Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' after the first 28 days of study.

Table 14.3-1.23 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption Following Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption following Cycle 1'.
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' after the first 28 days of study.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.24 - Summary of Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and Preferred Term Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced'".

Table 14.3-1.25 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and
Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced'".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.26 - Summary of Treatment-Emergent Adverse Events Leading to Dose Reduction within Cycle 1 by System Organ Class and
Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction within Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' within the first 28 days of study".

Table 14.3-1.27 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction within Cycle 1 by System Organ

Class and Preferred Term

Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction within Cycle 1.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' within the first 28 days of study".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.28 - Summary of all Treatment-Emergent Adverse Events Leading to Dose Reduction following Cycle 1 by System Organ Class and Preferred Term

Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction following Cycle 1.
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' after the first 28 days of study".

Table 14.3-1.29 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction following Cycle 1.
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' after the first 28 days of study".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.30 - Summary of Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term
Full Analysis Set

| System Organ Class<br>Preferred Term | Basket l<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE leading to death within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE leading to death within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

TEAEs leading to Death: any TEAE resulting in death, Outcome=Fatal, CTC Grade=5.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.31 - Summary of Related Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term Full Analysis Set


## PROGRAMMING NOTES:

Repeat Table 14.3-1.3

- Replace 'Any TEAE' by 'Any related TEAE leading to death'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

"TEAEs leading to Death: any TEAE resulting in death, Outcome=Fatal, CTC Grade=5."

Template Author: Andra Rusu Version 5.0 25Jun2020  BMSOP111/F2


Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Table 14.3-1.32 - Summary of Deaths
All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients who died during the study | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary cause of death Progressive Disease Adverse Event Unknown Patients who died after taking the first dose of | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ulixertinib Primary cause of death Progressive Disease Adverse Event Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.1 - Summary and Change from Baseline in Hematology Laboratory Results by Visit
Full Analysis Set

Parameter: XXXXX (XX)

| Visit | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Present for all hematology parameters: hematocrit, hemoglobin, platelets, white blood cells (WBC), neutrophil absolute, lymphocyte absolute with respective unit measure.
- Present for all available visits.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.3-2.2.1 - Gradable Hematology Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set

| Parameter (unit)<br>Cycle | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| CTCAE Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX (XXX) | | | | | | |
| Cycle 1 | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | | | | | |

Note: CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

• Present for all hematology parameters where CTCAE grades are defined as per the SAP appendix 14.2.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.2.2 - Non-gradable Hematology Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set


| Parameter (unit) | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Cycle | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| CTCAE Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX (XXX) | | | | | | |
| Cycle 1 | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | | | | | |

Note: CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

Present for all hematology parameters where CTCAE grades are not defined as per the SAP appendix 14.2.

Template Author: Andra Rusu  BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.3.1 - Shift Table of Gradable Hematology Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set


Filename: (Specify file name.rtf)

Basket: Basket 1 (N=XX)

| | | | W | orst CTCAE grade | during treatmer | nt period | | |
|---|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Normal | 1 | 2 | 3 | 4 | Missing | Total |
| (unit) | Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (XXX) | 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| | 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| | 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| | 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |

Note: CTCAE v5.0.

Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

### PROGRAMMING NOTES:

Present for each Basket and overall, and for all hematology parameters where CTCAE grades are defined as per the SAP appendix 14.2.

BMSOP111/F2

Template Author: Andra Rusu 
Version 5.0 25Jun 2020



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.3.2 - Shift Table of Non-gradable Hematology Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

Basket: Basket 1 (N=XX)

| Worst grade during treatment period | |
|-------------------------------------|-----------|
| Missing | Total |
| n (%) | n (%) |
| XX (XX.X) | XX (XX.X) |
| XX (XX.X) | XX (XX.X) |
| XX (XX.X) | XX (XX.X) |
| XX (XX.X) | XX (XX.X) |
| XX (XX.X) | XX (XX.X) |
| | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

### PROGRAMMING NOTES:

Present for all Baskets and overall, and for all hematology parameters where CTCAE grades are not defined as per the SAP appendix 14.2.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-2.4 - Summary and Change from Baseline in Biochemistry Laboratory Results by Visit
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat Table 14.3-2.1
- Present for all biochemistry parameters: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, carbon dioxide, calcium, chloride, cholesterol, creatinine, glucose, inorganic phosphorus, lactate dehydrogenase, potassium, total protein, sodium, total bilirubin, triglycerides, uric acid, urea nitrogen.
- Present for all available visits.

Table 14.3-2.5.1 - Gradable Biochemistry Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set

### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.2.1
- Present for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Table 14.3-2.5.2 - Non-gradable Biochemistry Laboratory Results - Worst On-treatment Value by Cycle
Full Analysis Set

### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.2.2
- Present for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Table 14.3-2.6.1 - Shift Table of Gradable Biochemistry Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.3.1
- . Present for all Baskets and overall, and for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-2.6.2 - Shift Table of Non-gradable Biochemistry Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.3.2
- Present for all Baskets and overall, and for all biochemistry parameters where CTCAE grades are not defined as per the SAP appendix 14.2.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-2.7 - Summary at Baseline in Coagulation Laboratory Results Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-2.1
- Present for all coagulation parameters: PT, INR, PTT




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.3-2.8 - Summary at Baseline in Urinalysis Laboratory Results
Full Analysis Set

Parameter: Specific gravity (XX)

| | | N=XX | N=XX | N=XX | N=XX |
|---|---|---|---|---|---|
| XX | XX | XX | XX | XX | XX |
| XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| | XX.X (XX.XX) | XX.X (XX.XX) XX.X (XX.XX) | XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) | XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) | XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X XX.X |

Note: Baseline is the last available assessment prior to first dose of study treatment.


Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Template Author: Andra Rusu Version 5.0 25Jun2020 BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.8 - Summary and Change from Baseline in Urinalysis Laboratory Results by Visit
Full Analysis Set

Parameter: Blood (XX)

| | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Visit | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Statistics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | | | | | | |
| Negative | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<cont.>

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

- Present for all urinalysis parameters: specific gravity, protein, glucose, occult blood, microscopic examination of RBC, microscopic examination of WBC, microscopic examination of casts.
- Present for all available visits.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.1 - Summary and Change from Baseline in Vital Signs by Visit Full Analysis Set

Parameter: XXXXX (XX)

| Visit | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Baseline | | | | | | |
| | XX | *** | *** | 00 | 99 | 99 |
| n | | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- Present for all vital signs: systolic blood pressure, diastolic blood pressure, pulse, respiratory rate, pulse oximetry and temperature with respective unit measure.
- Present for all available visits.


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.2 - Shift Table of Vital Signs Results - Baseline vs Worst On-treatment Value Full Analysis Set

Basket: Basket 1 (N=XX)

| | | | Worst value during on-treatment period | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Low | Normal | High | Very High | Missing | Total |
| (unit) | Value | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX | Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (XXX) | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Very High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

For Temperature, Low: < 36.4°C, Normal: 36.4°C - 37.7°C, High: > 37.7°C.

For Pulse, Low: < 55 bpm, Normal: 55-100 bpm, High: 101-150 bpm, Very high: > 150 bpm.

For Systolic blood pressure, Low: < 90 mmHg, Normal: 90-130 mmHg, High: 131-160 mmHg, Very high: ≥ 161 mmHg. For Diastolic blood pressure, Low: < 60 mmHg, Normal: 60-85 mmHg, High: 86-100 mmHg, Very high: ≥ 101 mmHg.

For Pulse oximetry, Very Low: < 90 %, Low: 90-95 %, Normal: ≥ 95 %.

For Respiratory Rate, Low: < 12 breaths/min, Normal: 12-16 breaths/min, High: > 16 breaths/min.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

### PROGRAMMING NOTES:

Present for each Basket and overall, and for all vital signs parameters.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.3 - Summary and Change from Baseline in ECG parameters by Visit
Full Analysis Set

Parameter: XXXXX (XX)

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to Cl | D8 | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- Present for all ECG parameters: heart rate, PR interval, QRS duration, RR interval, QT interval, QTcF with respective unit measure.
- Present for all available visits.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.4 - Summary of ECHO at Baseline Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Significant findings - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | | | | | - |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| LVEF | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.5 - Summary of Physical Examination at Baseline Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HEENT | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Thorax | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abdomen | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

Present for all Region/Body System parameters: HEENT, thorax, abdomen, skin and mucosae, neurological, extremities, urogenital, general
appearance, heart, back, lymph nodes.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.6 - Summary of ECOG Performance Status by Visit
Full Analysis Set

| Visit | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline [a] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| C1D8 [a] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| i | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 5 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| C1D15 [a] | | | | | | |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <cont.></cont.> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

- [a] (0) Fully active, able to carry on all pre-disease performance without restriction
  - (1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  - (2) Ambulatory and capable of all self-care but unable to carry out any work activities
  - (3) Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  - (4) Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  - (5) Death

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

### PROGRAMMING NOTES:

Present for all available visits.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.5-1.1 - Pharmacokinetic Concentration Data PK Analysis Set

| <i>l</i> isit<br>Analyte | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| CIDIS | | | | | | |
| BVD-523 (ng/mL) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XXX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Geometric Mean (CV%) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XXX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

GSD=Geometric Standard Deviation, SD=Standard Deviation

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.doc)

### PROGRAMMING NOTES:

Present for all available analytes (BVD-523, BVD-502/503,BVD-506, BVD-513) and visits


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.5-1.2 - Pharmacokinetic Parameters Data PK Analysis Set

Analyte: BVD-523

| Visit | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| C1D15 | | | | | | |
| C <sub>Max</sub> (ng/mL)<br>n<br>Mean (SD) | XX XX.XX (XX.XX) | XX<br>XX.XX (XX.XX) | XX<br>XX.XX (XX.XXX) | XX (XX.XX) | XX (XX.XX) | XX<br>XX.XX (XX.XX) |
| Geometric Mean (CV%)<br>Median<br>Min; Max | XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX.XX (XX.XXX) XX.XX XX.X; XX.X | XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX.XX (XX.XX) XX.XX XX.X; XX.X | XX.XX (XX.XX) XX.XX XX.X; XX.X |

GSD=Geometric Standard Deviation, SD=Standard Deviation

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)

### PROGRAMMING NOTES:

Present for all available analytes (BVD-523, BVD-502/503, BVD-506, BVD-513), PK parameters (AUC, Cmax, Cmin, t<sub>1/2</sub>, t<sub>max</sub>), and visits


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Figure 14.2-1.1 - Consort Diagram
Full Analysis Set



Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Y


Figure 14.2-1.2.1 - Spider plot of Percentage Change from Baseline in Sum of Longest Diameter
Full Analysis Set



Weeks since Treatment Initiation

Best overall response: CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progression Disease, NE=Not Evaluable.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

### PROGRAMMING NOTES:

- · Present all Baskets in separate figures and one figure with all patients.
- · Use a different line style for each BOR (dotted line, dashed line, etc).
- Add reference lines for +20% and -30%.

Figure 14.2-1.2.2 - Spider plot of Percentage Change from Baseline in Sum of Longest Diameter Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.2.1
- · Present data on Evaluable Analysis Set.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.3.1 - Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter Full Analysis Set


Basket = Basket X (N=XX)



Maximum percentage decrease from baseline in total tumor size is the maximum percentage decrease in the sum of longest diameters/short axis for all target lesions observed from baseline for each patient.

Best overall response: CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progression Disease, NE=Not Evaluable.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

### PROGRAMMING NOTES:

- Present each Basket on one figure and one figure with all patients. For overall figure, use a different color for each basket
- Each bar is an individual patient.
- Add reference lines for +20% and -30%.
- · Add the best overall response (CR, PR, SD, PD, NE) of each patient on the top of each bar.

Figure 14.2-1.3.2 - Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter
Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.3.1
- Present data on Evaluable Analysis Set.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Figure 14.2-1.4.1 - Swimmer Plot of Response Assessments Full Analysis Set



Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### PROGRAMMING NOTES:

- Present each Basket on one figure and a figure including all patients.
- · Display patient ID on the left outside the figure except for the figure where all patients are displayed.
- The bar displays time to PD/Death (PFS), with "PD" or "death" displayed at the end of the bar; if no PD/death occurred before cutoff date, the bar stops at cutoff date.
- For responders, display the date of first CR or PR, and display "Ongoing response" arrow if no PD or death occurred before cutoff date.
- "End of Treatment" is the date of treatment discontinuation, this must be displayed only for patients who discontinued the treatment before the
  cut-off date.

Figure 14.2-1.4.2 - Swimmer Plot of Response Assessments Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.4.1
- · Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.5.1 - Kaplan-Meier Estimate for Progression-Free survival (PFS)
Full Analysis Set




Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### PROGRAMMING NOTES:

- X-axis Label "Progression Free Survival (months)"
- Y-axis Label "Event-free probability (%)."
- Legend: overall number of events, "Median Duration of Response" and 95% Cl.
- Flag censored observations with '+' and add legend.
- If the median time to event has not been reached, present as "Median (95% CI) NR (xx.x, xx.x)" [replacing xx.x with '-' if there is no upper or lower confidence limit] and add footnote:
  - NR=Median time not reached.
- Present all Baskets on the same figure but with different colors and separate figures for each Basket. In the sample shell where it is 'Cohort' replace with 'Basket'

Figure 14.2-1.5.2 - Kaplan-Meier Estimate for Progression-Free survival (PFS)

Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.5.1
- Present data on Evaluable Analysis Set.

Figure 14.2-1.6.1 - Kaplan-Meier Estimate for Overall Survival (OS)
Full Analysis Set

### PROGRAMMING NOTES:

Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Overall Survival" in X-axis label and legend.

Figure 14.2-1.6.2 - Kaplan-Meier Estimate for Overall Survival (OS)
Evaluable Analysis Set

## PROGRAMMING NOTES:

- Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Overall Survival" in X-axis label and legend.
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Figure 14.2-1.7.1 - Kaplan-Meier Estimate for Duration of Response Full Analysis Set

# PROGRAMMING NOTES:

• Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Duration of Response" in X-axis label and legend.




Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Listing 16.2.1-1 - Patients informed consent All Patients Set

Basket: Basket 1

| | | | Main Infor | med Consent | Optional End of | Treatment Biopsy | | |
|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Age /<br>Gender | Protocol<br>Version | Consent Obtained / Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn | Consent Obtained /<br>Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn | Consent Obtained / Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn |
| xxxxxx | XX/M | 1.0 | Yes / Yes | DDMMMYYYY /<br>DDMMMYYYYY | Yes | DDMMMYYYY /<br>DDMMMYYYYY | Yes | DDMMMYYYY / |
| XXXXXX | XX/F | 1.0 | Yes / No | DDMMYYYY | Yes | DDMMYYYY | Yes | DDMMYYYYY |
| XXXXXX | XX/F | 1.0 | Yes / No | DDMMYYYYY | Yes | DDMMYYYY | Yes | DDMMYYYYY |
| XXXXXX | XX/F | 1.0 | No / Yes | DDMMYYYYY<br>DDMMYYYYY | No | DDMMYYYY | No | DDMMYYYY |
| <cont.></cont.> | | | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.doc)

# PROGRAMMING NOTE:

• For all Listings, repeat for each Basket. For All Patients Set present group Screen Failures




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.1-2 - Failed Inclusion and Exclusion Criteria
All Patients Set


Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Protocol<br>Version | Failed Inclusion /<br>Exclusion No. | Description |
|---|---|---|---|---|
| жж-жж | xx/M | 1.0 | INCL01 | XXXXXXXXXX |
| xx-xx | xx/M | 1.0 | EXCL01 | xxxxxxxxxx |
| xxx-xx | xx/M | 1.0 | EXCL02 | xxxxxxxxxxx |
| xxx-xx | xx/F | 1.0 | INCL02 | XXXXXXXXXXX |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

List all failed Inclusion / Exclusion criteria as per eCRF.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.1-3 - Patient Disposition All Patients Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Enrolled | Date of<br>Assignment | Gene/ Codon/<br>Amino acid<br>change | Completed<br>Screening /<br>Reason | Date of<br>Screening<br>Completion /<br>Discontinuation | Eligible for inclusion? | Rescreened? /<br>Previous patient<br>number |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Yes | DDMMYYYY | BRAF /D594 /<br>Alanine A | Yes | DDMMYYYY | Yes | No |
| xx-xx | xx/F | Yes | DDMMMYYYY | MEK1/MAP2K1 /<br>K601 /Arginine R | No /<br>Physician<br>Decision | DDMMYYYY | Yes | Yes /xxxxxxx |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Listing 16.2.1-3 - Patient Disposition All Patients Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Completed<br>Treatment /<br>Reason | Date of Treatment<br>Discontinuation | Date of Last Study<br>Dose | Completed Study /<br>If no, reason | Date of Completion |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | Yes | DDMMYYYYY | DDMMYYYYY | Yes | DDMMYYYYY |
| жж-жж | им/F | No/<br>Progressive<br>Disease | DDMMYYYYY | DDMMYYYYY | No/ xxxxxx | DDMMYYYY |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


### Listing 16.2.2-1 - Analysis Sets All Patients Set

#### Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | All Patients Set [a] | Full Analysis Set<br>[b] | Stage 1 Analysis Set<br>[c] | Evaluable Analysis<br>Set [d] | PK Analysis<br>Set [e] |
|---|---|---|---|---|---|---|
| хх-хх | xx/M | Yes | Yes | Yes | Yes | Yes |
| xx-xx | xx/F | Yes | Yes | Yes | Yes | Yes |

### Note: M=Male, F=Female.

- [a] Patients who were enrolled regardless of whether they received the study drug or not.
- [b] Patients who received at least 1 dose of the study drug.
- [c] First 13 patients who have completed at least one cycle of therapy and who have received a minimum of 75% of prescribed study therapy during Cycle 1
- [d] Patients who received at least one dose of study drug and have at least one post-treatment study evaluation or who have discontinued therapy prior to the first post-treatment study evaluation due to clinical progressive disease or drug-related adverse events.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.3-1 - Protocol Deviations Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Deviation<br>Category | Summary Term | Deviation<br>Description | Classification | Exclusion from<br>Analysis Sets |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | Inclusion<br>Criteria<br> | xxxxxxxxxx | XXXXXXXXXXXX | Important | Evaluable Analysis<br>Set |
| xx-xx | xx/F | Study<br>Assessments<br> | ********** | XXXXXXXXXXXX | Non-Important | Full Analysis Set |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

· Categories / Summary Term / Description to match the PDCF.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-1 - Demographics and Baseline Characteristics Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Childbearing/<br>Reproductive<br>Potential | Surgery<br>Name | Date of<br>Surgery/Post-<br>Menopausal | Date of Last<br>Menstrual<br>Period | Race | Ethnicity | Height at<br>Screening<br>(cm) | Weight at<br>Screening<br>(kg) |
|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Surgically<br>Sterile | Vasectomy | DDMMMYYY | | White | Hispanic or<br>Latino | xx | xx |
| xx-xx | xx/F | Able to Bear<br>Children | | | DDMMYYY | Other, | Not<br>Hispanic or<br>Latino | xx | ж |
| xx-xx | xx/F | Sterile -<br>Other Reason,<br>xxxxxx | | | DDMMMYYY | | | | |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-2 - Smoking History Full Analysis Set

Basket: Basket 1

| Danie . D | 45.200 1 | | | |
|---|---|---|---|---|
| Patient<br>ID | Age /<br>Gender | Smoking<br>History? | Substance | Usage |
| xx-xx | xx/M | Yes | Cigarettes | Former |
| xx-xx | xx/F | No | | |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-3 - Disease History Full Analysis Set

Basket: Basket 1

| Patient ID | Age /<br>Gender | Cancer<br>Diagnosis | Date of<br>Initial<br>Diagnosis | Time since<br>Initial<br>Diagnosis [a] | Stage at<br>Diagnosis | Method of<br>Diagnosis | Current<br>Stage at<br>Enrollment | Prior<br>Radiation<br>Therapies? |
|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Stomach | DDMMMYYYY | xx | 1 | Cytological | 1 | Yes |
| xxx-xx | xx/F | Other,<br>xxxxx | DDMMYYYY | xx | 2 | Histological | 4 | No |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-4 - Medical History and Concomitant Diseases Full Analysis Set


Basket: Basket 1

| Patient | Age / | | System Organ | | Start Date ( | (Day) | | |
|---|---|---|---|---|---|---|---|---|
| ID | Gender | Reported Term | Class | Preferred Term | /End Date (I | Day) | Ongoing | MH or Conc. |
| xx-xx | xx/M | xxxxxxx | xxxxxxxx | XXXXXXX | DDMMMYYYY (x | | No | МН |
| xx-xx | xx/F | xxxxxxx | xxxxxxxx | xxxxxxx | DDMMYYYYY (x | xx) | Yes | Conc. |

#### Note: M=Male, F=Female.

MedDRA <vx.x>.

Study day is calculated as (Event Date - Study treatment start date) for dates before Study treatment start date and (Event date - First treatment date + 1) for dates after Study treatment start date.

Medical history (MH): any conditions that started before the first study treatment date and were not ongoing at the first study treatment date.

Concomitant disease (Conc.): any conditions that started before first study treatment administration and were ongoing at first study treatment administration.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-5 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Line of<br>Therapy | Name of<br>Therapy | Start Date<br>(Day) | End Date<br>(Day) | Best Overall<br>Response | Date of Best<br>Overall<br>Response | Date of<br>Relapse/<br>Progression | Reason for<br>Discontinuati<br>on |
|---|---|---|---|---|---|---|---|---|---|
| хх-хх | xx/M | 1 | xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | Stable<br>Disease | DDMMYYYY | DDMMMYYYY | Intolerance |
| xx-xx | xx/M | 1 | XXXXX | DDMMYYYYY<br>(xx) | DDMMYYYYY<br>(xx) | Stable<br>Disease | DDMMYYYY | DDMMYYYY | Lack of<br>Efficacy |
| xx-xx | xx/F | 4 | xxxxx | DDMMMYYYY<br>(xx) | DDMMYYYY<br>(xx) | Partial<br>Response | DDMMYYYY | DDMMMYYYY | Other, |

Note: M=Male, F=Female.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication

date - First treatment date  $\dagger$  1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Data taken from 'Prior Cancer Medications' page.


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-6 - Prior Radiotherapy Courses Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Site of Radiotherapy | Dose (Unit) | Start Date (Day) | End Date (Day) | Duration<br>(months) [a] |
|---|---|---|---|---|---|---|
| xxx-xx | жж/М | Abdominal Cavity | xxx (xxx) | DDMMMYYYY (xx) | DDMMYYYYY (xx) | xx |
| xx-xx | xx/M | Adrenal Gland | xxx (xxx) | DDMMMYYYY (xx) | DDMMYYYY (xx) | жж |
| xx-xx | xx/F | Bile Duct | xxx (xxx) | DDMMMYYYY (xx) | DDMMYYYY (xx) | жx |

Note: M=Male, F=Female.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication date - First treatment date + 1) for dates after Study treatment start date.

[a] Duration of radiotherapy calculated as [(end date - start date) + 1] / 30.4375.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Data taken from 'Prior Radiotherapy' page.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-7 - Prior and Concomitant Medications Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Reported Term /<br>Preferred Term /<br>ATC Class | Indication | Start Date<br>(Day) | End<br>Date (Day) | Dose<br>(Units) /<br>Frequency | Route | Medication to<br>treat<br>adverse event? /<br>Adverse Event (ID) | Ongoing | Prior<br>/<br>Conc. |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Xxxxxxxxxxx /<br>xxxxxxxx /<br>xxxxxx | XXXXX | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | иии (ии)<br>/ Daily | Oral | Yes / xxxx (x) | Yes | Conc. |
| жж-жж | xx/F | ************************************** | XXXXXX | DDMMMYYYY<br>(xx) | Ongoing | xxx (xx)<br>/ Twice<br>per day | Oral,<br>xxxx | No | No | Prior |

Note: M=Male, F=Female, ATC=Anatomical Therapeutic Chemical.

WHOHD-B3 <vx.x>.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication date - First treatment date + 1) for dates after Study treatment start date.

Prior medication (Prior): any medications whose end date is before the first study treatment date.

Concomitant medication (Conc.): any medication whose start or end date is either the same or after the first dose of study treatment and up to the end of the on-treatment period.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- Data taken from 'Prior and Concomitant Medications' page.
- Adverse Event ID taken from collected ID.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Listing 16.2.4-8 - On Treatment Radiation Full Analysis Set

Cohort: Basket 1

| Patient<br>ID | Age /<br>Gender | Received<br>Radiation? | Site of<br>Radiotherapy | Dose (Unit) | Start Date (Day) | End Date (Day) |
|---|---|---|---|---|---|---|
| жж-жж | xx/M | Yes | Abdominal Cavity | xxx (xxx) | DDMMMYYYY (xx) | DDMMMYYYY (xx) |
| xx-xx | xx/M | Yes | Adrenal Gland | xxx (xxx) | DDMMMYYYY (xx) | DDMMMYYYY (xx) |
| xx-xx | xx/F | No | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

· Data taken from 'On Treatment Radiation' page.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-9 - On Treatment Surgery and Medical Procedures Full Analysis Set

Cohort: Basket 1

| Patient<br>ID | Age /<br>Gender | Any Surgeries/<br>Procedures | Name of Surgery/<br>Procedure | Indication? | Start Date (Day) | End Date (Day) | Ongoing? |
|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Yes | xxxxxxxxx | xxxxxxxxx | DDMMYYYY (xx) | DDMMMYYYY (xx) | No |
| xx-xx | xx/M | Yes | xxxxxxxxx | xxxxxxxxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | Yes |
| xx-xx | xx/F | No | | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Data taken from 'On Treatment Surgery and Medical Procedures' page.


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-10 - On Treatment Blood Transfusions Full Analysis Set


Filename: (Specify file name.rtf)

Cohort: Basket 1

| Patient ID | Age/<br>Gender | Any blood<br>transfusions | Transfusion ID | Date of Transfusion | Category of Transfusion | Units |
|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Yes | xxxxxxxxx | DDMMYYYY (xx) | Platelet transfusion | xx |
| | xx/M | Yes | xxxxxxxxx | DDMMMYYYY (xx) | Plasma | xx |
| xx-xx | xx/F | No | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## PROGRAMMING NOTES:

· Data taken from 'On Treatment Blood Transfusions' page.

Template Author: Andra Rusu Version 5.0 25Jun2020  BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Listing 16.2.4-11 - NGS Data Full Analysis Set

Cohort: Basket 1

| Patient ID | Age/<br>Gender | Gene / Codon /<br>Amino acid change | Vendor | Date of Report | Report Redacted | Report Uploaded |
|---|---|---|---|---|---|---|
| xx-xx | M/XX | BRAF /D594 /<br>Alanine A | STRATA | DDMMMYYYY (xx) | Yes | Yes |
| xxx-xx | xx/F | MEK1/MAP2K1 /<br>K601 /Arginine R | GUARDANT | | No | No |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-1 - Ulixertinib In-clinic Administration Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Treatment<br>Administered? | Dose (mg) | Dose Date and Time (day) |
|---|---|---|---|---|
| xx-xx | xx/M | Yes | xxx | DDMMYYYY hh:mm (xx) |
| xxx-xx | xx/F | Yes | xxx | DDMMYYYY hh:mm (xx) |
| xx-xx | xx/F | Yes | Xxx | DDMMMYYYY hh:mm (xx) |

Note: M=Male, F=Female.

Study day is calculated as Administration date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.5-2 - Hydroxychloroquine In-clinic Administration Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-1




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Listing 16.2.5-3 - Ulixertinib Interruptions and Adjustments Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Type of Change | Start Date / End Date /<br>Duration (days) | If Adjustment, new dose amount (mg) | Reason for<br>Interruption/Adjustment |
|---|---|---|---|---|---|
| xx-xx | xx/M | Interruption | DDMMYYYYY / DDMMYYYYY / (xx) | xxx | Adverse Event |
| xx-xx | xx/F | Adjustment | DDMMYYYY / DDMMYYYYY / (xx) | xxx | Other, |
| xx-xx | xx/F | | | | |

Note: M=Male, F=Female.

Study day is calculated as Interruption/Change date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.5-4 - Hydroxychloroquine Interruptions and Adjustments Full Analysis Set

### PROGRAMMING NOTES:

Repeat Listing 16.2.5-3




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.5-5 - Ulixertinib Exposure Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Number of<br>cycles<br>received [a] | Duration of<br>exposure<br>(months) [b] | Planned cumulative<br>dose (mg) | Actual cumulative dose received (mg)[c] | Relative dose intensity [d] |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | xx | xxx | жжж (mg) | xxx (mg) | xxx |
| xxx-xx | xx/F | жж | xxx | xxx (mg) | xxx (mg) | XXX |

Note: M=Male, F=Female.

- [a] Number of cycles received = Number of cycles where the patient received at least one dose.
- [b] Duration of exposure (months) = (Date of last known treatment dosing with ulixertinib- date of initial dosing with ulixertinib) + 1 / 30.4375.
- [c] Actual cumulative dose received (mg) = Sum of [(number of capsules dispensed number of capsules returned) x 150].
- [d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days). Planned cumulative dose is the number of cycles received x number of doses per day x mg prescribed per dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-6 - Hydroxychloroquine Exposure Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-5




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-7 - Ulixertinib Dispensed Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Mg<br>prescribed<br>per dose | Date<br>Bottles<br>Dispensed<br>(day) | Number of<br>Bottles<br>Dispensed | Lot Number<br>of the<br>bottles<br>dispensed | Different Lot<br>number<br>dispensed to<br>the patient? | Lot number<br>dispensed to<br>patient /No of<br>bottles | Total<br>Number of<br>Capsules<br>Dispensed |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | xxx | DDMMMYYYY<br>(xx) | xx | xxxx | Yes | Xxxx/XX | жж |
| xx-xx | xx/F | xxx | DDMMMYYYY<br>(xx) | xx | xxxx | No | | жж |

Note: M=Male, F=Female.

Study day is calculated as Dispensed date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-8 - Hydroxychloroquine Dispensed Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-7




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-9 - Ulixertinib Returned Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Cycle | Reason<br>capsules<br>not<br>returned | Date<br>Returned<br>(day) | Patient<br>compliant<br>since last<br>visit? If<br>no, reason | Missed dose<br>related to an<br>adverse event? | Number of<br>Bottles Returned | Lot Number<br>of the<br>bottles<br>returned | Total<br>Number of<br>Capsules<br>Returned |
|---|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | 2 | Lost | DDMMMYYYY<br>(xx) | Yes | Yes | xx | xxxx | xxx |
| xx-xx | xx/F | 3 | Other, xxxxx | DDMMMYYYY<br>(xx) | No, жжжж | Yes | xx | xxxx | xxx |

Note: M=Male, F=Female.

Study day is calculated as Returned date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-10 - Hydroxychloroquine Returned Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-9



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-1 - Target Lesions Full Analysis Set Page 1 of Y

Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Visit | Target<br>Lesions at<br>Screening? | Lesion<br>Number | Tumor<br>Type | Organ<br>Site | Method | Date of<br>Scan<br>(Day) | Longest<br>Diameter/<br>Short-<br>axis(mm) | Sum of Longest Diameter (mm)<br>/ Change from baseline / %<br>Change from baseline |
|---|---|---|---|---|---|---|---|---|---|---|
| хх-хх | xx/M | Screening<br>C2D1 | Yes | T01 | Primary | Bladder | CT<br>Scan | DDMMYYYYY<br>(xx) | xxx | XXX |
| хх-хх | xx/F | <br>Screening | Yes | T02 | Metastasis | Other, | MRI | DDMMYYYY<br>(xx) | xxx | xxx / xxx / xxx |
| xx-xx | xx/F | Screening<br> | Yes | T02 | Metastasis | | MRI | | xxx | xxx / xxx / xxx |

Note: M=Male, F=Female.

Study day is calculated as (Scan Date - Study treatment start date) for dates before Study treatment start date and (Scan date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.6-2 - Non-Target Lesions Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Visit | Assessment<br>Performed /<br>Reason | Non-Target<br>Lesions at<br>screening | Lesion Number | Organ<br>Site | Method | Date of Scan<br>(Day) | Result |
|---|---|---|---|---|---|---|---|---|---|
| xx-xx | жж/М | Screening<br>C2D1 | Yes<br>No, xxx | Yes | NT01 | Bladder | CT Scan | DDMMYYYY<br>(xx) | Present |
| ***-** | xx/F | Screening | Yes | Yes | NT02 | Other, | MRI | DDMMMYYYY<br>(xx) | Absent<br>(Disappeared) |

#### Note: M=Male, F=Female.

Study day is calculated as (Scan Date - Study treatment start date) for dates before Study treatment start date and (Scan date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


#### Listing 16.2.6-3 - New Lesions Full Analysis Set

Basket: Basket 1

| Patient | Age/ | | Any New | | | | |
|---|---|---|---|---|---|---|---|
| ID | Gender | Visit | Lesions | Lesion Number | Method | Date of Scan (Day) | Organ Site |
| xxx-xx | им/М | C2D29 | Yes | NL01 | CT Scan | DDMMMYYYY (xx) | Abdomen |
| хх-хх | xx/F | C2D29 | Yes | NL02 | Other, | DDMMMYYYY (xx) | Bone |

Note: M=Male, F=Female.

Study day is calculated as Scan date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.6-4 - Overall Response Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Best Overall<br>Response [a] | Assessment<br>Performed/<br>Reason | Date of Assessment (Day) | Target<br>Lesion<br>Response | Non-Target<br>Lesion<br>Response | New Lesions | Overall<br>Response |
|---|---|---|---|---|---|---|---|---|
| хх-хх | xx/M | CR | Yes | DDMMMYYYY (xx) | CR | CR | Yes | PD |
| ххх-хх | xx/F | PD | Yes | DDMMMYYYY (xx) | NE | PD | No | NE,<br>xxxx |

Note: M=Male, F=Female, CR=Complete Response, Non CR/Non PD=Non Complete Response/Non Progressive Disease, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

Study day is calculated as Assessment date - First treatment date + 1.

[a] Confirmed best overall response.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-5 - Progression-Free Survival (PFS) Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Treatment<br>Start Date | Date of<br>Last Tumor<br>Assessment | Date of Event/<br>Censoring | Event / Censoring<br>Reason | PFS (months) |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | DDMMYYYY | DDMMMYYYY | DDMMMYYYY | Death | жж.ж |
| xx-xx | xx/F | DDMMYYYYY | DDMMYYYY | DDMMYYYY | Censored: xxxxx | xx.x |

Note: M=Male, F=Female, PFS=Progression-Free Survival.

Event: progressive disease (PD) or death from any cause.

The PFS (in months) is defined as the time from the first ulixertinib dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-6 - Survival Status Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Completed<br>End of<br>Study? | Any Anti-Cancer<br>Treatment Since End<br>of treatment or<br>Last FUP/ Start<br>Date | Any Tumor Assessment Since<br>End of Study or Last FUP/<br>Assessment Date/<br>Overall Response | Survival<br>Status at<br>Follow-Up | Date of<br>Death | Last Known Date<br>Patient Alive [a] |
|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Yes | Yes/ DDMMYYYY | Yes/ DDMMMYYYY/ Complete<br>Response | Alive | | |
| xx-xx | xx/F | Yes | No | No | Dead | DDMMMYYYY | |

Note: M=Male, F=Female, FUP=Follow-up, CR=Complete Response, Non CR/Non PD=Non Complete Response/Non Progressive Disease, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

[a] If Survival status at the time of follow-up is unknown.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-7 - Duration of Response (DOR) Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Best Overall<br>Response [a] | Treatment<br>Start Date | Date of First<br>Response | Date of<br>Last Tumor<br>Assessment | Date of Event /<br>Censoring | Event /<br>Censoring Reason | Duration of<br>Response<br>(months) |
|---|---|---|---|---|---|---|---|---|
| ххх-хх | xx/M | CR | DDMMYYYY | DDMMYYYY | DDMMYYYY | DDMMYYYY | Death | xx.x |
| ххх-хх | xx/F | PR | DDMMYYYY | DDMMYYYYY | DD <b>MM</b> YYYYY | DDMMYYYY | Censored: xxxxx | xx.x |

Note: M=Male, F=Female, CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

Event: progressive disease (PD) or death from any cause.

This listing includes only patients with response (CR or PR).

Duration of response is the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause.

[a] Confirmed best overall response.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.7-1 - Adverse Events All Patients Set

Basket: Basket 1

| Dasies. Dasi | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Age /<br>Gender | ID | Reported Term | System Organ<br>Class | Preferred Term | Start Date (day) | End Date (day) | TEAE? | SAE? |
| xx-xx | xx/M | xx | XXXXXXXX | xxxxxxxx | xxxxxxxx | DDMMMYYYY (xx) | DDMMYYYYY (xx) | Yes | Yes |
| xx-xx | xx/F | ж | xxxxxxxx | xxxxxxxx | xxxxxxxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | No | No |

Note: M=Male, F=Female, TEAE=Treatment Emergent Adverse Event, SAE=Serious Adverse Event.

ID as collected in the databased. MedDRA <vx.x>. NCI CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.7-2 - Treatment-Emergent Adverse Events Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | ID | Reported Term<br>/ System Organ<br>Class<br>/Preferred<br>Term | Start Date<br>(Day) / End<br>Date (Day) /<br>Duration<br>(days) | SAE /<br>Serious<br>ness | NCI-<br>CTCAE<br>Grade | Relation<br>Ship to<br>Disease | Relation Ship to Ulixertin ib / Hydroxych loroquine | Action Taken with Ulixertinib / Hydroxychlo roquine | Medication<br>or<br>Therapies?<br>/<br>Medication<br>Name | Outcome<br>[a] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | xx | XXXXXXX/<br>XXXXXXXX/<br>XXXXXXXX | DDMMYYYYY<br>(xx) /<br>DDMMYYYYY<br>(xx) / xx | Yes /<br>Hospital<br>ization | 1 | Related | Related<br>/Related | Drug<br>Interrupted<br>/Drug<br>Interrupted | Yes<br>/xxxxxxxx,<br>xxxxxxx | Res'd |
| xx-xx | xx/F | xx | <br>********************************** | DDMMMYYYY<br>(xx) /<br>DDMMMYYYY<br>(xx) / xx | No | 3 | Possibly<br>Related | Possibly<br>Related<br>/Related | Drug<br>Interrupted<br>/Drug<br>Interrupted | Yes<br>/xxxxxxxx | Res'd<br>seq,<br>xxxxxx |

Note: M=Male, F=Female, TEAE=Treatment Emergent Adverse Event, SAE=Serious Adverse Event.

MedDRA <vx.x>. NCI CTCAE v5.0.

ID as collected in the databased.

Study day is calculated as TEAE date - First treatment date + 1.

[a] Res'd=Resolved, Res'd seq=Recovered/Resolved with sequelae, Ong=Ongoing, Unk=Unknown, Fatal=Fatal.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

### PROGRAMMING NOTES:

- · Sort by Basket, patient ID, ascending Adverse Event Start Date and Reported Term.
- Outcome = "Res'd seq" please specify sequelae.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.7-3 - Serious Adverse Events Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.7-2 and include only AEs classified as Serious.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.7-4 - Deaths All Patients Set

#### Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Date of Death (Day) | Autopsy Performed? /<br>Date of Autopsy | Primary Cause of Death | Treatment-Emergent Death |
|---|---|---|---|---|---|
| xx-xx | xx/M | DDMMYYYY (xx) | No | Progressive Disease | Yes |
| xx-xx | xx/F | DDMMMYYYY (xx) | Yes /DDMMYYYY | Adverse Event, xxxxxxx | No |

Note: M=Male, F=Female.

[a] A death is considered Treatment-Emergent if occurred after Ulixertinib administration.

Study day is calculated as Death date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

· Specify primary cause of death if not PD.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.8-1 - Hematology Full Analysis Set Page 1 of Y

Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Study<br>Visit | Sample Date and Time<br>(Day) | Parameter (Unit) | Result /<br>Reference Range<br>Indicator / CS?<br>[a] | LLN - ULN | CTC<br>Grade | Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| ххх-хх | xx/M | Screening | DDMMMYYYY / hh:mm (xx) | RBC (xxx) | жж / L / CS | хх - хх | xx | |
| | | C1D1<br> | DDMMYYYY / hh:mm (xx) | RBC (MMM) | иж / L / CS | хх - хх | xx | xx |
| xxx-xx | xx/F | Screening | DDMMMYYYY / hh:mm | RBC (xxx) | Not Done | | | |
| | | C1D1<br> | | - | | | | |

Note: M=Male, F=Female, L=Low, H=High, ULN=Upper Limit of Normal, LLN=Lower Limit of Normal, CS=Clinically Significant, NCS=Non Clinically Significant.

CTCAE v5.0.

Baseline is the last available assessment prior to first dose of study treatment.

Study day is calculated as (Sample Date - Study treatment start date) for dates before Study treatment start date and (Sample date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- Sort by Basket, patient ID, ascending Sample Date and Time and Parameter.
- Include all hematology parameters.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.8-2 - Biochemistry Full Analysis Set

## PROGRAMMING NOTES:

· Repeat Listing 16.2-8.1 for all biochemistry parameters.

Listing 16.2.8-3 - Coagulation Full Analysis Set

## PROGRAMMING NOTES:

· Repeat Listing 16.2-8.1 for all coagulation parameters.

Listing 16.2.8-4 - Urinalysis Full Analysis Set

### PROGRAMMING NOTES:

Repeat Listing 16.2-8.1 for all urinalysis parameters.

Listing 16.2.8-5 - Tumor Markers Full Analysis Set

## PROGRAMMING NOTES:

Repeat Listing 16.2-8.1 for all tumor marker parameters.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.8-6 - Pregnancy Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Sample<br>Type | Assessment<br>Performed? /Reason | Sample Date (Day) | Result |
|---|---|---|---|---|---|---|
| xx-xx | xx/F | Screening<br>Baseline | Serum | Yes | DDMMYYYY (xx) | Positive |
| xxx-xx | xx/F | Screening | Serum | No /xxxx | | |

Note: F=Female.

Baseline is the last available assessment prior to first dose of study treatment.

Study day is calculated as (Sample Date - Study treatment start date) for dates before Study treatment start date and (Sample date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, visit.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-1 - Vital Signs Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment Date<br>and Time (Day) | Parameter<br>(Unit) | Result/ Reference Range<br>Indicator / CS? [a] | Position | Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY hh:mm (xx) | Systolic Blood<br>Pressure (xxx) | жж / Н / CS | Sitting | |
| | | Baseline | Yes | DDMMMYYYY hh:mm (xx) | Systolic Blood<br>Pressure (xxx) | жж / Н / CS | Supine | |
| | | | | | *** | | | |
| xxx-xx | xx/F | Screening<br> | No / xxxxxx | | | Not Done | | |

Note: M=Male, F=Female, L=Low, H=High, VH=Very High, ND=Not Done, CS=Clinically Significant, NCS=Non Clinically Significant.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, ascending Assessment Date and Time and Parameter.


<sup>[</sup>a] If status = "Not Done" populate with "Not Done".

<sup>\*</sup> Baseline is the last available assessment prior to first dose of study treatment.

For temperature, Low if < 36.4°C; high if > 37.7°C.

For pulse, Low if < 55bpm; high if 101-150bpm; very high if > 150bpm.

For systolic blood pressure, Low if < 90mmHg; high if 131-160mmHg; very high if >= 161mmHg.

For diastolic blood pressure, Low if < 60mmHg; high if 86-100mmHg; very high if >= 101mmHg.

For Pulse oximetry, Very Low: < 90 %, Low: 90-95 %, Normal: ≥ 95 %.

For Respiratory Rate, Low: < 12 breaths/min, Normal: 12-16 breaths/min, High: > 16 breaths/min.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


#### Listing 16.2.9-2 - Electrocardiogram Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment Date and Time (Day) | Method/<br>Position | Parameter<br>(Unit) | Result /CS? | Change from baseline |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMMYYYY hh:mm (xx) | 12 Lead<br>Standard/<br>Supine | Heart Rate<br>(xxx) | xx /No | |
| xx-xx | xx/F | Screening | Yes | DDMMMYYYY hh:mm | 12 Lead<br>Standard/<br>Supine | Heart Rate (xxx) | xx /Yes | |

Note: M=Male, F=Female, L=Low, H=High.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, ascending Assessment Date and Time and Parameter.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-3 - ECHO Full Analysis Set

Basket: Basket 1

| Patient | Age / | Assessment<br>Performed? / | | | | |
|---|---|---|---|---|---|---|
| ID | Gender | Reason | Method | Assessment Date (Day) | Parameter (Unit) | Result /CS? |
| xxx-xx | xx/M | Yes | Echocardiography | DDMMYYYY (xx) | LVEF (xx) | xx /No |

Note: M=Male, F=Female, LVEF=Left Ventricular Ejection Fraction.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, ascending Assessment Date and Time.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-4 - Physical Examination Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment<br>Date | Region /Body<br>System | Result /CS? [a] | Abnormal<br>Findings |
|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY | HEENT | Abnormal/ CS | xxxxxx |
| xxx-xx | xx/F | Screening | Yes | DDMMYYYY | Thorax | Not Done | |

Note: M=Male, F=Female, CS=Clinically Significant, NCS=Non Clinically Significant.

[a] If status = "Not Done" populate with "Not Done".

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, Region/body system.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-5 - Ophthalmology Exam Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment<br>Date | Examination Test | Any Abnormal<br>Clinically<br>Significant<br>Result? | Eyes<br>Affecte<br>d | Abnormal Finding |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY | Best-corrected visual acuity | Yes | Left | xxxxxxxxx |
| xx-xx | xx/F | Screening | Yes | DDMMYYYY | ••• | Yes | Both | |

Note: M=Male, F=Female, CS=Clinically Significant, NCS=Non Clinically Significant.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, examination test name




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.9-6 - ECOG Performance Status Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Date of Assessment (Day) | ECOG Performance Status [a] |
|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY (xx) | (0) Fully Active |
| | | Baseline<br> | Yes | DDMMMYYYY (xx) | (0) Fully Active |
| xx-xx | xx/F | Screening | Yes | DDMMYYYY (xx) | (1) Restricted |
| | | Baseline<br> | No, xxxx | | |

Note: M=Male, F=Female.

Baseline is the last available assessment prior to first dose of study treatment.

- [a] (0) Fully active, able to carry on all pre-disease performance without restriction
  - (1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  - (2) Ambulatory and capable of all self-care but unable to carry out any work activities
  - (3) Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  - (4) Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  - (5) Death

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


#### PROGRAMMING NOTES:

Sort by Basket, patient ID, visit, assessment date.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.11-1 - Pharmacokinetic Concentration Data Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Collection Date/Time (Day) / Timepoint | Analyte | Concentration (Unit) |
|---|---|---|---|---|---|
| | | | | | xxxx (ng/mL) |
| xx-xx | xx/M | C1D15 | ddmmmyyyy hh:mm (xx) / Pre-dose | BVD-523 | |

---

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, assessment date and time.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.11-2 - Pharmacokinetic Parameters Data Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Visit | Analyte | PK Parameter | Result |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | C1D15 | C1D15 | BVD-523 | AUC | xxxx |

---

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit and analyte.


# **DocuSign**

#### Certificate Of Completion

Envelope Id: 9D451F5DDB6A406CBCF295C356DEEC6D

Subject: Complete with Docusign: BVD-523-HCQ\_SAP\_v2.0\_02Sep2024.pdf

Source Envelope:

Document Pages: 185 Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Status: Completed

Envelope Originator:

Julien Lucas

julien.lucas@aixial.com IP Address: 77.66.37.185

#### **Record Tracking**

Status: Original

02-Sep-2024 | 16:21

Holder: Julien Lucas

julien.lucas@aixial.com

Location: DocuSign

#### Signer Events

Anna Groover

agroover@biomed-valley.com

Senior Scientist

Security Level: Email, Account Authentication

(Required)

#### Signature

Signatures: 6

Initials: 0

—Signed by: Acce Acces

Signer Name: Anna Groover
Signing Reason: I approve this document

Signing Time: 03-Sep-2024 | 08:40 CDT -71380BDD08BC4D289E63FA3831CD4243

Signature Adoption: Pre-selected Style

Signature ID:

71380BDD-08BC-4D28-9E63-FA3831CD4243

Using IP Address: 136.37.127.159

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

Electronic Record and Signature Disclosure: Accepted: 03-Sep-2024 | 14:39

ID: 94d5e37d-2fb2-42f9-ab4e-2e7b997de2ae

Brent Kreider

bkreider@biomed-valley.com

President

Security Level: Email, Account Authentication

(Required)

Signed by:

Breat Kreider

Signer Name: Brent Kreider Signing Reason: I approve this document Signing Time: 04-Sep-2024 | 08:58 PDT

Signature Adoption: Pre-selected Style

Signature ID:

9FC8BD64-2186-4A97-88CC-D264914F8A6C

Using IP Address: 173.197.22.10

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

I approve this document

Electronic Record and Signature Disclosure: Accepted: 04-Sep-2024 | 16:58

ID: e1a5bfa5-34ac-47ef-af7d-11b59f1cd6cc

**Timestamp** 

Sent: 02-Sep-2024 | 16:33 Viewed: 03-Sep-2024 | 14:39 Signed: 03-Sep-2024 | 14:40

Sent: 02-Sep-2024 | 16:33

Viewed: 04-Sep-2024 | 16:58

Signed: 04-Sep-2024 | 16:58

| Signer Events | Signature | Timestamp |
|---|---|---|
| Julien Lucas | | Sent: 02-Sep-2024 16:33 |
| julien.lucas@aixial.com | Julien Lucas | Viewed: 02-Sep-2024 16:34 |
| Junior Statistician | | Signed: 09-Sep-2024 11:20 |
| Aixial Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: 1805EF25-9FF0-4719-80A6-4D0037F8D5D3 Using IP Address: 77.214.124.54 | |
| | With Signing Authentication via DocuSign passwor | d |
| | With Signing Reasons (on each tab): | |
| | I approve this document | |
| | I approve this document | |
| Electronic Record and Signature Disclosure: | | |

Accepted: 02-Sep-2024 | 16:34 ID: 14a3857a-35d7-4e97-a763-99d17ff61b10

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Natary Frants | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| , | _ | · |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | Timestamps 02-Sep-2024 16:33 |
| Envelope Summary Events Envelope Sent Certified Delivered | Status Hashed/Encrypted Security Checked | Timestamps 02-Sep-2024 16:33 02-Sep-2024 16:34 |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Status Hashed/Encrypted Security Checked Security Checked | Timestamps 02-Sep-2024 16:33 02-Sep-2024 16:34 09-Sep-2024 11:20 |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Cmed (Clinical Research Services) Limited (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Cmed (Clinical Research Services) Limited:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: dataprivacy@cmedresearch.com

#### To advise Cmed (Clinical Research Services) Limited of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at dataprivacy@cmedresearch.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Cmed (Clinical Research Services) Limited

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Cmed (Clinical Research Services) Limited

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

 decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Cmed (Clinical Research Services) Limited as described
  above, you consent to receive exclusively through electronic means all notices,
  disclosures, authorizations, acknowledgements, and other documents that are required to
  be provided or made available to you by Cmed (Clinical Research Services) Limited
  during the course of your relationship with Cmed (Clinical Research Services) Limited.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Ongoing medications are considered as concomitant medications.

The number and percentage of patients with prior and concomitant medications will be tabulated by basket and overall, by Anatomical Therapeutic Chemical Classification (ATC) and preferred term (PT) on the FAS. A by-patient listing will be produced for prior and concomitant medications as well as for all prior therapies.

On treatment Radiation, Surgery and Medical Procedures, and Blood Transfusions:

On treatment Radiation, Surgery and Medical Procedures, and Blood Transfusions will be listed on the FAS.

#### 9.6 STUDY DRUG EXPOSURE AND/OR COMPLIANCE

Duration on treatment and cumulative dose received will be calculated for both ulixertinib and hydroychloroquine as defined below with the same tables and listings.

- Number of cycles received =
   Number of cycles where the patient received at least one dose.
- Duration of exposure (months) =
  [(Date of last known treatment dosing with study treatment date of initial dosing with ulixertinib) + 1] / 30.4375
- Planned cumulative dose (mg) =
   Number of cycles received x number of doses per day x mg prescribed per dose.
- Actual cumulative dose received (mg) =
   For each time period reported in the eCRF:
   (Stop date Start date + 1)\*Dose
   Sum all available periods where dose was given.
- Relative dose intensity =

100 x Actual dose intensity / Planned dose intensity, with:

- Actual dose intensity (mg/day) = Actual cumulative dose received (mg) / Duration of exposure (days).
- Planned dose intensity (mg/day) = Planned cumulative dose (mg) / Duration of exposure (days).

Summary statistics will be presented for the number of cycles received, duration of exposure, actual cumulative dose, and relative dose intensity, by basket and overall on the FAS.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

The number and percentage of patients having at least one dosing interruption or adjustment will be tabulated with the corresponding reason by basket and overall on the FAS. A by-patient listing will be produced.

#### 9.7 PHARMACOKINETIC/ PHARMACODYNAMIC ENDPOINTS AND ANALYSES

#### 9.7.1 Pharmacokinetic Data

For patients enrolled in stage 1 of each basket, PK concentrations of ulixertinib and hydroxychloroquine will be determined pre-dose and post-dose in plasma at cycle 1 day 15. Summary parameters such as AUC, Cmax, Cmin, t1/2, tmax will be calculated.

PK parameters in plasma will be tabulated and summarized, by basket, using descriptive statistics (e.g., sample size, arithmetic and geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum).

For patients enrolled in stage 2 of each basket, PK concentration of ulixertinib will be measured on cycle 1 day 15. This will be a single timepoint collection prior to taking study drug on this day.

PK values will be presented in by-patient listings.

PK analysis will be conducted on the PK analysis set.

#### 9.7.2 Pharmacodynamic Data

Not applicable.

#### 9.8 EFFICACY DATA ENDPOINTS AND ANALYSES

#### 9.8.1 Primary Efficacy

#### 9.8.1.1 Overall Response Rate (ORR)

Tumor response will be assessed by the Investigator using RECIST 1.1 criteria1.

Disease assessments must include all known or suspected sites of disease; therefore, the decision for body areas to be scanned will depend on the extent of disease. The minimum recommended body areas to be scanned is chest, abdomen, and pelvis.

Disease assessments will be evaluated radiologically and conducted at baseline (within 28 days prior to the first dose of study treatment) and then every 8 weeks thereafter  $\leq$  7 days prior to the start of the following cycle (e.g., prior to cycle 3 day one, cycle 5 day 1, cycle 7 day 1, etc.). If a response is observed (CR or PR), confirmation of response is required  $\geq$  4 weeks from the first documentation of response. Disease assessments will continue until disease progression, the



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

initiation of subsequent anti-cancer therapy, or death. In addition, radiological tumor assessments will be conducted whenever disease progression is suspected (e.g., symptomatic deterioration) or when clinically indicated. The schedule of tumor assessments should be fixed according to the calendar, starting with cycle one day one, regardless of treatment delays or interruptions due to toxicity.

Brain CT or MRI scans are required at baseline for all patients with stable brain lesions and for those for whom Central Nervous System (CNS) involvement is suspected. If stable brain metastases are present at baseline, brain imaging should be repeated at each tumor assessment. Otherwise, brain imaging will be conducted post-baseline only when clinically indicated.

The table below provides a summary of the overall response status determination at each time point.

**Table 5. Evaluation of Overall Response** 

| Target lesions | Non-target lesions | New lesions | Overall response |
|---|---|---|---|
| CR | CR (or no non-target lesions) | No | CR |
| No target lesion a | CR | No | CR |
| CR | NE b | No | PR |
| CR | Non-CR/non-PD | No | PR |
| PR | Non-PD and NE (or no non-target lesions) b | No | PR |
| SD | Non-PD and NE (or no non-target lesions) b | No | SD |
| Not all evaluated | Non-PD | No | NE |
| No target lesion a | Not all evaluated | No | NE |
| No target lesion a | Non-CR/non-PD | No | Non-CR/non-PD |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |
| No target lesion a | Unequivocal PD | Yes or No | PD |
| No target lesion a | Any | Yes | PD |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, and NE = not evaluable

The ORR is defined as the number of patients having a confirmed response of either CR or PR divided by the total number of patients in the FAS/EAS. ORR will be calculated with the 95% confidence intervals (CIs), by basket and overall on the FAS and EAS. The 95% CIs will be estimated using the Clopper-Pearson method.

Complete and partial response must be confirmed by a repeat assessment performed ≥ 4 weeks after the criteria for response are first met. Date of confirmed CR/PR will be the date of the first CR/PR that qualifies for confirmation. Additionally, patients with no post-baseline efficacy measurement due to reasons accountable for disease progression, will be assessed as non-evaluable and will count in the denominator of the ORR.

Defined as no target lesion at baseline.

<sup>&</sup>lt;sup>b</sup> Not evaluable is defined as when either no or only a subset of lesion measurements is made at an assessment.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BOR will be assessed based on the tumor response at different evaluation time points from baseline until the first documented disease progression for RECIST or the last response assessment if there is no documented disease progression at the time of the analysis. The order used to determine BOR is CR>PR>SD>PD, ignoring visits with missing tumor assessments. For SD to qualify for BOR, the SD assessment should be at least 6 weeks after first ulixertinib dose. BOR date in this case will be the date of the first SD/PR/CR documented after 6 weeks.

The following table, based on Table 3 from the RECIST 1.1 guidelines<sup>1</sup>, summarizes the algorithm describing how confirmed response and BOR are determined from the overall tumor assessments.

Table 6. Evaluation of Confirmed BOR

| | Overall | Overall response | |
|---|---|---|---|
| | response | subsequent | |
| Case | first timepoint | timepoint | Confirmed response/BOR |
| 1 | CR | CR | CR (if assessments at least 28 days apart). (note: sequence of CR – |
| | | | NE – CR would be considered as confirmed CR) |
| 2 | CR | PR | SD, PD, or PR |
| | | | If CR truly met at first timepoint, any subsequent assessment |
| | | | of PR should make the disease PD at that point. That is, |
| | | | neither a PR nor SD may follow CR. |
| | | | Therefore, SD, if CR assessment >=6 weeks (42 days after date) |
| | | | of first treatment), otherwise PD. |
| | | | However, BOR may be PR if subsequent scans suggest small |
| | | | lesions were still present at first assessment (in which case |
| | | | first assessment of CR should be changed to PR) |
| 3 | CR | SD | SD or PD |
| | | | <ul> <li>SD, if CR or SD assessment &gt;=6 weeks (42 days) after date of</li> </ul> |
| | | | first treatment, |
| | | | otherwise PD |
| 4 | CR | PD | SD or PD |
| | | | SD, if CR assessment >=6 weeks (42 days after date of first |
| | | | treatment), |
| 5 | CD. | NE | otherwise PD |
| 5 | CR | NE | SD or NE |
| | | | <ul> <li>SD, if CR assessment &gt;=6 weeks (42 days after date of first<br/>treatment</li> </ul> |
| | | | otherwise NE |
| 6 | PR | CR | PR (if assessments at least 28 days apart). |
| 7 | PR | PR | PR (if assessments at least 28 days apart). PR (if assessments at least 28 days apart). (note: sequence of PR — |
| ľ | 1 | ' N | NE – PR would be considered as confirmed PR) |
| | | | Where there are cases of more than one SD assessment between |
| | | | two PR assessments, then this should be discussed. |
| 8 | PR | SD | SD |
| 9 | PR | PD | SD or PD |
| | | | SD, if PR assessment >=6 weeks (42 days after date of first |
| | | | treatment), |
| | | | otherwise PD |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| 6 | Overall response | Overall response subsequent | Confirmed account (DOD |
|---|---|---|---|
| Case | | timepoint | Confirmed response/BOR |
| 10 | PR | NE | SD or NE SD, if PR assessment >= 6 weeks (42 days after date of first treatment), otherwise NE |
| 11 | SD | SD, PR, CR | SD |
| 12 | SD | PD | SD or PD SD, if SD assessment >=6 weeks (42 days after date of first treatment), otherwise PD |
| 13 | SD | NE | SD or NE SD, if SD assessment >= 6 weeks (42 days after date of first treatment), otherwise NE |
| 14 | NE, - | SD | SD |
| 15 | CR, PR, SD | - | SD or NE SD, if assessment >=6 weeks (42 days after date of first treatment) and does not qualify for CR or PR, otherwise NE. |
| 16 | PD | | PD. Ignore all assessments after initial overall response of PD. |
| 17 | NE | NE | NE<br>Where all assessments are Not evaluable |

For changes in target tumor size, spider and waterfall plots will be presented. For all response assessments, swimmer plots will be presented. Target and Non-Target Lesions response assessments and incidence of new lesions will be summarized by visit and listed. All response assessments will be listed.

#### 9.8.2 Secondary Efficacy

#### **9.8.2.1** Progression-free Survival (PFS)

The PFS (in months) is defined as the time from the first ulixertinib dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

PFS = [(Date of first PD/death - Date of first study treatment) + 1] / 30.4375

Patients with no documented progression or death will be censored at the last available tumor assessment (last assessment that is CR, PR or SD):

PFS = [(Date of last assessment where patient is PD free – Date of first study treatment) + 1] / 30.4375



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

For patients with no post baseline tumor assessment a censored PFS at day 1 will be considered.

PFS = (Date of first study treatment - Date of first study treatment) + 1

The analysis of PFS will be performed with a Kaplan-Meier method (product-limit estimates) and a summary of associated statistics will be presented including corresponding two-sided 95% CI. The CI for the median will be calculated according to Brookmeyer and Crowley and CI for the survival function estimates at Month 3, 6, 9, 12, and 18 will be derived using the log-log transformation (SAS PROC LIFETEST CONFTYPE=LOGLOG). However, the final choice of timepoints may be updated dependent upon the data.

#### 9.8.3 Exploratory Efficacy

#### 9.8.3.1 Duration of Response (DOR)

The DOR (in months) is defined as the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause. Only patients with BOR of CR or PR (i.e. responders) will be included in the analysis of DOR.

DOR = [(Date of first PD/death - Date of first recorded confirmed CR/PR) + 1] / 30.4375

Patients with no documented progression or death after CR or PR will be censored at the last available tumor assessment (last assessment that is CR, PR, or SD):

DOR = [(Date of last assessment where patient is PD free – Date of first recorded CR/PR) + 1] / 30.4375

The analysis of DOR will be performed with a Kaplan-Meier method (product-limit estimates) and a summary of associated statistics will be presented including corresponding two-sided 95% CI. The CI for the median will be calculated according to Brookmeyer and Crowley and CI for the survival function estimates at Month 3, 6, 9, 12, and 18 will be derived using the log-log transformation (SAS PROC LIFETEST CONFTYPE=LOGLOG), only if there are sufficient data for responders. However, the final choice of timepoints may be updated dependent upon the data.

#### 9.8.3.2 Overall Survival (OS)

The OS (in months) is defined as the time from first treatment to death. Patients who did not die during the study will be censored at the last known alive date.

OS = [(Date of death – Date of first study treatment) + 1] / 30.4375

For censored patients:



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

OS = [(Last known alive date - Date of first study treatment) + 1] / 30.4375

The last known alive date will be determined among study treatment administrations, any visits where at least one assessment has been completed, or any follow-up assessment where the patient has been confirmed to be alive.

OS will be analyzed using the same Kaplan-Meier method used to analyze the DOR.

#### 9.9 SAFETY DATA ENDPOINTS AND ANALYSES

All safety analyses will be performed by basket and overall on the FAS, using descriptive statistics.

#### 9.9.1 Adverse Events (AEs)

The following definitions will be used:

- Treatment-emergent AEs (TEAEs): Treatment-emergent adverse event (TEAE) is defined
  as any AE that emerges during on-treatment period.
- Related AEs: AEs suspected by the Investigator and/or Sponsor to have a relationship to study treatment (as recorded on the AE eCRF page, Causality = Related, Possibly Related, or missing), including ulixertinib or hydroxychloroquine or both.
- Serious Adverse Events (SAE): serious AEs (as recorded on the AE eCRF page, Does AE Meet the Definition of an SAE = Yes).
- AEs leading to treatment discontinuation: AEs leading to permanent discontinuation of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Drug withdrawn).
- AEs leading to dose reduction: AEs leading to dose reduction of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Dose Reduced).
- AEs leading to treatment interruption: AEs leading to treatment interruption of study treatment (as recorded on the AE eCRF page, Action taken with study treatment = Drug Interrupted).
- AEs leading to Death: adverse event leading to death (as recorded on the AE eCRF page, Results in death, or Outcome = Fatal, or Grade = 5).

An overview summary table will present the number and percentage of patients with a TEAE, all treatment-related adverse events will be indicated as Ulixertinib-related or Hydroxychloroquine-related or both, including:

- TEAEs / TEAEs related to study treatment
- SAEs / SAEs related to study treatment
- TEAEs leading to treatment discontinuation / TEAEs related to study treatment leading to treatment discontinuation



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

- TEAEs leading to treatment discontinuation within 1 cycle / TEAEs related to study treatment leading to treatment discontinuation within 1 cycle
- TEAEs leading to treatment discontinuation following 1 cycle / TEAEs related to study treatment leading to treatment discontinuation following 1 cycle
- TEAEs leading to treatment interruption / TEAEs related to study treatment leading to treatment interruption
- TEAEs leading to treatment interruption within 1 cycle / TEAEs related to study treatment leading to treatment interruption within 1 cycle
- TEAEs leading to treatment interruption following 1 cycle / TEAEs related to study treatment leading to treatment interruption following 1 cycle
- TEAEs leading to dose reduction / TEAEs related to study treatment leading to dose reduction
- TEAEs leading to dose reduction within 1 cycle / TEAEs related to study treatment leading to dose reduction within cycle 1
- TEAEs leading to dose reduction following 1 cycle / TEAEs related to study treatment leading to dose reduction following cycle 1
- TEAEs leading to death / TEAEs related to study treatment leading to death
- TEAEs with grade ≥ 3 / TEAEs related to study treatment with grade ≥ 3

In addition, the following tables will be produced by SOC and PT:

- TEAEs / TEAEs related to study treatment
- Serious TEAEs / Serious TEAEs related to study treatment
- TEAEs and maximum CTCAE grade / TEAEs related to study treatment and maximum CTCAE grade
- TEAEs leading to treatment discontinuation within/following cycle 1 / TEAEs related to study treatment leading to treatment discontinuation within/following cycle 1
- TEAEs leading to treatment interruption within/following cycle 1 / TEAEs related to study treatment leading to treatment interruption within/following cycle 1
- TEAEs leading to dose reduction within/following cycle 1 / TEAEs related to study treatment leading to dose reduction within/following cycle 1
- TEAEs leading to death / TEAEs related to study treatment leading to death

The following tables will be produced by PT:

- TEAEs / TEAEs related to study treatment
- Serious TEAEs / Serious TEAEs related to study treatment

A patient with multiple occurrences of an AE will be counted only once in the AE category. SOCs will be sorted by descending order of frequency for the overall group, PTs will be sorted by descending order of frequency for the overall group within each SOC.

All deaths will be summarized and listed with the corresponding reasons, split by overall deaths, and deaths occurring after the first dose of ulixertinib.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

The following listings will be provided:

- All AEs (All Patient Set)
- TEAEs (FAS)
- SAEs (FAS)
- Deaths (FAS)

#### 9.9.2 Clinical Safety Laboratory Evaluation

All haematology, biochemistry, coagulation and urinalysis laboratory tests collected will be reported.

The numerical measurements and change from baseline of all haematology, biochemistry, and urinalysis laboratory tests will be summarized using descriptive summary statistics for each visit.

For laboratory tests covered by the NCI-CTCAE (version 5), laboratory data will be graded accordingly. 'Normal' will be assigned for all non-missing values not graded as 1 or higher. For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classifications based on laboratory normal ranges as collected in the CRF. Separate tables will be created for Gradable and Non-gradable laboratory values.

Haematology and biochemistry laboratory tests will be summarized by:

- Tables (Gradable and Non-gradable) to describe the worst on-treatment value by cycle.
- Shift tables (Gradable and Non-gradable) to compare baseline to the worst on-treatment value.

Listings of all laboratory data with values flagged to show the corresponding NCI-CTCAE grades and the classifications relative to the laboratory normal ranges will also be provided. Also results of serum pregnancy tests and tumor markers will be listed.

#### 9.9.3 Other Safety data

#### **9.9.3.1** Vital signs

Vital signs include the following parameters: systolic blood pressure (SBP) (mmHg), diastolic blood pressure (DBP) (mmHg), pulse (beats/min), respiratory rate (breaths/min), pulse oximetry (%) and temperature (°C).

The numerical measurements and change from baseline of all vital signs parameters will be summarized using descriptive summary statistics for each visit.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Shift tables of baseline to worst on-treatment result (low, normal, high, very high) will be presented.

Table 7. Thresholds for classification of vital signs test results

| Vital Sign | Criteria | Flag |
|------------------|-------------------|-----------|
| Temperature | < 36.4°C | Low |
| | 36.4°C - 37.7°C | Normal |
| | > 37.7°C | High |
| Pulse | < 55 bpm | Low |
| | 55-100 bpm | Normal |
| | 101-150 bpm | High |
| | > 150 bpm | Very High |
| Respiratory rate | <12 breaths/min | Low |
| | 12-16 breaths/min | Normal |
| | >16 breaths/min | High |
| Pulse oximetry | <90 % | Very Low |
| | 90-95 % | Low |
| | ≥95 % | Normal |
| Systolic Blood | < 90 mmHg | Low |
| Pressure | 90-130 mmHg | Normal |
| | 131-160 mmHg | High |
| | ≥161 mmHg | Very High |
| Diastolic Blood | < 60 mmHg | Low |
| Pressure | 60-85 mmHg | Normal |
| | 86-100 mmHg | High |
| | ≥ 101 mmHg | Very High |

All Vital Signs will be Listed.

#### 9.9.3.2 Electrocardiogram (ECG)

ECG includes the following parameters: Heart Rate (beats/min), PR Interval (msec), QRS Duration (msec), RR Interval (msec), QT Interval (msec), and QT interval corrected for heart rate by the Fridericia's formula (QTcF) Interval (msec).

The numerical measurements and change from baseline of all ECG parameters will be summarized using descriptive summary statistics for each visit.

A listing of ECG evaluations will be created.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### 9.9.3.3 ECHO

ECHO assessments at baseline will be summarized using descriptive summary statistics.

A listing of ECHO evaluations will be created.

#### 9.9.3.4 Physical Examination

Physical Examination includes the following parameters: HEENT, Thorax, Abdomen, Skin and Mucosae, Neurological, Extremities, Urogenital, General Appearance, Heart, Back, and Lymph Nodes.

All physical examination assessments at baseline will be summarized using descriptive summary statistics.

A listing of physical examination evaluations will be created.

#### 9.9.3.5 Ophthalmology exam

A listing of ophthalmological examination assessments will be created.

#### 9.9.3.6 ECOG Performance status

The number and percentages of patients will be tabulated for ECOG performance score categories at each visit.

A listing of all ECOG Performance status at all visits will be presented.

## 10 Interim Analyses

No interim analysis is planned.

# 11 Changes to Planned Analyses

No major changes to analyses planned in the protocol are expected.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 12 Document History

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 17Jul2023 | 1.0 | David Manteigas | First SAP Version. |
| 20-Aug-2024 | 1.1 | Julien Lucas | Updated version to include required changes after the study was terminated early. |
| 02-Sep-2024 | 2.0 | Julien Lucas | Second SAP version. |

## 13 References

 Eisenhauer EA, Therasse P, Bogaerts J, et al. (2009), New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer; 45:228-47.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# 14 Appendices

## 14.1 Schedule of events

| | | | On-Trea | tment Period | : One Cycle | = 28 days | | Pos | t-Treatment P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | cle 2 | Cycle 3+ | EOT" | Safety<br>Follow-<br>Up <sup>Ⅲ</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1™ | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| Informed Consent | х | | | | | | | | | |
| Demographics | х | | | | | | | | | |
| Cancer History <sup>v</sup> | х | | | | | | | | | |
| Medical History | х | | | | | | | | | |
| Eligibility Criteria | х | | | | | | | | | |
| Clinical Assessments | | | | | | | | | | |
| Vital Signs <sup>vl</sup> | Х | X | X | X | X | X | X | X | X | |
| Physical Exam <sup>vll</sup> | Х | Х | х | X | X | X | X | X | X | |
| ECOG Score | Х | Х | х | X | X | X | X | X | X | |
| ECG | х | | x | X | x | | | X | | |
| Echocardiogram | Х | | ACI | | | | | | | |



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

| | | | On-Trea | tment Period | l: One Cycle | = 28 days | | Pos | st-Treatment P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | cle 2 | Cycle 3+ | EOTII | Safety<br>Follow-<br>Up <sup>™</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1₩ | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| Ophthalmologic Exam <sup>vill</sup> | Х | | | | X | | X | | | |
| Adverse event collection | Х | | | | | X | | | _ | |
| Concomitant medications | Х | | | | X | | | | | |
| Laboratory Studies <sup>lx</sup> | | | | | | | | | | |
| Hematology | х | X | x | x | x | x | X | X | X | |
| Chemistry | Х | Х | X | X | X | X | X | X | X | |
| Creatine kinase <sup>x</sup> | х | | | Α | CI | | | | | |
| LDH and Phosphorus | х | х | x | х | x | Α | CI | | | |
| Coagulation | Х | | | A | CI | | | | | |
| Urinalysis | Х | | ACI | | | | | | | |
| Tumor Marker <sup>xl</sup> | | Х | | | X | | X | X | | |
| Pregnancy Test <sup>xli</sup> | х | ACI | | | | | | | | |
| Disease Assessments | | | | | | | | | | |
| CT Scans or MRIXII | Х | | | | | | X | х | | Xxiv |



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

| | | | On-Trea | tment Period | : One Cycle | = 28 days | | Pos | t-Treatment P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities | Screening | | Cycle 1 | | Сус | ile 2 | Cycle 3+ | EOT" | Safety<br>Follow-<br>Up <sup>™</sup> | |
| Day of Cycle<br>(Visit Window) | (≤ -28 days) | 1₩ | 8<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | 15<br>(± 2 days) | 1<br>(± 2 days) | (+7 days) | (± 7 days) | Follow-Up |
| RECIST 1.1 Assessment | Х | | | | | | Х | X | | Х |
| Treatment Compliance ar | nd Distribution | | | | | | | | | |
| Hydroxychloroquine | | X | | | X | | х | | | |
| Ulixertinib | | X | | | X | | X | | | |
| Treatment administration on site | | | | X <sup>15</sup> | | | x | | | |
| Meal provided by site | 4 44 . 4. | | | Х | | | X16 | | | |

Abbreviations: ACI = as clinically indicated; LDH = lactate dehydrogenase; CT = computed tomography; MRI = magnetic resonance imaging; ECG = electrocardiogram; EOT = end of treatment



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

¹ Screening procedures must be completed ≤ 28 days prior to C1D1 unless noted otherwise.

- <sup>2</sup> The end of treatment visit should occur when the decision to discontinue treatment is made. If this visit overlaps with a regularly scheduled visit, only the procedures listed in the calendar for the EOT visit will be performed. All end of treatment procedures should be completed within 7 days after the decision to discontinue treatment has been made.
- 3 Patients will have a safety follow-up visit 60 days (± 7 days) after last dose of study drug.
- 4 C1D1 procedures do not need to be repeated if screening procedures were performed ≤ 7 days of the start of treatment.
- <sup>5</sup> Oncologic history of the malignancy under study including prior regimens (duration of therapy, best response on therapy, date of discontinuation, and reason for discontinuation), surgery, and radiation therapy.
- <sup>6</sup> Vital signs include systolic/diastolic blood pressure, heart rate, respiration rate, pulse oximetry, weight, and body temperature. Height will be captured at screening only.
- 7 If necessary to facilitate scheduling, the physical exam may occur one day prior to study treatment.
- <sup>8</sup> A standard ophthalmologic exam must be completed at screening, C2D1, and every 3 cycles thereafter (i.e. C5D1, C8D1, etc.) and as clinically indicated to assess for retinopathies. All assessments must be conducted up to 7 days prior to the clinic visit to enable timely results review.
- <sup>9</sup> Labs may be performed ≤ 3 days prior to a scheduled day one visit except for C1D1 labs which may be completed ≤ 7 days prior to C1D1.
- 10 After screening, creatine kinase should only be drawn if creatinine is elevated.
- <sup>11</sup> Tumor marker should be drawn on day one of each cycle. Tumor markers will be disease specific: pancreatic adenocarcinoma only CA 19-9; colorectal carcinoma only CEA; cholangiocarcinoma only CEA and CA 19-9. Tumor markers are not required for patients with esophageal or stomach cancers.
- <sup>12</sup> Pregnancy test (serum or urine) must be obtained at screening ≤ 7 days prior to C1D1 for all women of childbearing potential and as clinically indicated while on treatment.
- <sup>13</sup> Disease assessment will be repeated every 8 weeks (± 7 days) regardless of dose holds or delays. Patients who discontinue treatment for reasons other than progression will have computed tomography (CT) scans at the EOT visit (unless their previous restaging was performed within 6 weeks).
- 14 Patients that discontinue study treatment for any reason other than disease progression, must continue to have disease assessments every 8 weeks (± 7 days) until disease progression or initiation of subsequent anticancer therapy.
- 15 Patient should be instructed to not take their study treatment before arriving at clinic. Study treatment and meal should be provided after the pre-dose PK draw.
- 16 Meal is only required to be given at C3D1, i.e., at the time of drug administration for ctDNA and tumor biopsy for stage 1.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

#### 14.2 Schedule of Correlative Sample Collection

| | | | . C1D15 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Correlative<br>Test | | | Pre-<br>Dose | | | ı | Post-D | ose | | | C3D1 | EOT |
| Time Point<br>(hour) | Screening | C1D1 | | 0.5 | 1 | 2 | 4 | 6 | 8 | 12 | ± 7 | |
| Window (min) | | | ≤ 60 | ±2 | ±3 | ±6 | ±12 | ±18 | ±24 | ±36 | days | |
| | | | | STA | GE 1 | | | | | | | |
| PK Blood <sup>1</sup> | | | X | X | Х | Х | Х | Х | Х | X | | |
| ctDNA | | X | | | | | | | | | X <sup>2</sup> | X <sup>3</sup> |
| Biopsy | X | | | | | | | | | | X | X |
| | STAGE 2 | | | | | | | | | | | |
| PK Blood <sup>4</sup> | | | Х | | | | | | | | | |

Abbreviations: C = cycle; ctDNA = circulating tumor DNA; D = day; EOT = end of treatment; PK = pharmacokinetics.

<sup>&</sup>lt;sup>1</sup>To accommodate PK blood draws, patients should be instructed not to take their morning doses of both medications until told to do so in the clinic. A meal should be provided by the site when taking the medications in the clinic. Pre-dose PK sample should be collected prior to the administration of study drugs. Post-dose PK samples should be collected at the appropriate time points following administration of study drugs. PK samples should be drawn while patients are at steady state, which is 5 days, or 10 consecutive doses.

<sup>&</sup>lt;sup>2</sup>To be drawn at the time of the tumor biopsy.

<sup>&</sup>lt;sup>3</sup>Required blood draw at EOT. If optional biopsy is collected at EOT, ctDNA should be drawn at the time of the tumor biopsy.

<sup>&</sup>lt;sup>4</sup>Biopsies at screening and C3D1 (± 7 days) are required. When blood is being drawn at D3D1, site will provide a meal when study drugs are taken. An optional biopsy will be offered at the time when the decision to discontinue treatment is made (+ 7 days).



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

## 14.3 CTCAE v5.0 Grading for Laboratory Values

**Table 8. Hematology Tests** 

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Hematocrit | No | | |
| Hemoglobin | Yes | Blood and lymphatic<br>system disorders | Anemia |
| | | Investigations | Hemoglobin increased |
| Platelets | Yes | Investigations | Platelet count decreased |
| White blood cells | Yes | Investigations | White blood cell decreased |
| | | Blood and lymphatic<br>system disorders | Leukocytosis |
| Neutrophils absolute | Yes | Investigations | Neutrophil count decreased |
| Lymphocytes absolute | Yes | Investigations | Lymphocyte count decreased |
| | | | Lymphocyte count increased |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 9. Coagulation Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|-----------|-----------------|----------------|-----------------|
| PT | No | | |
| INR | Yes | Investigations | INR increased |
| PTT | No | | |

<sup>†</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 10. Serum Chemistry Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Albumin | Yes | Metabolism and<br>nutrition disorders | Hypoalbuminemia |
| Alkaline phosphatase | Yes | Investigations | Alkaline phosphatase increased |
| ALT | Yes | Investigations | Alanine aminotransferase increased |
| AST | Yes | Investigations | Aspartate aminotransferase increased |
| Blood urea nitrogen | No | | |
| Uric acid | No | | |
| Chloride | No | | |
| Calcium | Yes | Metabolism and | Hypocalcemia |
| | | nutrition disorders | Hypocalcemia |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

1.0 / 27-Jul-2023

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Creatinine | Yes | Investigations | Creatinine increased |
| Lactate Dehydrogenase | Yes | Investigations | Lactate Dehydrogenase increased |
| Glucose | Yes | Metabolism and | Hyperglycemia |
| | | nutrition disorders | Hypoglycemia |
| Potassium | Yes | Metabolism and | Hyperkalemia |
| | | nutrition disorders | Hypokalemia |
| Sodium | Yes | Metabolism and | Hypernatremia |
| | | nutrition disorders | Hyponatremia |
| Inorganic Phosphorus | No | | |
| Total bilirubin | Yes | Investigations | Blood bilirubin increased |
| Direct bilirubin | No | | |
| Total protein | No | | |
| Urea Nitrogen | No | | |
| Carbon Dioxide | No | ĺ | Ì |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.

Table 11. Urinalysis Tests

| Parameter | CTCAE Gradable† | SOC | CTCAE v5.0 Term |
|---|---|---|---|
| Dipstick Evaluation Of | No | | |
| Bilirubin | | | |
| Dipstick Evaluation Of<br>Blood | No | | |
| Dipstick Evaluation Of<br>Glucose | No | | |
| Dipstick Evaluation Of<br>Ketones | No | | |
| Dipstick Evaluation Of<br>Leukocytes | No | | |
| Dipstick Evaluation Of<br>Protein | No | | |
| Microscopic<br>Examination Of Casts | No | | |
| Microscopic<br>Examination Of Rbc | No | | |
| Microscopic<br>Examination Of Wbc | No | | |
| pH | No | | |
| Specific Gravity | No | | |

<sup>+</sup> For laboratory tests where grades are not defined by NCI-CTCAE, results will be graded by the low/normal/high classification based on laboratory normal ranges.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# **SPONSOR:**

# **BioMed Valley Discoveries**

## PROTOCOL NUMBER:

BVD-523-HCQ

# STATISTICAL ANALYSIS PLAN TFL SHELLS

| Author: | Julien Lucas |
|----------|--------------|
| Version: | 2.0 |
| Date: | 02-Sep-2024 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## 1 Cover and signature pages

| Sponsor: | BioMed Valley Discoveries |
|---|---|
| Protocol Number: | BVD-523-HCQ |
| Study Title: | A phase 2 basket trial of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring MAPK pathway mutations (BVD-523-HCQ) |
| Document Version No | 1.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorize its approval.

#### Statistician

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|---|---|---|---|
| | Biostat III | | Signed by: Julium (mas Signer Name: Julien Lucas Signing Reason: I approve this document Signing Time: 09-Sep-2024 11:20 BST 1805EF259FF0471980A64D0037F8D5D3 |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### **Client Representative**

| Name | Title [text box when using eSignatures]: | Date | Signature |
|---|---|---|---|
| | Senior Scientist | | Signed by: Assec Alexand Signer Name: Anna Groover Signing Reason: I approve this document Signing Time: 03-Sep-2024 08:40 CDT 71380BDD08BC4D289E63FA3831CD4243 |
| | President | | Signed by: Brent Kreides Signer Name: Brent Kreider Signing Reason: I approve this document Signing Time: 04-Sep-2024 08:58 PDT 9FC8BD6421864A9788CCD264914F8A6C |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# 2 Document History

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 27Jul2023 | 1.0 | David Manteigas | First SAP version |
| 20Aug2024 | 1.1 | Julien Lucas | Updated version to include required changes after the study was early terminated. |
| 02Sep2024 | 2.0 | Julien Lucas | Second SAP version. |

# 3 List of Tables, Figures and Listings

| TFL | TFL | Title | Population | SMC* | Included |
|---|---|---|---|---|---|
| Type | Number | | | | in Final |
| | | | | | Analysis |
| 14.1 | | Demographic Data | | | |
| Table | 14.1-1.1 | Patient Disposition | All Patients Set | Y | Y |
| Table | 14.1-1.2 | Number of Patients in the Analysis Sets | All Patients Set | | Y |
| Table | 14.1-1.3 | Summary of Important Protocol Deviations | Full Analysis Set | | Y |
| Table | 14.1-2.1 | Demographics and Baseline Characteristics | Full Analysis Set | Y | Y |
| Table | 14.1-2.2 | Disease History | Full Analysis Set | Y | Y |
| Table | 14.1-2.3 | Summary of Medical History | Full Analysis Set | | Y |
| Table | 14.1-2.4 | Summary of Concomitant Diseases | Full Analysis Set | | Y |
| Table | 14.1-3.1 | Prior Systemic Anti-Cancer Therapies | Full Analysis Set | Y | Y |
| Table | 14.1-3.2 | Prior Radiotherapy Courses | Full Analysis Set | Υ | Y |
| Table | 14.1-3.3 | Prior Medications | Full Analysis Set | | Y |
| Table | 14.1-3.4 | Concomitant Medications | Full Analysis Set | | Y |
| Table | 14.1-4.1.1 | Treatment Exposure (Ulixertinib) | Full Analysis Set | Υ | Y |
| Table | 14.1-4.1.2 | Treatment Exposure (Hydroxychloroquine) | Full Analysis Set | Υ | Y |
| Table | 14.1-4.2.1 | Dosing Interruptions and Adjustments (Ulixertinib) | Full Analysis Set | Υ | Y |
| Table | 14.1-4.2.2 | Dosing Interruptions and Adjustments | Full Analysis Set | Y | Y |
| | | (Hydroxychloroquine) | | | |
| 14.2 | | Efficacy Data | | | |
| Table | 14.2-1.1.1 | Best Overall Response and Overall Response Rate | Full Analysis Set | | Y |
| Table | 14.2-1.1.2 | Best Overall Response and Overall Response Rate | Evaluable Analysis Set | | |
| Table | 14.2-1.2.1 | Overall, Target and Non-Target Lesion Response | Full Analysis Set | | Y |
| Table | 14.2-1.2.2 | Overall, Target and Non-Target Lesion Response | Evaluable Analysis Set | | |
| Table | 14.2-1.3.1 | Incidence of New Lesions | Full Analysis Set | | Y |
| Table | 14.2-1.3.2 | Incidence of New Lesions | Evaluable Analysis Set | | |
| Table | 14.2-1.4.1 | Progression-free Survival (PFS) | Full Analysis Set | | Y |
| Table | 14.2-1.4.2 | Progression-free Survival (PFS) | Evaluable Analysis Set | | |
| Table | 14.2-1.5.1 | Overall Survival (OS) | Full Analysis Set | | Y |
| Table | 14.2-1.5.2 | Overall Survival (OS) | Evaluable Analysis Set | | |
| Table | 14.2-1.6.1 | Duration of Response (DOR) | Full Analysis Set | | |
| 14.3 | | Safety Data | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| Table | 14.3-1.1 | Overview Summary of Treatment-Emergent Adverse Events | Full Analysis Set | Y | Y |
|---|---|---|---|---|---|
| Table | 14.3-1.2 | Summary of Treatment-Emergent Adverse Events by | Full Analysis Set | Y | Y |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.3 | Summary of Related Treatment-Emergent Adverse<br>Events by System Organ Class and Preferred Term | Full Analysis Set | Y | Y |
| Table | 14.3-1.4 | Summary of Serious Treatment-Emergent Adverse | Full Analysis Set | Υ | Y |
| Tubic | 14.5 1.4 | Events by System Organ Class and Preferred Term | Tall Allalysis Sec | Ι' | 1. |
| Table | 14215 | Summary of Related Serious Treatment-Emergent | Full Analysis Set | Y | Y |
| Table | 14.3-1.5 | | ruii Analysis set | 1' | 1 |
| | | Adverse Events by System Organ Class and Preferred | | | |
| | 44046 | Term | 5 11 4 1 1 5 5 1 | | |
| Table | 14.3-1.6 | Summary of Treatment-Emergent Adverse Events by | Full Analysis Set | | |
| | | Preferred Term | | | |
| Table | 14.3-1.7 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | |
| | | Events by Preferred Term | | | |
| Table | 14.3-1.8 | Summary of Serious Treatment-emergent Adverse | Full Analysis Set | | |
| | | Events by Preferred Term | | | |
| Table | 14.3-1.9 | Summary of Related Serious Treatment-emergent | Full Analysis Set | | |
| | | Adverse Events by Preferred Term | | | |
| Table | 14.3-1.10 | Summary of Treatment-Emergent Adverse Events by | Full Analysis Set | | Υ |
| | | System Organ Class and Preferred Term for Maximum | | | |
| | | CTCAE grade | | | |
| Table | 14.3-1.11 | Summary of Related Treatment-Emergent Adverse | Full Analysis Set | Υ | Y |
| | | Events by System Organ Class and Preferred Term for | | | |
| | | Maximum CTCAE grade | | | |
| Table | 14.3-1.12 | Summary of Treatment-emergent Adverse Leading to | Full Analysis Set | Y | Y |
| 10010 | 11.0 1.11 | Treatment Discontinuation Events by System Organ | Tan ranary sis sec | 1. | 1. |
| | | Class and Preferred Term | | | |
| Table | 14.3-1.13 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | Y | Y |
| Tubic | 14.5 1.15 | Events Leading to Treatment Discontinuation by | Tuli Analysis sec | 1' | Ι' |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.14 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | Y | Y |
| Table | 14.5-1.14 | _ | ruii Anaiysis set | 1' | ' |
| | | Leading to Treatment Discontinuation within Cycle 1 | | | |
| T-bl- | 142115 | by System Organ Class and Preferred Term | Full Applicate Coa | Y | v |
| Table | 14.3-1.15 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | Y | Y |
| | | Events Leading to Treatment Discontinuation within | | | |
| | | Cycle 1 by System Organ Class and Preferred Term | | <b>—</b> | |
| Table | 14.3-1.16 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | Υ | Y |
| | l | Leading to Treatment Discontinuation following Cycle | | | |
| | | 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.17 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | Υ | Y |
| | | Events Leading to Treatment Discontinuation following | | | |
| | | Cycle 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.18 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Treatment Interruption by System Organ | | | |
| | | Class and Preferred Term | | | |
| Table | 14.3-1.19 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Treatment Interruption by System | | | |
| | | Organ Class and Preferred Term | | | |
| Table | 14.3-1.20 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | Υ | Υ |
| | | Leading to Treatment Interruption within Cycle 1 by | | | |
| | l | System Organ Class and Preferred Term | | | |
| | | -, | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| Table | 14.3-1.21 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | Y | Y |
|---|---|---|---|---|---|
| | | Events Leading to Treatment Interruption within Cycle | | | |
| | | 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.22 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Treatment Interruption following Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.23 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Treatment Interruption following | | | |
| | | Cycle 1 by System Organ Class and Preferred Term | | | |
| Table | 14.3-1.24 | Summary of Treatment-emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Dose Reduction by System Organ Class and | | | |
| | | Preferred Term | | | |
| Table | 14.3-1.25 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Dose Reduction by System Organ | | | |
| | | Class and Preferred Term | | | |
| Table | 14.3-1.26 | Summary of Treatment-Emergent Adverse Events | Full Analysis Set | Y | Y |
| | | Leading to Dose Reduction within Cycle 1 by System | | | |
| | | Organ Class and Preferred Term | | | |
| Table | 14.3-1.27 | Summary of Related Treatment-Emergent Adverse | Full Analysis Set | Y | Y |
| | | Events Leading to Dose Reduction within Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.28 | Summary of Treatment-Emergent Adverse Events | Full Analysis Set | | Y |
| | | Leading to Dose Reduction following Cycle 1 by System | | | |
| | | Organ Class and Preferred Term | | | |
| Table | 14.3-1.29 | Summary of Related Treatment-Emergent Adverse | Full Analysis Set | | Y |
| | | Events Leading to Dose Reduction following Cycle 1 by | | | |
| | | System Organ Class and Preferred Term | | | |
| Table | 14.3-1.30 | Summary of Treatment-emergent Adverse Events by | Full Analysis Set | | Y |
| | | System Organ Class and Preferred Term Leading to | | | |
| | | Death | | | |
| Table | 14.3-1.31 | Summary of Related Treatment-emergent Adverse | Full Analysis Set | | Y |
| | | Events by System Organ Class and Preferred Term | | | |
| | | Leading to Death | | | |
| Table | 14.3-1.32 | Summary of Deaths | All Patients Set | Y | Y |
| Table | 14.3-2.1 | Summary and Change from Baseline in Hematology | Full Analysis Set | | Y |
| | | Laboratory Results by Visit | | | |
| Table | 14.3-2.2.1 | Gradable Hematology Laboratory Results - Worst On- | Full Analysis Set | | |
| | | treatment Value by Cycle | | | |
| Table | 14.3-2.2.2 | Non-gradable Hematology Laboratory Results – Worst | Full Analysis Set | | |
| | | On-treatment Value by Cycle | | | |
| Table | 14.3-2.3.1 | Shift Table of Gradable Hematology Laboratory Results | Full Analysis Set | Y | Y |
| | | – Baseline vs Worst On-treatment Value | | | |
| Table | 14.3-2.3.2 | Shift Table of Non-gradable Hematology Laboratory | Full Analysis Set | | Y |
| | | Results – Baseline vs Worst On-treatment Value | | | |
| Table | 14.3-2.4 | Summary and Change from Baseline in Biochemistry | Full Analysis Set | | Y |
| | l —— | Laboratory Results by Visit | | | |
| | | Gradable Biochemistry Laboratory Results – Worst On- | Full Analysis Set | | |
| Table | 14.3-2.5.1 | Gradable blochemistry Laboratory Results – Worst Oil- | | | 1 |
| Table | 14.3-2.5.1 | treatment Value by Cycle | | | |
| Table<br>Table | | | Full Analysis Set | + | |
| | 14.3-2.5.1<br>14.3-2.5.2 | treatment Value by Cycle | Full Analysis Set | | |
| | | treatment Value by Cycle Non-gradable Biochemistry Laboratory Results — | Full Analysis Set | Y | Y |


Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| | | | T | т — | T |
|---|---|---|---|---|---|
| Table | 14.3-2.6.2 | Shift Table of Non-gradable Biochemistry Laboratory Results – Baseline vs Worst On-treatment Value | Full Analysis Set | | Y |
| T-bl- | 14227 | | Full Applicate Con | <del> </del> | Y |
| Table | <u>14.3-2.7</u> | Summary at Baseline in Coagulation Laboratory<br>Results by Visit | Full Analysis Set | | T |
| Table | 14.3-2.8 | Summary at Baseline in Urinalysis Laboratory Results<br>by Visit | Full Analysis Set | | |
| Table | <u>14.3-3.1</u> | Summary and Change from Baseline in Vital Signs by<br>Visit | Full Analysis Set | | Y |
| Table | 14.3-3.2 | Shift table of Vital Signs – Baseline vs worst on-<br>treatment value | Full Analysis Set | | Υ |
| Table | 14.3-3.3 | Summary and Change from Baseline in ECG parameters by Visit | Full Analysis Set | Y | Y |
| Table | 14.3-3.4 | Summary of ECHO at Baseline | Full Analysis Set | <del> </del> | |
| Table | 14.3-3.5 | Summary of Physical Examination at Baseline | Full Analysis Set | | |
| Table | 14.3-3.6 | Summary of ECOG Performance Status by Visit | Full Analysis Set | Υ | |
| 14.4 | | Other Efficacy Data | | | |
| 14.5 | | Pharmacokinetic Data | | | |
| Table | 14.5-1.1 | Pharmacokinetic Concentration Data | PK Analysis Set | | Υ |
| Table | 14.5-1.2 | Pharmacokinetic Parameters Data | PK Analysis Set | <u> </u> | Υ |
| 14.2 | | Figures | | | |
| Figure | 14.2-1.1 | Consort Diagram | Full Analysis Set | Υ | Υ |
| Figure | 14.2-1.2.1 | Spider plot of Percentage Change from Baseline in<br>Sum of Longest Diameter | Full Analysis Set | | Y |
| Figure | 14.2-1.2.2 | Spider plot of Percentage Change from Baseline in<br>Sum of Longest Diameter | Evaluable Analysis Set | | |
| Figure | 14.2-1.3.1 | Waterfall plot of Maximum Percentage Change from<br>Baseline in Sum of Longest Diameter | Full Analysis Set | | Υ |
| Figure | 14.2-1.3.2 | Waterfall plot of Maximum Percentage Change from<br>Baseline in Sum of Longest Diameter | Evaluable Analysis Set | | |
| Figure | 14.2-1.4.1 | Swimmer Plot of Response Assessments | Full Analysis Set | | Υ |
| Figure | 14.2-1.4.2 | Swimmer Plot of Response Assessments | Evaluable Analysis Set | | |
| Figure | 14.2-1.5.1 | Kaplan-Meier Estimate for Progression-free Survival (PFS) | Full Analysis Set | | Y |
| Figure | 14.2-1.5.2 | Kaplan-Meier Estimate for Progression-free Survival (PFS) | Evaluable Analysis Set | | |
| Figure | 14.2-1.6.1 | Kaplan-Meier Estimate for Overall Survival (OS) | Full Analysis Set | | Υ |
| Figure | 14.2-1.6.2 | Kaplan-Meier Estimate for Overall Survival (OS) | Evaluable Analysis Set | 1 | |
| Figure | 14.2-1.7.1 | Kaplan-Meier Estimate for Duration of Response (DOR) | Full Analysis Set | | |
| 16.2 | • | Patient Data Listings | | 1 | |
| 16.2.1 | | Patient Disposition | | 1 | |
| Listing | 16.2.1-1 | Patient Informed Consent | All Patients Set | 1 | Υ |
| Listing | 16.2.1-2 | Failed Inclusion and Exclusion Criteria | All Patients Set | | Υ |
| Listing | 16.2.1-3 | Patient Disposition | All Patients Set | | Υ |
| 16.2.2 | | Analysis Sets | | | |
| Listing | 16.2.2-1 | Analysis Sets | All Patients Set | | |
| 16.2.3 | | Protocol Deviations | | | |
| Listing | 16.2.3-1 | Protocol Deviations | Full Analysis Set | | Υ |
| 16.2.4 | | Demographic Data | | | |
| Listing | 16.2.4-1 | Demographics and Baseline Characteristics | Full Analysis Set | | Υ |
| Listing | 16.2.4-2 | Smoking History | Full Analysis Set | | |
| | | 3 | | | |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

| Listing 16.2.4-4 Medical History and Concomitant Diseases Full Analysis Set Y Listing 16.2.4-5 Prior Systemic Anti-Cancer Therapies Full Analysis Set Y Listing 16.2.4-5 Prior Radiotherapy Courses Full Analysis Set Y Listing 16.2.4-7 Prior and Concomitant Medications Full Analysis Set Y Listing 16.2.4-8 On Treatment Radiation Full Analysis Set U Listing 16.2.4-9 On Treatment Radiation Full Analysis Set U Listing 16.2.4-10 On Treatment Boload Transfusions Full Analysis Set U Listing 16.2.4-11 NGS Data Full Analysis Set U Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set U Listing 16.2.5-2 Ulixertinib In-clinic Administration Full Analysis Set U Listing 16.2.5-3 Ulixertinib In-clinic Administration Full Analysis Set U Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Y Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set I Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set I Listing 16.2.5-1 Target Lesions Full Analysis Set I Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.8-1 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Biochemistry Fu | Licting | 16.2.4-3 | Disease History | Full Analysis Sot | Υ |
|---|---|---|---|---|---|
| Listing 16.2.4-5 Prior Systemic Anti-Cancer Therapies Full Analysis Set Y Listing 16.2.4-6 Prior Radiotherapy Courses Full Analysis Set Y Listing 16.2.4-8 Prior and Concomitant Medications Full Analysis Set Y Listing 16.2.4-8 On Treatment Radiation Full Analysis Set U Listing 16.2.4-9 On Treatment Surgery and Medical Procedures Full Analysis Set Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set U Listing 16.2.4-11 NGS Data Full Analysis Set V Listing 16.2.4-11 NGS Data Full Analysis Set V Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set U Listing 16.2.5-2 Ulixertinib In-clinic Administration Full Analysis Set V Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set V Listing 16.2.5-3 Ulixertinib Exposure Full Analysis Set V Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set V Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set V Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set V Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set V Listing 16.2.5-9 Ulixertinib Dispensed Full Analysis Set V Listing 16.2.5-9 Ulixertinib Dispensed Full Analysis Set V Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set V Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set V Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set V Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set V Listing 16.2.5-1 Target Lesions Full Analysis Set V Listing 16.2.6-2 Non-Target Lesions Full Analysis Set V Listing 16.2.6-3 New Lesions Full Analysis Set V Listing 16.2.6-4 Overall Response Full Analysis Set V Listing 16.2.6-5 Frogression-Free Survival (PFS Full Analysis Set V Listing 16.2.6-6 Survival Status Full Analysis Set V Listing 16.2.7-1 Adverse Events Full Analysis Set V Listing 16.2.7-1 Adverse Events Full Analysis Set V Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set V Listing 16.2.7-3 Serious Adverse Events Full Analysis Set V Listing 16.2.8-1 Hematology Full Analysis Set V Listing 16.2.8-3 Rem | Listing | | | Full Analysis Set | |
| Listing 16.2.4-6 Prior Radiotherapy Courses Full Analysis Set Y Listing 16.2.4-7 Prior and Concomitant Medications Full Analysis Set Y Listing 16.2.4-8 On Treatment Radiation Full Analysis Set U Listing 16.2.4-9 On Treatment Surgery and Medical Procedures Full Analysis Set Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set Listing 16.2.4-11 NGS Data Full Analysis Set U Listing 16.2.5-11 VIII NGS Data Full Analysis Set U Listing 16.2.5-12 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set U Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-3 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-8 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set U Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set U Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set U Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set U Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set U Listing 16.2.5-1 Target Lesions Full Analysis Set U Listing 16.2.6-1 Target Lesions Full Analysis Set U Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-5 New Lesions Full Analysis Set Y Listing 16.2.6-6 Survival Seturned Full Analysis Set Y Listing 16.2.6-6 Survival Seturned Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-3 Serious Adverse Events Full Analysis Set Y Listing 16. | | _ | • | | |
| Listing 16.2.4-7 Prior and Concomitant Medications Full Analysis Set Y Listing 16.2.4-8 On Treatment Radiation Full Analysis Set Listing 16.2.4-9 On Treatment Surgery and Medical Procedures Full Analysis Set Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set Listing 16.2.4-11 NGS Data Full Analysis Set Y Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-8 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-9 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Exposure Full Analysis Set I Listing 16.2.5-1 Ulixertinib Returned Full Analysis Set I Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.8-2 Blochemistry Full Analysis Set Y Listing 16.2.8-3 Deaths Adverse Events Full Analysis Set Y Listing 16.2.8-3 Deaths Adverse | | _ | | | |
| Listing 16.2.4-8 On Treatment Radiation Full Analysis Set Listing 16.2.4-10 On Treatment Surgery and Medical Procedures Full Analysis Set Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set Listing 16.2.4-11 NGS Data Full Analysis Set Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-8 Hydroxychloroquine Exposure Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-1 Hydroxychloroquine Exposure Listing 16.2.5-1 Target Lesions Full Analysis Set Listing 16.2.5-1 Hydroxychloroquine Full Full Analysis Set Listing 16.2.5-1 Hydroxychloroquine Full Full Analysis Set Listing 16.2.5-1 Target Lesions Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Listing 16.2.7-1 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Listing 16.2.7-4 Deaths Adverse Events Full Analysis Set Listing 16.2.8-1 Hematology Full Analysis Set Listing 16.2.8-3 Biochemistry Full Analysis Set Listing 16.2.8-3 Biochemistry Full Analysis Set Listing 16.2.8-3 Biochemistr | | _ | | _ | |
| Listing 16.2.4-9 On Treatment Surgery and Medical Procedures Full Analysis Set Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set Listing 16.2.4-11 NGS Data Full Analysis Set 16.2.5-1 Compliance and/or Drug Concentration Data Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Listing 16.2.5-5 Ulixertinib Exposure Listing 16.2.5-6 Hydroxychloroquine Exposure Listing 16.2.5-6 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-1 Ulixertinib Returned Full Analysis Set Listing 16.2.5-1 Ulixertinib Returned Full Analysis Set Listing 16.2.5-1 Ulixertinib Returned Full Analysis Set Listing 16.2.5-1 Ulixertinib Returned Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Biochemistry Full Analysis Set Y | | | | | Ť |
| Listing 16.2.4-10 On Treatment Blood Transfusions Full Analysis Set I 16.2.5 Compliance and/or Drug Concentration Data Listing 16.2.5-1 Ulikertinib In-clinic Administration Full Analysis Set Y Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set I 15.1 Set I 16.2.5-3 Ulikertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-3 Ulikertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulikertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-7 Ulikertinib Exposure Full Analysis Set Y Listing 16.2.5-8 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-9 Ulikertinib Dispensed Full Analysis Set I 15.1 Set I 16.2.5-9 Ulikertinib Reprosure Full Analysis Set I 15.1 Set I 16.2.5-9 Ulikertinib Reprosure Full Analysis Set I 15.1 Set I 16.2.5-1 Ulikertinib Reprosure Full Analysis Set I 15.1 Set I 16.2.5-1 Ulikertinib Reprosure Full Analysis Set I 15.1 Set I 16.2.5-1 Ulikertinib Reprosure Full Analysis Set I 15.1 Set I 16.2.5-1 Ulikertinib Returned Full Analysis Set I 16.2.5-1 Ulikertinib Returned Full Analysis Set I 16.2.5-1 Ulikertinib Returned Full Analysis Set I 16.2.5-1 Undividual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Toeaths | | _ | | | |
| Listing 16.2.4-11 NGS Data Full Analysis Set Y 16.2.5 Compliance and/or Drug Concentration Data Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Full Analysis Set Full Analysis Set Ilisting 16.2.5-2 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Y Listing 16.2.5-8 Hydroxychloroquine Exposure Full Analysis Set Ilisting 16.2.5-9 Ulixertinib Dispensed Full Analysis Set Ilisting 16.2.5-9 Ulixertinib Returned Full Analysis Set Ilisting 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Ilisting 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Ilisting 16.2.5-10 Individual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Survival Status Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y Listing 16.2.8-3 United Set Y Listing 16.2.8-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-3 Serious Adverse Events Full Anal | | | | | |
| Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Hematology Full Analysis Set Y Listing 16.2.8-3 Serious Adverse Events Full Analysis Set Y | | _ | | _ | v |
| Listing 16.2.5-1 Ulixertinib In-clinic Administration Full Analysis Set Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Full Analysis Set I Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Full Analysis Set I Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set I Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set I Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set I Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-2 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | | 16.2.4-11 | | ruii Andiysis set | ı |
| Listing 16.2.5-2 Hydroxychloroquine In-clinic Administration Full Analysis Set Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Listing 16.2.6-4 Overall Response Full Analysis Set Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Listing 16.2.6-6 Survival Status Full Analysis Set Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Listing 16.2.7-1 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Listing 16.2.7-4 Deaths Listing 16.2.8-3 Laboratory Data Listing 16.2.8-3 Coagulation Full Analysis Set Listing 16.2.8-3 Coagulation Full Analysis Set Listing 16.2.8-3 Coagulation Full Analysis Set Listing 16.2.8-3 Coagulation Full Analysis Set | | 16 2 5 1 | | Full Applysis Cot | |
| Listing 16.2.5-3 Ulixertinib Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Ulixertinib Exposure Full Analysis Set Ulixertinib Dispensed Full Analysis Set Full Analysis Set Ulixertinib Returned Full Analysis Set Ulixertinib Returned Full Analysis Set Ulixertinib Returned Full Analysis Set Individual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-7 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | _ | | | | |
| Listing 16.2.5-4 Hydroxychloroquine Interruptions and Adjustments Full Analysis Set Y Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Full Analysis Se | | _ | <u> </u> | • | v |
| Listing 16.2.5-5 Ulixertinib Exposure Full Analysis Set Y Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Full Analysi | | | | • | |
| Listing 16.2.5-6 Hydroxychloroquine Exposure Full Analysis Set Y Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Listing 16.2.6-4 Overall Response Full Analysis Set Listing 16.2.6-6 Survival Status Full Analysis Set Listing 16.2.6-6 Survival Status Full Analysis Set Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Listing 16.2.7-1 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Listing 16.2.7-4 Deaths Listing 16.2.8-1 Hematology Full Analysis Set Listing 16.2.8-2 Biochemistry Listing 16.2.8-3 Coagulation Full Analysis Set Listing 16.2.8-3 Coagulation Full Analysis Set | | _ | | | |
| Listing 16.2.5-7 Ulixertinib Dispensed Full Analysis Set Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set Listing 16.2.6-1 Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Listing 16.2.6-3 New Lesions Full Analysis Set Listing 16.2.6-4 Overall Response Full Analysis Set Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Listing 16.2.6-6 Survival Status Full Analysis Set Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Listing 16.2.7-1 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Listing 16.2.7-3 Serious Adverse Events Listing 16.2.7-4 Deaths Listing 16.2.8-1 Hematology Full Analysis Set Listing 16.2.8-2 Biochemistry Listing 16.2.8-3 Coagulation Full Analysis Set | | _ | · | | |
| Listing 16.2.5-8 Hydroxychloroquine Dispensed Full Analysis Set Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set 16.2.6 Individual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | | | | | Y |
| Listing 16.2.5-9 Ulixertinib Returned Full Analysis Set Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set 16.2.6 Individual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | | _ | • | | |
| Listing 16.2.5-10 Hydroxychloroquine Returned Full Analysis Set 16.2.6 Individual Efficacy Response data Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Y Listing 16.2.7-1 Adverse Events Full Analysis Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | | _ | | • | |
| Individual Efficacy Response data | _ | <u>16.2.5-9</u> | | Full Analysis Set | |
| Listing 16.2.6-1 Target Lesions Full Analysis Set Y Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Full Analysis Set Full Analysis Set | Listing | <u>16.2.5-10</u> | | Full Analysis Set | |
| Listing 16.2.6-2 Non-Target Lesions Full Analysis Set Y Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set Listing 16.2.7-1 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | 16.2.6 | | Individual Efficacy Response data | | |
| Listing 16.2.6-3 New Lesions Full Analysis Set Y Listing 16.2.6-4 Overall Response Full Analysis Set Y Listing 16.2.6-5 Progression-Free Survival (PFS Full Analysis Set Y Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set 16.2.7 Adverse Events Full Analysis Set Listing 16.2.7-1 Adverse Events All Patients Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | | Target Lesions | Full Analysis Set | |
| Listing16.2.6-4Overall ResponseFull Analysis SetYListing16.2.6-5Progression-Free Survival (PFSFull Analysis SetYListing16.2.6-6Survival StatusFull Analysis SetYListing16.2.6-7Duration of Response (DOR)Full Analysis SetY16.2.7Adverse EventsFull Analysis SetYListing16.2.7-1Adverse EventsAll Patients SetYListing16.2.7-2Treatment Emergent Adverse EventsFull Analysis SetYListing16.2.7-3Serious Adverse EventsFull Analysis SetYListing16.2.7-4DeathsAll Patients SetY16.2.8Laboratory DataFull Analysis SetYListing16.2.8-1HematologyFull Analysis SetYListing16.2.8-2BiochemistryFull Analysis SetYListing16.2.8-3CoagulationFull Analysis SetY | Listing | | Non-Target Lesions | Full Analysis Set | Y |
| Listing16.2.6-5Progression-Free Survival (PFSFull Analysis SetYListing16.2.6-6Survival StatusFull Analysis SetYListing16.2.6-7Duration of Response (DOR)Full Analysis SetY16.2.7Adverse EventsFull Analysis SetYListing16.2.7-1Adverse EventsAll Patients SetYListing16.2.7-2Treatment Emergent Adverse EventsFull Analysis SetYListing16.2.7-3Serious Adverse EventsFull Analysis SetYListing16.2.7-4DeathsAll Patients SetY16.2.8Laboratory DataFull Analysis SetYListing16.2.8-1HematologyFull Analysis SetYListing16.2.8-2BiochemistryFull Analysis SetYListing16.2.8-3CoagulationFull Analysis SetY | Listing | 16.2.6-3 | New Lesions | Full Analysis Set | Υ |
| Listing 16.2.6-6 Survival Status Full Analysis Set Y Listing 16.2.6-7 Duration of Response (DOR) Full Analysis Set 16.2.7 Adverse Events Full Analysis Set Listing 16.2.7-1 Adverse Events All Patients Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | 16.2.6-4 | Overall Response | Full Analysis Set | Υ |
| Listing 16.2.6-7 Duration of Response (DOR) 16.2.7 Adverse Events Listing 16.2.7-1 Adverse Events Listing 16.2.7-2 Treatment Emergent Adverse Events Listing 16.2.7-3 Serious Adverse Events Listing 16.2.7-4 Deaths Listing 16.2.7-4 Deaths Laboratory Data Listing 16.2.8-1 Hematology Listing 16.2.8-2 Biochemistry Listing 16.2.8-3 Coagulation Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y Listing 16.2.8-3 Full Analysis Set Y | Listing | 16.2.6-5 | Progression-Free Survival (PFS | Full Analysis Set | Υ |
| 16.2.7 Adverse Events Full Analysis Set Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | <u>16.2.6-6</u> | Survival Status | Full Analysis Set | Υ |
| Listing 16.2.7-1 Adverse Events All Patients Set Y Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | <u>16.2.6-7</u> | Duration of Response (DOR) | Full Analysis Set | |
| Listing 16.2.7-2 Treatment Emergent Adverse Events Full Analysis Set Y Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | 16.2.7 | | Adverse Events | Full Analysis Set | |
| Listing 16.2.7-3 Serious Adverse Events Full Analysis Set Y Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | <u>16.2.7-1</u> | Adverse Events | All Patients Set | Y |
| Listing 16.2.7-4 Deaths All Patients Set Y 16.2.8 Laboratory Data Full Analysis Set Y Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | <u>16.2.7-2</u> | Treatment Emergent Adverse Events | Full Analysis Set | Y |
| 16.2.8 Laboratory Data Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | 16.2.7-3 | Serious Adverse Events | Full Analysis Set | Y |
| Listing 16.2.8-1 Hematology Full Analysis Set Y Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | 16.2.7-4 | Deaths | All Patients Set | Y |
| Listing 16.2.8-2 Biochemistry Full Analysis Set Y Listing 16.2.8-3 Coagulation Full Analysis Set Y | 16.2.8 | | Laboratory Data | | |
| Listing 16.2.8-3 Coagulation Full Analysis Set Y | Listing | 16.2.8-1 | Hematology | Full Analysis Set | Υ |
| | Listing | 16.2.8-2 | Biochemistry | Full Analysis Set | Υ |
| Licting 16.2.8-4 Urinalysis Full Analysis Set V | Listing | 16.2.8-3 | Coagulation | Full Analysis Set | Υ |
| Listing 10.2.07 Officiallysis Set | Listing | 16.2.8-4 | Urinalysis | Full Analysis Set | Υ |
| Listing 16.2.8-5 Tumor Markers Full Analysis Set | Listing | 16.2.8-5 | Tumor Markers | Full Analysis Set | |
| Listing 16.2.8-6 Pregnancy Full Analysis Set | | 16.2.8-6 | Pregnancy | Full Analysis Set | |
| 16.2.9 Other Safety Data | 16.2.9 | | Other Safety Data | | |
| Listing 16.2.9-1 Vital Signs Full Analysis Set Y | Listing | <u>16.2.9-1</u> | Vital Signs | Full Analysis Set | Y |
| Listing 16.2.9-2 Electrocardiogram Full Analysis Set Y | Listing | 16.2.9-2 | Electrocardiogram | Full Analysis Set | Y |
| Listing 16.2.9-3 ECHO/MUGA Full Analysis Set Y | Listing | 16.2.9-3 | ECHO/MUGA | Full Analysis Set | Υ |
| Listing 16.2.9-4 Physical Examination Full Analysis Set Y | | 16.2.9-4 | Physical Examination | Full Analysis Set | Υ |
| Listing 16.2.9-5 Ophthalmology exam Full Analysis Set Y | Listing | | | | Υ |
| Listing 16.2.9-6 ECOG Performance Status Full Analysis Set Y | _ | | | Full Analysis Set | Υ |
| 16.2.11 Pharmacokinetic Data | | | | · | |
| Listing 16.2.11-1 Pharmacokinetic Concentration Data PK Analysis Set Y | | 16.2.11-1 | | PK Analysis Set | Υ |
| Listing 16.2.11-2 Pharmacokinetic Parameters Data PK Analysis Set Y | | _ | | | Υ |

<sup>\*</sup>Table, Figure or Listing that will be used for SMC purposes. Y=Yes



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

# 4 General programming notes

All tables will be reported by treatment Basket.

An 'Overall' column will be included in all tables.

| Column headers | | | | | |
|----------------|----------|----------|----------|----------|---------|
| Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |

For tables reporting data on All Patients Set, a screening failures column will be added.

The full-page header to be included for each delivery is indicated in the table below:

| Delivery | Туре | Page Header |
|----------------|---------|-------------|
| Dry run | Dry run | Dry-run |
| SMC N* | Final | Final |
| Final analysis | Draft | Draft |
| | Final | Final |

<sup>\*</sup>N references to the SMC chronological number

For the listings, all cases where 'Other' is present, please present the respective 'Other' specification.

All Listings will be sorted by Basket and patient ID. A programming note will be added to each Listing when another variable is needed to make the sorting meaningful (e.g., assessment date).



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.1 - Patient Disposition
All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients enrolled [a] | XX | XX | XX | XX | XX | XX | XX |
| Patients completed screening [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued from screening [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary reason for discontinuation [c] | | | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Screen Failure | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Technical Problems | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients rescreened [b] | | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients eligible for inclusion in the study [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Patients treated with study drug [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

<sup>[</sup>a] Patients who signed the informed consent.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Percentages are calculated from the number of patients enrolled.

<sup>[</sup>c] Percentages are calculated from the number of patients who discontinued from screening.

<sup>[</sup>d] Percentages are calculated from the number of patients who were treated with study drug.

<sup>[</sup>e] Percentages are calculated from the number of patients who discontinued from treatment.

<sup>[</sup>f] Percentages are calculated from the number of patients who discontinued from study.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-1.1 - Patient Disposition All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients completed treatment [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Discontinued from treatment [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Primary reason for discontinuation [e] | | | | | | | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

<sup>[</sup>a] Patients who signed the informed consent.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>[</sup>b] Percentages are calculated from the number of patients enrolled.

<sup>[</sup>c] Percentages are calculated from the number of patients who discontinued from screening.

<sup>[</sup>d] Percentages are calculated from the number of patients who were treated with study drug.

<sup>[</sup>e] Percentages are calculated from the number of patients who discontinued from treatment.

<sup>[</sup>f] Percentages are calculated from the number of patients who discontinued from study.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.1 - Patient Disposition
All Patients Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients completed study [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Primary reason for completion [f] | | | | | , | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Pregnancy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Sponsor Request | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Protocol-Specified Withdrawal Criterion Met | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

- [a] Patients who signed the informed consent.
- [b] Percentages are calculated from the number of patients enrolled.
- [c] Percentages are calculated from the number of patients who discontinued from screening.
- [d] Percentages are calculated from the number of patients who were treated with study drug.
- [e] Percentages are calculated from the number of patients who discontinued from treatment.
- [f] Percentages are calculated from the number of patients who completed the study.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


# PROGRAMMING NOTES:

· Display all possible reasons, either reported for at least one patient or not.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.2 - Number of Patients in the Analysis Sets


| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| All Patients Set [a] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Full Analysis Set [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Stage 1 Analysis Set [c] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| Evaluable Analysis Set [d] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| PK Analysis Set [e] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |

- [a] Patients who were enrolled regardless of whether they received the study drug or not.
- [b] Patients who received at least 1 dose of the study drug.
- [c] First 13 patients who have completed at least one cycle of therapy and who have received a minimum of 75% of prescribed study therapy during Cycle 1
- [d] Patients who received at least one dose of study drug and have at least one post-treatment study evaluation or who have discontinued therapy prior to the first post-treatment study evaluation due to clinical progressive disease or drug-related adverse events.
- [e] Patients who received at least one dose of study medication and have at least one post dose PK measurement.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-1.3 - Summary of Important Protocol Deviations Full Analysis Set Page 1 of Y

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Number of patients with at least one important protocol deviation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Deviation category 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| - | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Deviation category 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Summary term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *********** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: A patient with multiple occurences of a protocol deviation is counted only once in this deviation category/summary term.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

- Categories / Summary terms to match the PDCF.
- Present only important protocol deviations with at least one occurrence (where classification=Important).




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set

| XX<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX<br>XX.XX (XX.XXX)<br>XX.XX<br>XX.X; XX.X | XX<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X |
|---|---|---|---|---|
| XX.XX (XX.XX)<br>XX.XX | XX.XX (XX.XXX)<br>XX.XX | XX.XX (XX.XX)<br>XX.XX | XX.XX (XX.XX)<br>XX.XX | XX.XX (XX.XX) |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | **** /**** *** | **** | | **** |
| | | | | XX (XX.X)<br>XX (XX.X) |
| | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


BMSOP111/F2


<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set Page 2 of Y

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Race - n (%) | | | _ | _ | _ | |
| American Indian or | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Alaska Native | | | | | | |
| Asian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pacific Islander | | | | | | |
| White | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Ethnicity - n (%) | | | | | | |
| Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 1 | | | | | |
| Weight (kg) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set Page 3 of Y

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Height (cm) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| ECOG performance at Baseline | e - n | | | | | |
| (%) [b] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Smoking History - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Current | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Former | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)


<sup>[</sup>b] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.1 - Demographics and Baseline Characteristics Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Gene/Codon/Amino acid change | | | | | | |
| HRAS/G469/Alanine A | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) |
| KRAS/G469/Arginine R | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) |
| NRAS/G469/Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.doc)


BMSOP111/F2


<sup>[</sup>a] Last non-missing value prior to first dose of study treatment.

<sup>[</sup>b] Body Mass Index (BMI)=Weight (kg) / Height(m)^2.

<sup>[</sup>c] 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities.



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.2 - Disease History Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| ancer Diagnosis - n (%) | | | | | | |
| Intrahepatic cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Perihilar cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Extrahepatic cholangiocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pancreatic adenocarcinoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ime since initial diagnosis | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| isease stage at enrollment - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

[a] Calculated as (date of first dose of study treatment - date of diagnosis) / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Table 14.1-2.2 - Disease History Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Disease stage at initial | | | | | | |
| diagnosis - n (%) | | | | | | |
| i | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Method of diagnosis - n (%) | | | | | | |
| Cytological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Histological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Prior Radiation Therapies - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | | | | | | |

[a] Calculated as (date of first dose of study treatment - date of diagnosis) / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-2.3 - Summary of Medical History Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any relevant medical history | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>.

If there is more than one medical history within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one medical history within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within primary SOC.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-2.4 - Summary of Concomitant Diseases Full Analysis Set Page 1 of Y

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any relevant concomitant disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *********** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *************************************** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>.

If there is more than one concomitant disease within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one concomitant disease within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within primary SOC.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Received at least one systemic prior anti-cancer Therapy - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lines of systemic prior anti-cancer therapies - n $(%)$ | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mean (SD) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) | XX.X<br>(XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Most recent therapy before study treatment start Regimen name - n (%) | | | | | | |
| xxxxxxx | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| xxxxxxx | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| xxxxxxx | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies
Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Best Response - n (%) | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Duration of therapy (months) [a] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Time since Best Overall Response | | | | | | |
| (months) [b] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


Filename: (Specify file name.rtf)

<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-3.1 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Time since Relapse/Progression | | | | | | |
| (months) [c] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Reason for discontinuation - n (%) | | | | | | |
| Intolerance | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lack of Efficacy (incl. PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed Therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Calculated as [(date of first study treatment - date of BOR)+1] / 30.4375.

<sup>[</sup>c] Calculated as [(date of first study treatment - date of Relapse/Progression)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


## Table 14.1-3.2 - Prior Radiotherapy Courses Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Received at least one prior radiotherapy - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total number of prior radiotherapy courses - $n$ (%) | | | | | | |
| 1 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Site of prior radiotherapy - n (%) [a] Abdominal Cavity Adrenal Gland | XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Most recent prior radiotherapy before study<br>treatment start<br>Site of prior radiotherapy - n (%)<br>Abdominal Cavity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Duration of therapy (months) [b] | | | | | | |
| n<br>Mean (SD)<br>Median<br>Min; Max | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX | XX<br>XX.X<br>(XX.XX)<br>XX.X<br>XX; XX |

<sup>[</sup>a] Patients can have more than 1 site of prior radiotherapy if they had multiple prior radiotherapies.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


<sup>[</sup>b] Calculated as [(end date of therapy - start date of therapy)+1] / 30.4375.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.1-3.3 - Prior Medications Full Analysis Set

| ATC Class Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| FIGURE TELIA | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0) |
| Any Prior Medications | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *********** | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: WHOHD-B3 <vx.x>. ATC=Anatomical Therapeutic Chemical.

If there is more than one medication within an ATC class, the patient is counted only once under that ATC class. If there is more than one medication within an ATC class and preferred term (PT), the patient is counted only once in that ATC class and PT.

ATC classes are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within ATC class.

Prior medication is defined as any medications whose end date is before the first study treatment date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.1-3.4 - Concomitant Medications Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.1-3.3
- Present concomitant medications.
- Replace footnote 'Prior medication is defined as...' with the following footnote:
   (Concomitant medication is defined as any medication ongoing at first day of study drug or started after first day of study drug up to the end of the ontreatment period.'




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.1.1 - Treatment exposure (Ulixertinib)
Full Analysis Set

| | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Number of cycles received | | | | | | |
| [a] - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | ( | () | () | (************************************** | () | () |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| Duration of exposure to | | | | | | |
| ulixertinib (months) [b] - n | | | | | | |
| (%) | | | | | | |
| < 1 month | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1-2 months | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2-3 months | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

<sup>[</sup>a] Number of cycles received = Number of cycles where the patient received at least one dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)

<sup>[</sup>b] Duration of exposure (months) = [(Date of last known treatment dosing with drug - date of initial dosing with drug) + 1] / 30.4375.

<sup>[</sup>c] Actual cumulative dose received (mg) = Sum of [(Stop date - Start date for each time period reported in the dairy) x Dose].

<sup>[</sup>d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days).



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.1.1 - Treatment exposure (Ulixertinib) Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Actual cumulative dose on | | | | | | |
| alixertinib (mg) [c] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |
| Relative dose intensity [d] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

<sup>[</sup>a] Number of cycles received = Number of cycles where the patient received at least one dose.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)


BMSOP111/F2


Filename: (Specify file name.rtf)

<sup>[</sup>b] Duration of exposure (months) = [(Date of last known treatment dosing with drug - date of initial dosing with drug) + 1] / 30.4375.

<sup>[</sup>c] Actual cumulative dose received (mg) = Sum of [(Stop date - Start date for each time period reported in the dairy) x Dose].

<sup>[</sup>d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days).



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.1-4.1.2 - Treatment exposure (Hydroxychloroquine) Full Analysis Set

## PROGRAMMING NOTES:

• Repeat Table 14.1-4.1.1



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.1-4.2.1 - Dosing Interruptions and Adjustments (Ulixertinib) Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| At least one dose adjustment - n (%) Reason dose changed - n (%) [a] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Parental/Guardian decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Consent withdrawal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Consent Withdiawai | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | AA (AA.A) | AA (AA.A) | AA (AA.A) | AA (AA.A) | AA (AA.A) | AA (AA.A) |
| Other | | | | | | |
| Dose changed to - n (%) [b] | | | | | | |
| 150mg | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 300mg | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 450mg | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| At least one dose interruption - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason dose interrupted [a] | | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dispensing Error | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Investigator Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Consent Withdrawal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patient Decision | | | | | | |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] A patient can be counted under several reasons if they had multiple different dose changes/interruptions.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


<sup>[</sup>b] A patient can be counted under more than one dose level if they had multiple different dose changes.



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.1-4.2.2 - Dosing Interruptions and Adjustments (Hydroxychloroquine) Full Analysis Set

# PROGRAMMING NOTES:

• Repeat Table 14.1-4.2.1




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.2-1.1.1 - Best Overall Response and Overall Response Rate Full Analysis Set

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Best overall response - n (%) [a] | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| verall response rate (CR+PR) - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 5 % CI for Overall response rate | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Disease control rate (CR+PR+SD) - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 95 % CI for Disease Control rate | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Non-responders (SD+PD+NE) - n (%) [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable , CI=Confidence Interval.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


<sup>95%</sup> CI is estimated using the Clopper-Pearson method.

<sup>[</sup>a] Confirmed Best overall response as per RECIST 1.1

<sup>[</sup>b] Non responders: Patients without a confirmed response or a missing baseline/screening tumor assessment will be considered non-responders



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.2-1.1.2 - Best Overall Response and Overall Response Rate
Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.1.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.2-1.2.1 - Overall, Target and Non-Target Lesion Response Full Analysis Set

| | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| C3D1 | | | | | | |
| Target Lesion Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Target Lesion Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Complete Response/Non | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | | | | | | |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Applicable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Overall Response - n (%) | | | | | | |
| Complete response (CR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response (PR) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive disease (PD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Evaluable (NE) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| D | | | | | | |
| Programming Note: Repeat for all | | | | | | |
| available assessments | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.2.2 - Overall, Target and Non-Target Lesion Response Evaluable Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.2-1.2.1
- Present data on Evaluable AnalysisSet.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.2-1.3.1 - Incidence of New Lesions Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3D1 | | | | | | |
| New Lesions - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of New Lesions - n (%) | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.3.2 - Incidence of New Lesions Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.3.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.2-1.4.1 - Progression-Free Survival (PFS)
Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with events - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PFS (months) [a] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| CM probability estimates for PFS (95% | | | | | | |
| CI) [b] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X |

Note: CI=Confidence Interval.

Progression-Free Survival (PFS) is the time from the first ulixertinib dose dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

- [a] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [b] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


<sup>\*</sup> Censored observation at maximum value.



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.4.2 - Progression-Free Survival (PFS) Evaluable Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.2-1.4.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Table 14.2-1.5.1 - Overall Survival (OS) Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with events - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| OS (months) [a] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| KM probability estimates for PFS (95% | | | | | | |
| CI) [b] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |

Note: CI=Confidence Interval.

Overall Survival is defined as the time from first treatment to death.

- [a] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [b] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


<sup>\*</sup> Censored observation at maximum value.


Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.2-1.5.2 - Overall Survival (OS) Evaluable Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.2-1.4.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.2-1.6.1 - Duration of Response Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Patients with response (CR+PR) | XX | XX | XX | XX | XX | XX |
| Patients with events - n (%) [a] Patients censored - n (%) [a] | XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| DOR (months) [b] | | | | | | |
| Median (95% CI) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| Min, Max | XX, XX* | XX, XX | XX, XX | XX, XX* | XX, XX | XX, XX |
| KM probability estimates for PFS (95% CI) [c] | | | | | | |
| 3 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 6 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 9 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 12 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |
| 18 Months | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) | XX (X.X, X.X) |

Note: CI=Confidence Interval, CR=Complete Response, PR=Partial Response.

Duration of response is the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause. +1

- [a] Percentage calculated on patients with response. Events are death or disease progression.
- [b] Product-limit (Kaplan-Meier) estimates. 95% CI for median calculated using the Brookmeyer and Crowley method.
- [c] Based upon Kaplan-Meier (KM) estimates and 95% CI use the log-log transformation.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>\*</sup> Censored observation at maximum value.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.3-1.1 - Overview Summary of Treatment-Emergent Adverse Events Full Analysis Set

| | Basket :<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| 7.1 | | | | | | |
| Number of patients with: | | | **** | **** (**** **) | **** (**** **) | **** /*** *** |
| Any TEAE | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to Both | XX (XX.) | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to Uli. | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE to HCQ. | XX (XX.) | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any SAE | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related SAE | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation | XX (XX.) | (XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation within 1 cycle | XX (XX.) | (XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation within 1 cycle | XX (XX. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment discontinuation following 1 cycle | XX (XX. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment discontinuation | XX (XX.) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| following 1 cycle | 00 /00 | , , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | XX (XX.X) | 00 /00 01 | XX (XX.X) | עם עט עט |
| Any TEAE leading to treatment interruption | XX (XX.) | | | XX (XX.X) | | XX (XX.X) |
| Any Related TEAE leading to treatment interruption | XX (XX. | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment interruption within 1 cycle | XX (XX.) | (XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment interruption within 1 cycle | XX (XX.) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to treatment interruption following 1 cycle | XX (XX.) | (XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to treatment interruption following 1 cycle | XX (XX.) | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: SAE=Serious Adverse Events, TEAE=Treatment-Emergent Adverse Events

Note 2: Any related TEAE includes TEAEs that are considered related to either hydroxychloroquine or ulixertinib.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


# Table 14.3-1.1 - Overview Summary of Treatment-Emergent Adverse Events

#### Full Analysis Set

| | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| umber of patients with: | | | | | | |
| Any TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any related TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE leading to dose reduction within | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 1 | | | | | | |
| Any Related TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| within Cycle 1 | | | | | | |
| Any TEAE leading to dose reduction following | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 1 | | | | | | |
| Any Related TEAE leading to dose reduction | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| following Cycle 1 | | | | | | |
| Any TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any TEAE with Grade >= 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any Related TEAE with Grade >= 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: SAE=Serious Adverse Events, TEAE=Treatment-Emergent Adverse Events

Note 2: Any related TEAE includes TEAEs that are considered related to either hydroxychloroquine or ulixertinib.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

# Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

"Related TEAE to Both", "Related TEAE to Uli." and "Related TEAE to HCQ." will be presented for all treatment-related adverse events [...]" in the above table.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.2 - Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within each SOC.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.3-1.3 - Summary of Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term
Full Analysis Set

| System | | Basket 1 | | | Basket 2 | ! | | Basket 3 | 1 | | Basket 4 | | | Basket 5 | | | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ | | N=XX | | | N=XX | | | N=XX | | | N=XX | | | N=XX | | | N=XX | |
| Class | | n (%) | | | n (%) | | | n (%) | | | n (%) | | | n (%) | | | n (%) | |
| Preferred | | | | | | | | | | | | | | | | | | |
| Term | | | | | | | | | | | | | | | | | | |
| | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ |
| Any | ХX | xx | xx | хx | xx | xx | ХX | xx | xx | xx | xx | xx | ХX | xx | xx | ХX | xx | xx |
| related | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) |
| TEAE | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) | (AA.A) |
| System<br>organ | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) |
| class 1 | ,, | ( | ( | ,, | ( | (, | (, | (, | (, | ( | (, | ( | ( | ( | ( | ,, | ,, | ( |
| | XX | XX | XX | xx | XX | XX | XX | XX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX |
| Preferred<br>term 1 | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) |
| | XX | XX | XX | XX | XX | XX | XX | XX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX |
| Preferred<br>term 2 | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) | (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

Note 2: Both = TEAE related to both treatments, Uli = TEAE related to ulixertinib, HCQ = TEAE related to Hydroxychloriquine.

Related TEAE: TEAEs with causality=Related, Possibly Related or missing.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted by descending order of frequency for the overall Basket within each SOC.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.4 - Summary of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.2
- Present Serious TEAE: TEAEs with SAE =" Yes".
- Add footnote:

"Serious TEAE: TEAEs with SAE =" Yes"."

Table 14.3-1.5 - Summary of Related Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Present Related Serious TEAE: SAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"SAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Table 14.3-1.6 - Summary of Treatment-Emergent Adverse Events by Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1<br>Preferred term 2 | XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a preferred term (PT), the patient is counted only once in that PT.

PTs are sorted in descending order of frequency for the overall Basket.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


# Table 14.3-1.7 - Summary of Related Treatment-emergent Adverse Events by Preferred Term Full Analysis Set

| Preferred<br>Term | | Basket 1<br>N=XX<br>n (%) | | | Basket 2<br>N=XX<br>n (%) | ! | | Basket 3<br>N=XX<br>n (%) | | | Basket 4<br>N=XX<br>n (%) | | | Basket 5<br>N=XX<br>n (%) | | | Overall<br>N=XX<br>n (%) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ | Both | Uli | HCQ |
| Any<br>related<br>TEAE | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| Preferred<br>term 1 | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| Preferred<br>term 2 | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) | XX<br>(XX.X) | (XX.X) | (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | (XX.X) | (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

Note 2: Both = TEAE related to both treatments, Uli = TEAE related to ulixertinib, HCQ = TEAE related to Hydroxychloriquine.

Related TEAE: TEAEs with causality=Related, Possibly Related or missing.

If there is more than one TEAE within a preferred term (PT), the patient is counted only once in that PT.

PTs are sorted in descending order of frequency for the overall Basket.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.8 - Summary of Serious Treatment-emergent Adverse Events by Preferred Term Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.6
- Present Serious TEAE: TEAEs with SAE =" Yes".
- Add footnote:

"Serious TEAE: TEAEs with SAE =" Yes"."

Table 14.3-1.9 - Summary of Related Serious Treatment-emergent Adverse Events by Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.7
- Present Related Serious TEAE: SAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"SAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.10 - Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term for Maximum CTCAE Grade
Full Analysis Set

Basket: Basket X

| System Organ Class<br>Preferred Term | Any CTC Grade<br>n (%) [Events] | CTC Grade 1<br>n (%) | CTC Grade 2<br>n (%) | CTC Grade 3<br>n (%) | CTC Grade 4<br>n (%) | CTC Grade 5<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *************************************** | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| *********** | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>; CTCAE v5.0. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC and maximum severity. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC, PT and maximum severity. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

[Events] presents the number of TEAEs reported overall, by primary SOC and PT regardless of severity.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

Present for each Basket and overall.


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.11 - Summary of Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term for Maximum CTCAE Grade

Full Analysis Set


Basket: Basket X, Related to both study treatments

| System Organ Class<br>Preferred Term | Any CTC Grade<br>n (%) [Events] | CTC Grade 1<br>n (%) | CTC Grade 2<br>n (%) | CTC Grade 3<br>n (%) | CTC Grade 4<br>n (%) | CTC Grade 5<br>n (%) |
|---|---|---|---|---|---|---|
| Any related TEAE | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ********** | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) [XX] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>; CTCAE v5.0. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE within a system organ class (SOC), the patient is counted only once under that SOC and maximum severity. If there is more than one TEAE within a SOC and preferred term (PT), the patient is counted only once in that SOC, PT and maximum severity. Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

[Events] presents the number of TEAEs reported overall, by primary SOC and PT regardless of severity.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Present for each Basket and overall. For each Basket and Overall present TEAEs that are Related to both study treatments, related to ulixertinib and related to hydroxychloriquine
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Template Author: Andra Rusu  BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Table 14.3-1.12 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class<br>Preferred Term | Basket l<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE leading to treatment discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE leading to treatment discontinuation within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE leading to treatment discontinuation within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.13 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation by System Organ Class and
Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Table 14.3-1.14 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Within Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn within the first 28 days of study."

Table 14.3-1.15 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Within Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

## PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation within cycle 1'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn within the first 28 days of study."

Template Author: Andra Rusu  BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.16 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Add footnote:

"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn after the first 28 days of study." 
"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Table 14.3-1.17 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Discontinuation Following Cycle 1 by

System Organ Class and Preferred Term

Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any TEAE leading to treatment discontinuation following cycle 1'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:


"TEAEs leading to treatment discontinuation: any TEAEs with Action taken with study treatment=Drug withdrawn after the first 28 days of study." 
"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

Template Author: Andra Rusu  BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.18 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption by System Organ Class and Preferred
Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- · Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption.'
- Add footnote:
- "Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted'.

Table 14.3-1.19 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption by System Organ Class and
Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted'.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.20 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption Within Cycle 1 by System Organ Class and Preferred Term

Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption within Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' within the first 28 days of study.

Table 14.3-1.21 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption Within Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption within Cycle 1.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' within the first 28 days of study.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.22 - Summary of Treatment-Emergent Adverse Events Leading to Treatment Interruption Following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to treatment interruption following Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' after the first 28 days of study.

Table 14.3-1.23 - Summary of Related Treatment-Emergent Adverse Events Leading to Treatment Interruption Following Cycle 1 by System
Organ Class and Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to treatment interruption following Cycle 1'.
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Drug Interrupted' after the first 28 days of study.

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.24 - Summary of Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and Preferred Term Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced'".

Table 14.3-1.25 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and
Preferred Term
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced'".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-1.26 - Summary of Treatment-Emergent Adverse Events Leading to Dose Reduction within Cycle 1 by System Organ Class and
Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction within Cycle 1.'
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' within the first 28 days of study".

Table 14.3-1.27 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction within Cycle 1 by System Organ

Class and Preferred Term

Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction within Cycle 1.'
- Add footnotes:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' within the first 28 days of study".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

Table 14.3-1.28 - Summary of all Treatment-Emergent Adverse Events Leading to Dose Reduction following Cycle 1 by System Organ Class and Preferred Term

Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.12
- Replace 'Any TEAE' by 'Any TEAE leading to dose reduction following Cycle 1.
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' after the first 28 days of study".

Table 14.3-1.29 - Summary of Related Treatment-Emergent Adverse Events Leading to Dose Reduction following Cycle 1 by System Organ
Class and Preferred Term
Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to dose reduction following Cycle 1.
- Add footnote:

"Includes TEAE with 'Action Taken with treatment' = 'Dose Reduced' after the first 28 days of study".

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Filename: (Specify file name.rtf)

Table 14.3-1.30 - Summary of Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term
Full Analysis Set

| System Organ Class<br>Preferred Term | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|
| Any TEAE leading to death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: MedDRA <vx.x>. TEAE=Treatment-Emergent Adverse Events.

If there is more than one TEAE leading to death within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one TEAE leading to death within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.

Primary SOCs are presented by descending order of frequency for the overall Basket, PTs are sorted within primary SOC descending order of frequency for the overall Basket within each SOC.

BMSOP111/F2

TEAEs leading to Death: any TEAE resulting in death, Outcome=Fatal, CTC Grade=5.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


Template Author: Andra Rusu 



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.31 - Summary of Related Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term Full Analysis Set


#### PROGRAMMING NOTES:

- Repeat Table 14.3-1.3
- Replace 'Any TEAE' by 'Any related TEAE leading to death'
- Present Related TEAE: TEAEs with causality=Related, Possibly Related or missing.
- Add footnote:

"Related TEAE: TEAEs with causality=Related, Possibly Related or missing."

"TEAEs leading to Death: any TEAE resulting in death, Outcome=Fatal, CTC Grade=5."

Template Author: Andra Rusu Version 5.0 25Jun2020  BMSOP111/F2



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-1.32 - Summary of Deaths All Patients Set Page 1 of Y

| | Basket 1<br>N=XX<br>n (%) | Basket 2<br>N=XX<br>n (%) | Basket 3<br>N=XX<br>n (%) | Basket 4<br>N=XX<br>n (%) | Basket 5<br>N=XX<br>n (%) | Screen<br>Failures<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|---|---|---|
| Patients who died during the study | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary cause of death<br>Progressive Disease<br>Adverse Event<br>Unknown | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Patients who died after<br>taking the first dose of<br>ulixertinib | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary cause of death<br>Progressive Disease<br>Adverse Event<br>Unknown | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.1 - Summary and Change from Baseline in Hematology Laboratory Results by Visit Full Analysis Set

Parameter: XXXXX (XX)

| Visit | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- Present for all hematology parameters: hematocrit, hemoglobin, platelets, white blood cells (WBC), neutrophil absolute, lymphocyte absolute with respective unit measure.
- Present for all available visits.


BMSOP111/F2




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Table 14.3-2.2.1 - Gradable Hematology Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set

| Parameter (unit)<br>Cycle | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| CTCAE Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX (XXX) | | | | | | |
| Cycle 1 | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | | | | | |

Note: CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

• Present for all hematology parameters where CTCAE grades are defined as per the SAP appendix 14.2.


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.2.2 - Non-gradable Hematology Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set


| Parameter (unit) | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Cycle | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| CTCAE Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX (XXX) | | | | | | |
| Cycle 1 | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | | | | | |

Note: CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

Present for all hematology parameters where CTCAE grades are not defined as per the SAP appendix 14.2.

Template Author: Andra Rusu  BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.3.1 - Shift Table of Gradable Hematology Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set


Basket: Basket 1 (N=XX)

| | | | Wo | orst CTCAE grade | during treatmen | t period | | |
|---|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Normal | 1 | 2 | 3 | 4 | Missing | Total |
| (unit) | Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXXX | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (XXX) | 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: CTCAE v5.0.

Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

BMSOP111/F2

# PROGRAMMING NOTES:

Present for each Basket and overall, and for all hematology parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Template Author: Andra Rusu 



Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.3.2 - Shift Table of Non-gradable Hematology Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

Basket: Basket 1 (N=XX)

BioMed Valley Discoveries

| Worst grade during treatment period | | | | | |
|---|---|---|---|---|---|
| Baseline | Low | Normal | High | Missing | Total |
| Grade | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Grade<br>Low<br>Normal<br>High<br>Missing | Crade n (%) | Baseline | Baseline Low Normal High Grade n (%) n (%) n (%) Low XX (XX.X) XX (XX.X) XX (XX.X) Normal XX (XX.X) XX (XX.X) XX (XX.X) High XX (XX.X) XX (XX.X) XX (XX.X) Missing XX (XX.X) XX (XX.X) XX (XX.X) | Baseline Low Normal High Missing Grade n (%) n (%) n (%) n (%) Low XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Normal XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) High XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Missing XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

Present for all Baskets and overall, and for all hematology parameters where CTCAE grades are not defined as per the SAP appendix 14.2.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

Table 14.3-2.4 - Summary and Change from Baseline in Biochemistry Laboratory Results by Visit
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat Table 14.3-2.1
- Present for all biochemistry parameters: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, carbon dioxide, calcium, chloride, cholesterol, creatinine, glucose, inorganic phosphorus, lactate dehydrogenase, potassium, total protein, sodium, total bilirubin, triglycerides, uric acid, urea nitrogen.
- Present for all available visits.

Table 14.3-2.5.1 - Gradable Biochemistry Laboratory Results - Worst On-treatment Value by Cycle Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.2.1
- Present for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Table 14.3-2.5.2 - Non-gradable Biochemistry Laboratory Results - Worst On-treatment Value by Cycle
Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.2.2
- Present for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Table 14.3-2.6.1 - Shift Table of Gradable Biochemistry Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

BMSOP111/F2

#### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.3.1
- . Present for all Baskets and overall, and for all biochemistry parameters where CTCAE grades are defined as per the SAP appendix 14.2.

Template Author: Andra Rusu 



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.3-2.6.2 - Shift Table of Non-gradable Biochemistry Laboratory Results - Baseline vs Worst On-treatment Value Full Analysis Set

#### PROGRAMMING NOTES:

- Repeat of Table 14.3-2.3.2
- Present for all Baskets and overall, and for all biochemistry parameters where CTCAE grades are not defined as per the SAP appendix 14.2.




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Table 14.3-2.7 - Summary at Baseline in Coagulation Laboratory Results Full Analysis Set

# PROGRAMMING NOTES:

- Repeat Table 14.3-2.1
- · Present for all coagulation parameters: PT, INR, PTT




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.8 - Summary at Baseline in Urinalysis Laboratory Results
Full Analysis Set


Filename: (Specify file name.rtf)

Parameter: Specific gravity (XX)

| Visit<br>Statistics | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.


Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-2.8 - Summary and Change from Baseline in Urinalysis Laboratory Results by Visit
Full Analysis Set

Parameter: Blood (XX)

| Visit | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Statistics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | | | | | | |
| Negative | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4+ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<cont.>

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

- Present for all urinalysis parameters: specific gravity, protein, glucose, occult blood, microscopic examination of RBC, microscopic examination of WBC, microscopic examination of casts.
- Present for all available visits.


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.1 - Summary and Change from Baseline in Vital Signs by Visit Full Analysis Set

Parameter: XXXXX (XX)

| Visit | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

- Present for all vital signs: systolic blood pressure, diastolic blood pressure, pulse, respiratory rate, pulse oximetry and temperature with respective unit measure.
- Present for all available visits.


BMSOP111/F2




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.2 - Shift Table of Vital Signs Results - Baseline vs Worst On-treatment Value Full Analysis Set

Basket: Basket 1 (N=XX)

| | | | Worst value during on-treatment period | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Low | Normal | High | Very High | Missing | Total |
| (unit) | Value | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| XXXX | Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX) | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Very High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Percentages are based on the number of patients in the Basket.

For Temperature, Low: < 36.4°C, Normal: 36.4°C - 37.7°C, High: > 37.7°C.

For Pulse, Low: < 55 bpm, Normal: 55-100 bpm, High: 101-150 bpm, Very high: > 150 bpm.

For Systolic blood pressure, Low: < 90 mmHg, Normal: 90-130 mmHg, High: 131-160 mmHg, Very high: ≥ 161 mmHg. For Diastolic blood pressure, Low: < 60 mmHg, Normal: 60-85 mmHg, High: 86-100 mmHg, Very high: ≥ 101 mmHg.

For Pulse oximetry, Very Low: < 90 %, Low: 90-95 %, Normal: ≥ 95 %.

For Respiratory Rate, Low: < 12 breaths/min, Normal: 12-16 breaths/min, High: > 16 breaths/min.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

Present for each Basket and overall, and for all vital signs parameters.


BMSOP111/F2


Filename: (Specify file name.rtf)


Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.3 - Summary and Change from Baseline in ECG parameters by Visit
Full Analysis Set

Parameter: XXXXX (XX)

| | Basket l<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| C1D8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |
| Change from Baseline to Cll | D8 | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

- Present for all ECG parameters: heart rate, PR interval, QRS duration, RR interval, QT interval, QTcF with respective unit measure.
- Present for all available visits.


BMSOP111/F2



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.4 - Summary of ECHO at Baseline Full Analysis Set

| | Basket 1 | Basket 2 | Basket 3 | Basket 4 | Basket 5 | Overall |
|---|---|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Significant findings - n (%) | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| LVEF | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min; Max | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX | XX; XX |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.5 - Summary of Physical Examination at Baseline Full Analysis Set

| | Basket 1<br>N=XX | Basket 2 Basket 3<br>N=XX N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX | |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HEENT | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Thorax | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abdomen | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Done | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Present for all Region/Body System parameters: HEENT, thorax, abdomen, skin and mucosae, neurological, extremities, urogenital, general
appearance, heart, back, lymph nodes.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.3-3.6 - Summary of ECOG Performance Status by Visit
Full Analysis Set

| Visit | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| Grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline [a] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| C1D8 [a] | | | | | | |
| 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| i | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 5 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| C1D15 [a] | | | | | | |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <cont.></cont.> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available assessment prior to first dose of study treatment.

- [a] (0) Fully active, able to carry on all pre-disease performance without restriction
  - (1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  - (2) Ambulatory and capable of all self-care but unable to carry out any work activities
  - (3) Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  - (4) Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  - (5) Death

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## PROGRAMMING NOTES:

Present for all available visits.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.5-1.1 - Pharmacokinetic Concentration Data PK Analysis Set

| Jisit<br>Analyte | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| CIDIS | | | | | | |
| BVD-523 (ng/mL) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XXX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Geometric Mean (CV%) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XXX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min; Max | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X | XX.X; XX.X |

GSD=Geometric Standard Deviation, SD=Standard Deviation

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.doc)

### PROGRAMMING NOTES:

Present for all available analytes (BVD-523, BVD-502/503,BVD-506, BVD-513) and visits


BMSOP111/F2



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Table 14.5-1.2 - Pharmacokinetic Parameters Data PK Analysis Set

Analyte: BVD-523

| Visit | Basket 1<br>N=XX | Basket 2<br>N=XX | Basket 3<br>N=XX | Basket 4<br>N=XX | Basket 5<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|---|---|
| ClD15 | | | | | | |
| CMax (ng/mL)<br>n<br>Mean (SD)<br>Geometric Mean (CV%)<br>Median<br>Min; Max | XX<br>XX.XX (XX.XX)<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X | XX<br>XX.XX (XX.XX)<br>XX.XX (XX.XX)<br>XX.XX; XX.X | XX XX.XX (XX.XXX) XX.XX (XX.XXX) | XX<br>XX.XX (XX.XX)<br>XX.XX (XX.XX)<br>XX.XX<br>XX.XX | XX<br>XX.XX (XX.XX)<br>XX.XX (XX.XX)<br>XX.XX<br>XX.XX | XX<br>XX.XX (XX.XX)<br>XX.XX (XX.XX)<br>XX.XX<br>XX.X; XX.X |

GSD=Geometric Standard Deviation, SD=Standard Deviation

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.doc)

## PROGRAMMING NOTES:

Present for all available analytes (BVD-523, BVD-502/503, BVD-506, BVD-513), PK parameters (AUC, Cmax, Cmin, t<sub>1/2</sub>, t<sub>max</sub>), and visits


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Full Analysis Set

Figure 14.2-1.1 - Consort Diagram



Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.2.1 - Spider plot of Percentage Change from Baseline in Sum of Longest Diameter
Full Analysis Set


Filename: (Specify file name.rtf)





Weeks since Treatment Initiation

Best overall response: CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progression Disease, NE=Not Evaluable.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

## PROGRAMMING NOTES:

- · Present all Baskets in separate figures and one figure with all patients.
- Use a different line style for each BOR (dotted line, dashed line, etc).
- Add reference lines for +20% and -30%.

Figure 14.2-1.2.2 - Spider plot of Percentage Change from Baseline in Sum of Longest Diameter Evaluable Analysis Set

## PROGRAMMING NOTES:

- Repeat Figure 14.2-1.2.1
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.3.1 - Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter
Full Analysis Set


Basket = Basket X (N=XX)



Maximum percentage decrease from baseline in total tumor size is the maximum percentage decrease in the sum of longest diameters/short axis for all target lesions observed from baseline for each patient.

Best overall response: CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progression Disease, NE=Not Evaluable.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

## PROGRAMMING NOTES:

- Present each Basket on one figure and one figure with all patients. For overall figure, use a different color for each basket
- Each bar is an individual patient.
- Add reference lines for +20% and -30%.
- · Add the best overall response (CR, PR, SD, PD, NE) of each patient on the top of each bar.

Figure 14.2-1.3.2 - Waterfall plot of Maximum Percentage Change from Baseline in Sum of Longest Diameter
Evaluable Analysis Set

## PROGRAMMING NOTES:

- Repeat Figure 14.2-1.3.1
- Present data on Evaluable Analysis Set.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.4.1 - Swimmer Plot of Response Assessments
Full Analysis Set




Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### PROGRAMMING NOTES:

- Present each Basket on one figure and a figure including all patients.
- · Display patient ID on the left outside the figure except for the figure where all patients are displayed.
- The bar displays time to PD/Death (PFS), with "PD" or "death" displayed at the end of the bar; if no PD/death occurred before cutoff date, the bar stops at cutoff date.
- For responders, display the date of first CR or PR, and display "Ongoing response" arrow if no PD or death occurred before cutoff date.
- "End of Treatment" is the date of treatment discontinuation, this must be displayed only for patients who discontinued the treatment before the
  cut-off date.

Figure 14.2-1.4.2 - Swimmer Plot of Response Assessments Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.4.1
- Present data on Evaluable Analysis Set.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Figure 14.2-1.5.1 - Kaplan-Meier Estimate for Progression-Free survival (PFS)
Full Analysis Set




Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

#### PROGRAMMING NOTES:

- X-axis Label "Progression Free Survival (months)"
- Y-axis Label "Event-free probability (%)."
- · Legend: overall number of events, "Median Duration of Response" and 95% Cl.
- Flag censored observations with '+' and add legend.
- If the median time to event has not been reached, present as "Median (95% CI) NR (xx.x, xx.x)" [replacing xx.x with '-' if there is no upper or lower confidence limit] and add footnote:
  - NR=Median time not reached.
- Present all Baskets on the same figure but with different colors and separate figures for each Basket. In the sample shell where it is 'Cohort' replace with 'Basket'

Figure 14.2-1.5.2 - Kaplan-Meier Estimate for Progression-Free survival (PFS)

Evaluable Analysis Set

### PROGRAMMING NOTES:

- Repeat Figure 14.2-1.5.1
- Present data on Evaluable Analysis Set.

Figure 14.2-1.6.1 - Kaplan-Meier Estimate for Overall Survival (OS)
Full Analysis Set

### PROGRAMMING NOTES:

Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Overall Survival" in X-axis label and legend.

Figure 14.2-1.6.2 - Kaplan-Meier Estimate for Overall Survival (OS)
Evaluable Analysis Set

## PROGRAMMING NOTES:

- Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Overall Survival" in X-axis label and legend.
- Present data on Evaluable Analysis Set.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

Figure 14.2-1.7.1 - Kaplan-Meier Estimate for Duration of Response Full Analysis Set

# PROGRAMMING NOTES:

• Replicate figure 14.2-1.5.1, replacing "Progression Free Survival" by "Duration of Response" in X-axis label and legend.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Listing 16.2.1-1 - Patients informed consent All Patients Set

Basket: Basket 1

| | | | Main Infor | Sample banking for future Biospecimen Main Informed Consent research consent | | | | Optional End of Treatment Biopsy |
|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Age /<br>Gender | Protocol<br>Version | Consent Obtained /<br>Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn | Consent Obtained /<br>Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn | Consent Obtained / Withdrawn? | Date Consent<br>Obtained /<br>Withdrawn |
| XXXXXX | XX/M | 1.0 | Yes / Yes | DDMMYYYYY /<br>DDMMYYYYY | Yes | DDMMMYYYY /<br>DDMMMYYYY | Yes | DDMMYYYYY /<br>DDMMYYYYY |
| XXXXXX | XX/F | 1.0 | Yes / No<br>Yes / No | DDMMYYYYY | Yes<br>Yes | DDMMYYYY | Yes<br>Yes | DDMMYYYYY |
| XXXXXX | XX/F | 1.0 | No / Yes | DDMMMYYYY<br>DDMMMYYYY | No | DDMMMYYYY | No | DDMMMYYYY |
| <cont.></cont.> | | | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.doc)

## PROGRAMMING NOTE:

• For all Listings, repeat for each Basket. For All Patients Set present group Screen Failures




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.1-2 - Failed Inclusion and Exclusion Criteria
All Patients Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Protocol<br>Version | Failed Inclusion /<br>Exclusion No. | Description |
|---|---|---|---|---|
| хх-хх | xx/M | 1.0 | INCL01 | xxxxxxxxxx |
| xxx-xx | xx/M | 1.0 | EXCL01 | xxxxxxxxxx |
| xx-xx | xx/M | 1.0 | EXCL02 | XXXXXXXXXXX |
| xxx-xx | xx/F | 1.0 | INCL02 | xxxxxxxxxx |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

List all failed Inclusion / Exclusion criteria as per eCRF.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.1-3 - Patient Disposition All Patients Set Page 1 of Y

Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Enrolled | Date of<br>Assignment | Gene/ Codon/<br>Amino acid<br>change | Completed<br>Screening /<br>Reason | Date of<br>Screening<br>Completion /<br>Discontinuation | Eligible for inclusion? | Rescreened? /<br>Previous patient<br>number |
|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Yes | DDMMYYYY | BRAF /D594 /<br>Alanine A | Yes | DDMMMYYYY | Yes | No |
| xxx-xx | xx/F | Yes | DDMMYYYY | MEK1/MAP2K1 /<br>K601 /Arginine R | No /<br>Physician<br>Decision | DDMMYYYY | Yes | Yes /xxxxxxx |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Listing 16.2.1-3 - Patient Disposition All Patients Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Completed<br>Treatment /<br>Reason | Date of Treatment<br>Discontinuation | Date of Last Study<br>Dose | Completed Study /<br>If no, reason | Date of Completion |
|---|---|---|---|---|---|---|
| xx-xx | M/xx | Yes | DDMMYYYY | DDMMYYYY | Yes | DDMMYYYY |
| xx-xx | жж/F | No/<br>Progressive<br>Disease | DDMMYYYYY | DDMMYYYY | No/ xxxxxx | DDMMMYYYY |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


### Listing 16.2.2-1 - Analysis Sets All Patients Set

### Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | All Patients Set [a] | Full Analysis Set<br>[b] | Stage 1 Analysis Set<br>[c] | Evaluable Analysis<br>Set [d] | PK Analysis<br>Set [e] |
|---|---|---|---|---|---|---|
| хх-хх | xx/M | Yes | Yes | Yes | Yes | Yes |
| xx-xx | xx/F | Yes | Yes | Yes | Yes | Yes |

### Note: M=Male, F=Female.

- [a] Patients who were enrolled regardless of whether they received the study drug or not.
- [b] Patients who received at least 1 dose of the study drug.
- [c] First 13 patients who have completed at least one cycle of therapy and who have received a minimum of 75% of prescribed study therapy during Cycle 1
- [d] Patients who received at least one dose of study drug and have at least one post-treatment study evaluation or who have discontinued therapy prior to the first post-treatment study evaluation due to clinical progressive disease or drug-related adverse events.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Listing 16.2.3-1 - Protocol Deviations Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Deviation<br>Category | Summary Term | Deviation<br>Description | Classification | Exclusion from<br>Analysis Sets |
|---|---|---|---|---|---|---|
| хх-хх | xx/M | Inclusion<br>Criteria<br> | ******* | XXXXXXXXXXXX | Important | Evaluable Analysis<br>Set |
| ххх-хх | xx/F | Study<br>Assessments<br> | ************ | XXXXXXXXXXX | Non-Important | Full Analysis Set |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Categories / Summary Term / Description to match the PDCF.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-1 - Demographics and Baseline Characteristics


Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Childbearing/<br>Reproductive<br>Potential | Surgery<br>Name | Date of<br>Surgery/Post-<br>Menopausal | Date of Last<br>Menstrual<br>Period | Race | Ethnicity | Height at<br>Screening<br>(cm) | Weight at<br>Screening<br>(kg) |
|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Surgically<br>Sterile | Vasectomy | DDMMYYY | | White | Hispanic or<br>Latino | xx | жж |
| xx-xx | xx/F | Able to Bear<br>Children | | | DDMMYYY | Other, | Not<br>Hispanic or<br>Latino | xx | xx |
| xxx-xx | xx/F | Sterile -<br>Other Reason,<br>xxxxxx | | | DDMMYYY | | | | |

Full Analysis Set

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-2 - Smoking History Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Smoking<br>History? | Substance | Usage |
|---|---|---|---|---|
| xx-xx | xx/M | Yes | Cigarettes | Former |
| xx-xx | xx/F | No | | |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-3 - Disease History Full Analysis Set

Basket: Basket 1

| Patient ID | Age /<br>Gender | Cancer<br>Diagnosis | Date of<br>Initial<br>Diagnosis | Time since<br>Initial<br>Diagnosis [a] | Stage at<br>Diagnosis | Method of<br>Diagnosis | Current<br>Stage at<br>Enrollment | Prior<br>Radiation<br>Therapies? |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Stomach | DDMMMYYYY | xx | 1 | Cytological | 1 | Yes |
| xx-xx | xx/F | Other,<br>xxxxx | DDMMMYYYY | xx | 2 | Histological | 4 | No |



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-4 - Medical History and Concomitant Diseases Full Analysis Set Page 1 of Y

Basket: Basket 1

| Dasket. E | | | | | | | |
|---|---|---|---|---|---|---|---|
| Patient | Age / | | System Organ | | Start Date (Day) | | |
| ID | Gender | Reported Term | Class | Preferred Term | /End Date (Day) | Ongoing | MH or Conc. |
| xxx-xx | xx/M | xxxxxxx | XXXXXXXX | ххххххх | DDMMYYYY (xx) /<br>DDMMYYYYY (xx) | No | МН |
| xxx-xx | xx/F | XXXXXXX | xxxxxxxx | XXXXXXX | DDMMMYYYY (xx) | Yes | Conc. |

Note: M=Male, F=Female.

MedDRA <vx.x>.

Study day is calculated as (Event Date - Study treatment start date) for dates before Study treatment start date and (Event date - First treatment date + 1) for dates after Study treatment start date.

Medical history (MH): any conditions that started before the first study treatment date and were not ongoing at the first study treatment date.

Concomitant disease (Conc.): any conditions that started before first study treatment administration and were ongoing at first study treatment administration.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-5 - Prior Systemic Anti-Cancer Therapies Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Line of<br>Therapy | Name of<br>Therapy | Start Date<br>(Day) | End Date<br>(Day) | Best Overall<br>Response | Date of Best<br>Overall<br>Response | Date of<br>Relapse/<br>Progression | Reason for<br>Discontinuati<br>on |
|---|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | 1 | xxxxxx | DDMMMYYYY<br>(xx) | DDMMYYYYY<br>(xx) | Stable<br>Disease | DDMMYYYY | DDMMMYYYY | Intolerance |
| xx-xx | xx/M | 1 | XXXXX | DDMMYYYYY<br>(xx) | DDMMYYYYY<br>(xx) | Stable<br>Disease | DDMMYYYY | DDMMYYYY | Lack of<br>Efficacy |
| хж-жж | xx/F | 4 | XXXXX | DDMMYYYY<br>(xx) | (xx)<br>DDMMYYYY | Partial<br>Response | DDMMYYYY | DDMMMYYYY | Other,<br>xxxxx |

Note: M=Male, F=Female.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM)

# PROGRAMMING NOTES:

Data taken from 'Prior Cancer Medications' page.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-6 - Prior Radiotherapy Courses Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Site of Radiotherapy | Dose (Unit) | Start Date (Day) | End Date (Day) | Duration (months) [a] |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | Abdominal Cavity | xxx (xxx) | DDMMMYYYY (xx) | DDMMYYYYY (xx) | xx |
| xxx-xx | xx/M | Adrenal Gland | xxx (xxx) | DDMMYYYY (xx) | DDMMYYYY (xx) | xx |
| xxx-xx | xx/F | Bile Duct | xxx (xxx) | DDMMMYYYY (xx) | DDMMYYYY (xx) | жж |

Note: M=Male, F=Female.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication date - First treatment date + 1) for dates after Study treatment start date.

[a] Duration of radiotherapy calculated as [(end date - start date) + 1] / 30.4375.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

# PROGRAMMING NOTES:

· Data taken from 'Prior Radiotherapy' page.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-7 - Prior and Concomitant Medications Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Reported Term /<br>Preferred Term /<br>ATC Class | Indication | Start Date<br>(Day) | End<br>Date (Day) | Dose<br>(Units) /<br>Frequency | Route | Medication to<br>treat<br>adverse event? /<br>Adverse Event (ID) | Ongoing | Prior<br>/<br>Conc. |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Xxxxxxxxxxx /<br>xxxxxxxxxx /<br>xxxxxx | xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | иии (ии)<br>/ Daily | Oral | Yes / xxxx (x) | Yes | Conc. |
| жж-жж | xx/F | ************************************** | XXXXXX | DDMMMYYYY<br>(xx) | Ongoing | xxx (xx)<br>/ Twice<br>per day | Oral,<br>xxxx | No | No | Prior |

Note: M=Male, F=Female, ATC=Anatomical Therapeutic Chemical.

WHOHD-B3 <vx.x>.

Study day is calculated as (Medication Date - Study treatment start date) for dates before Study treatment start date and (Medication date - First treatment date + 1) for dates after Study treatment start date.

Prior medication (Prior): any medications whose end date is before the first study treatment date.

Concomitant medication (Conc.): any medication whose start or end date is either the same or after the first dose of study treatment and up to the end of the on-treatment period.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

- Data taken from 'Prior and Concomitant Medications' page.
- Adverse Event ID taken from collected ID.


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY


Listing 16.2.4-8 - On Treatment Radiation Full Analysis Set

Cohort: Basket 1

| Patient<br>ID | Age /<br>Gender | Received<br>Radiation? | Site of<br>Radiotherapy | Dose (Unit) | Start Date (Day) | End Date (Day) |
|---|---|---|---|---|---|---|
| ххх-ххх | xx/M | Yes | Abdominal Cavity | xxx (xxx) | DDMMYYYYY (xx) | DDMMMYYYY (xx) |
| хх-хх | xx/M | Yes | Adrenal Gland | xxx (xxx) | DDMMYYYYY (xx) | DDMMYYYY (xx) |
| XX-XX | xx/F | No | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Data taken from 'On Treatment Radiation' page.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYYY

Listing 16.2.4-9 - On Treatment Surgery and Medical Procedures Full Analysis Set

Cohort: Basket 1

| Patient<br>ID | Age /<br>Gender | Any Surgeries/<br>Procedures | Name of Surgery/<br>Procedure | Indication? | Start Date (Day) | End Date (Day) | Ongoing? |
|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Yes | xxxxxxxxx | xxxxxxxxx | DDMMMYYYY (xx) | DDMMYYYYY (xx) | No |
| xx-xx | xx/M | Yes | xxxxxxxxx | xxxxxxxxx | DDMMMYYYY (xx) | DDMMYYYYY (xx) | Yes |
| xx-xx | xx/F | No | | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

# PROGRAMMING NOTES:

· Data taken from 'On Treatment Surgery and Medical Procedures' page.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.4-10 - On Treatment Blood Transfusions Full Analysis Set Page 1 of Y

Filename: (Specify file name.rtf)

Cohort: Basket 1

| Patient ID | Age/<br>Gender | Any blood<br>transfusions | Transfusion ID | Date of Transfusion | Category of Transfusion | Units |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | Yes | xxxxxxxxx | DDMMYYYY (xx) | Platelet transfusion | жx |
| | xx/M | Yes | xxxxxxxxx | DDMMMYYYY (xx) | Plasma | xx |
| xx-xx | xx/F | No | | | | |

Note: M=Male, F=Female.

Study day is calculated as Procedure date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

# PROGRAMMING NOTES:

· Data taken from 'On Treatment Blood Transfusions' page.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.4-11 - NGS Data Full Analysis Set

Cohort: Basket 1

| Patient ID | Age/<br>Gender | Gene / Codon /<br>Amino acid change | Vendor | Date of Report | Report Redacted | Report Uploaded |
|---|---|---|---|---|---|---|
| xxx-xx | жж/М | BRAF /D594 /<br>Alanine A | STRATA | DDMMYYYYY (xx) | Yes | Yes |
| xxx-xx | xx/F | MEK1/MAP2K1 /<br>K601 /Arginine R | GUARDANT | | No | No |

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-1 - Ulixertinib In-clinic Administration Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Treatment<br>Administered? | Dose (mg) | Dose Date and Time (day) |
|---|---|---|---|---|
| xx-xx | xx/M | Yes | xxx | DDMMMYYYY hh:mm (xx) |
| xx-xx | xx/F | Yes | xxx | DDMMMYYYY hh:mm (xx) |
| xx-xx | xx/F | Yes | Xxx | DDMMMYYYY hh:mm (xx) |

Note: M=Male, F=Female.

Study day is calculated as Administration date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-2 - Hydroxychloroquine In-clinic Administration Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-1




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-3 - Ulixertinib Interruptions and Adjustments Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Type of Change | Start Date / End Date /<br>Duration (days) | If Adjustment, new dose amount (mg) | Reason for<br>Interruption/Adjustment |
|---|---|---|---|---|---|
| xx-xx | xx/M | Interruption | DDMMYYYY / DDMMYYYYY / (xx) | xxx | Adverse Event |
| xx-xx | xx/F | Adjustment | DDMMYYYY / DDMMYYYYY / (xx) | xxx | Other, |
| xx-xx | xx/F | | | | |

Note: M=Male, F=Female.

Study day is calculated as Interruption/Change date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2


Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-4 - Hydroxychloroquine Interruptions and Adjustments Full Analysis Set

#### PROGRAMMING NOTES:

Repeat Listing 16.2.5-3




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.5-5 - Ulixertinib Exposure Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Number of<br>cycles<br>received [a] | Duration of<br>exposure<br>(months) [b] | Planned cumulative<br>dose (mg) | Actual cumulative dose received (mg)[c] | Relative dose intensity [d] |
|---|---|---|---|---|---|---|
| xxx-xx | xx/M | xx | xxx | xxx (mg) | xxx (mg) | xxx |
| xx-xx | xx/F | xx | xxx | xxx (mg) | ххх (mg) | xxx |

#### Note: M=Male, F=Female.

- [a] Number of cycles received = Number of cycles where the patient received at least one dose.
- [b] Duration of exposure (months) = (Date of last known treatment dosing with ulixertinib- date of initial dosing with ulixertinib) + 1 / 30.4375.
- [c] Actual cumulative dose received (mg) = Sum of [(number of capsules dispensed number of capsules returned) x 150].
- [d] Relative dose intensity = 100 x Actual dose intensity / Planned dose intensity. Actual dose intensity (mg/day) is defined as Actual cumulative dose received (mg) / Duration of exposure (days). Planned dose intensity (mg/day) is defined as Planned cumulative dose (mg) / Duration of exposure (days). Planned cumulative dose is the number of cycles received x number of doses per day x mg prescribed per dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-6 - Hydroxychloroquine Exposure Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-5




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-7 - Ulixertinib Dispensed Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Mg<br>prescribed<br>per dose | Date<br>Bottles<br>Dispensed<br>(day) | Number of<br>Bottles<br>Dispensed | Lot Number<br>of the<br>bottles<br>dispensed | Different Lot<br>number<br>dispensed to<br>the patient? | Lot number<br>dispensed to<br>patient /No of<br>bottles | Total<br>Number of<br>Capsules<br>Dispensed |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | xxx | DDMMYYYYY<br>(xx) | xx | xxxx | Yes | Xxxx/XX | xx |
| xx-xx | xx/F | xxx | DDMMMYYYY<br>(xx) | xx | xxxx | No | | xx |

Note: M=Male, F=Female.

Study day is calculated as Dispensed date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.5-8 - Hydroxychloroquine Dispensed Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-7




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.5-9 - Ulixertinib Returned Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Cycle | Reason<br>capsules<br>not<br>returned | Date<br>Returned<br>(day) | Patient<br>compliant<br>since last<br>visit? If<br>no, reason | Missed dose<br>related to an<br>adverse event? | Number of<br>Bottles Returned | Lot Number<br>of the<br>bottles<br>returned | Total<br>Number of<br>Capsules<br>Returned |
|---|---|---|---|---|---|---|---|---|---|
| xx-xx | mx/M | 2 | Lost | DDMMYYYYY<br>(xx) | Yes | Yes | xx | xxxx | xxx |
| xx-xx | xx/F | 3 | Other, xxxxx | DDMMYYYY<br>(xx) | No, xxxxx | Yes | xx | xxxx | xxx |

Note: M=Male, F=Female.

Study day is calculated as Returned date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.5-10 - Hydroxychloroquine Returned Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.5-9




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-1 - Target Lesions Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Visit | Target<br>Lesions at<br>Screening? | Lesion<br>Number | Tumor<br>Type | Organ<br>Site | Method | Date of<br>Scan<br>(Day) | Longest<br>Diameter/<br>Short-<br>axis(mm) | Sum of Longest Diameter (mm)<br>/ Change from baseline / %<br>Change from baseline |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening<br>C2D1 | Yes | T01 | Primary | Bladder | CT<br>Scan | DDMMMYYYY<br>(xx) | xxx | XXX |
| | | ••• | | | | | | | | |
| xx-xx | xx/F | Screening | Yes | T02 | Metastasis | Other, | MRI | DDMMYYYY<br>(xx) | xxx | xxx / xxx / xxx |
| | | ••• | | | | | | | | |

Note: M=Male, F=Female.

Study day is calculated as (Scan Date - Study treatment start date) for dates before Study treatment start date and (Scan date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit.


BMSOP111/F2


Filename: (Specify file name.rtf)



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

Listing 16.2.6-2 - Non-Target Lesions Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Visit | Assessment<br>Performed /<br>Reason | Non-Target<br>Lesions at<br>screening | Lesion Number | Organ<br>Site | Method | Date of Scan | Result |
|---|---|---|---|---|---|---|---|---|---|
| xxx-xx | жж/М | Screening | Yes | Yes | NT01 | Bladder | CT Scan | DDMMYYYYY<br>(xx) | Present |
| | | C2D1<br> | No, xxx | | | | | | |
| xx-xx | xx/F | Screening | Yes | Yes | NT02 | Other, | MRI | DDMMYYYYY<br>(xx) | Absent<br>(Disappeared) |

## Note: M=Male, F=Female.

Study day is calculated as (Scan Date - Study treatment start date) for dates before Study treatment start date and (Scan date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-3 - New Lesions Full Analysis Set

Basket: Basket 1

| Patient | Age/ | | Any New | | | | |
|---|---|---|---|---|---|---|---|
| ID | Gender | Visit | Lesions | Lesion Number | Method | Date of Scan (Day) | Organ Site |
| xx-xx | xx/M | C2D29 | Yes | NL01 | CT Scan | DDMMYYYY (xx) | Abdomen |
| хх-хх | xx/F | C2D29 | Yes | NL02 | Other, | DDMMYYYY (xx) | Bone |

Note: M=Male, F=Female.

Study day is calculated as Scan date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


#### Listing 16.2.6-4 - Overall Response Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Best Overall<br>Response [a] | Assessment<br>Performed/<br>Reason | Date of Assessment<br>(Day) | Target<br>Lesion<br>Response | Non-Target<br>Lesion<br>Response | New Lesions | Overall<br>Response |
|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | CR | Yes | DDMMYYYY (xx) | CR | CR | Yes | PD |
| xx-xx | xx/F | PD | Yes | DDMMMYYYY (xx) | NE | PD | No | NE,<br>xxxx |

Note: M=Male, F=Female, CR=Complete Response, Non CR/Non PD=Non Complete Response/Non Progressive Disease, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

Study day is calculated as Assessment date - First treatment date + 1.

[a] Confirmed best overall response.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-5 - Progression-Free Survival (PFS) Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Treatment<br>Start Date | Date of<br>Last Tumor<br>Assessment | Date of Event/<br>Censoring | Event / Censoring<br>Reason | PFS (months) |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | DDMMYYYY | DDMMMYYYY | DDMMMYYYY | Death | xx.x |
| xx-xx | xx/F | DDMMYYYY | DDMMMYYYY | DDMMYYYY | Censored: xxxxx | xx.x |

Note: M=Male, F=Female, PFS=Progression-Free Survival.

Event: progressive disease (PD) or death from any cause.

The PFS (in months) is defined as the time from the first ulixertinib dose until the first radiographically documented progression of disease or death from any cause, whichever occurs first.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-6 - Survival Status Full Analysis Set Page 1 of Y

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Completed<br>End of<br>Study? | Any Anti-Cancer<br>Treatment Since End<br>of treatment or<br>Last FUP/ Start<br>Date | Any Tumor Assessment Since<br>End of Study or Last FUP/<br>Assessment Date/<br>Overall Response | Survival<br>Status at<br>Follow-Up | Date of<br>Death | Last Known Date<br>Patient Alive [a] |
|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | Yes | Yes/ DDMMYYYY | Yes/ DDMMMYYYY/ Complete<br>Response | Alive | | |
| xx-xx | xx/F | Yes | No | No | Dead | DDMMYYYY | |

Note: M=Male, F=Female, FUP=Follow-up, CR=Complete Response, Non CR/Non PD=Non Complete Response/Non Progressive Disease, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

[a] If Survival status at the time of follow-up is unknown.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.6-7 - Duration of Response (DOR) Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Best Overall<br>Response [a] | Treatment<br>Start Date | Date of First<br>Response | Date of<br>Last Tumor<br>Assessment | Date of Event /<br>Censoring | Event /<br>Censoring Reason | Duration of<br>Response<br>(months) |
|---|---|---|---|---|---|---|---|---|
| xxx-xx | xx/M | CR | DDMMYYYYY | DDMMYYYY | DDMMMYYYY | DDMMMYYYY | Death | xx.x |
| ххх-хх | xx/F | PR | DDMMYYYYY | DDMMYYYYY | DDMMMYYYY | DDMMMYYYY | Censored: xxxxx | xx.x |

Note: M=Male, F=Female, CR=Complete Response, PR=Partial Response, SD=Stable Disease, PD=Progressive Disease, NE=Not Evaluable.

Event: progressive disease (PD) or death from any cause.

This listing includes only patients with response (CR or PR).

Duration of response is the period from the date of initial confirmed PR or CR until the date of first radiographically documented progressive disease or death from any cause.

[a] Confirmed best overall response.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)


BMSOP111/F2



Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.7-1 - Adverse Events All Patients Set

Basket: Basket 1

| Patient | Age / | | | System Organ | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| ID | Gender | ID | Reported Term | Class | Preferred Term | Start Date (day) | End Date (day) | TEAE? | SAE? |
| xx-xx | xx/M | xx | XXXXXXXX | XXXXXXXX | xxxxxxxx | DDMMYYYY (xx) | DDMMYYYY (xx) | Yes | Yes |
| xx-xx | xx/F | xx | xxxxxxxx | xxxxxxxx | xxxxxxxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | No | No |

Note: M=Male, F=Female, TEAE=Treatment Emergent Adverse Event, SAE=Serious Adverse Event.


ID as collected in the databased. MedDRA <vx.x>. NCI CTCAE v5.0.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

Template Author: Andra Rusu Version 5.0 25Jun2020 BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.7-2 - Treatment-Emergent Adverse Events Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | ID | Reported Term<br>/ System Organ<br>Class<br>/Preferred<br>Term | Start Date<br>(Day) / End<br>Date (Day) /<br>Duration<br>(days) | SAE /<br>Serious<br>ness | NCI-<br>CTCAE<br>Grade | Relation<br>Ship to<br>Disease | Relation Ship to Ulixertin ib / Hydroxych loroquine | Action<br>Taken with<br>Ulixertinib<br>/<br>Hydroxychlo<br>roquine | Medication<br>or<br>Therapies?<br>/<br>Medication<br>Name | Outcome<br>[a] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | xx | XXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | DDMMMYYYY<br>(xx) /<br>DDMMMYYYY<br>(xx) / xx | Yes /<br>Hospital<br>ization | 1 | Related | Related<br>/Related | Drug<br>Interrupted<br>/Drug<br>Interrupted | Yes<br>/xxxxxxxx,<br>xxxxxxx | Res'd |
| xx-xx | xx/F | xx | <br>************/<br>********************* | DDMMMYYYY (xx) / xx DDMMMYYYYY | No | 3 | Possibly<br>Related | Possibly<br>Related<br>/Related | Drug<br>Interrupted<br>/Drug<br>Interrupted | Yes<br>/xxxxxxxx | Res'd<br>seq,<br>xxxxxx |

Note: M=Male, F=Female, TEAE=Treatment Emergent Adverse Event, SAE=Serious Adverse Event.

MedDRA <vx.x>. NCI CTCAE v5.0.

ID as collected in the databased.

Study day is calculated as TEAE date - First treatment date + 1.

[a] Res'd=Resolved, Res'd seg=Recovered/Resolved with sequelae, Ong=Ongoing, Unk=Unknown, Fatal=Fatal.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

- · Sort by Basket, patient ID, ascending Adverse Event Start Date and Reported Term.
- Outcome = "Res'd seq" please specify sequelae.


BMSOP111/F2



Protocol: BVD-523-HCQ

**Statistical Analysis Plan:** 

2.0 / 02-Sep-2024

Listing 16.2.7-3 - Serious Adverse Events Full Analysis Set

# PROGRAMMING NOTES:

Repeat Listing 16.2.7-2 and include only AEs classified as Serious.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.7-4 - Deaths All Patients Set Page 1 of Y

Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Date of Death (Day) | Autopsy Performed? /<br>Date of Autopsy | Primary Cause of Death | Treatment-Emergent Death |
|---|---|---|---|---|---|
| жж-жж | xx/M | DDMMMYYYY (xx) | No | Progressive Disease | Yes |
| xx-xx | xx/F | DDMMMYYYY (xx) | Yes /DDMMYYYY | Adverse Event, xxxxxxx | No |

Note: M=Male, F=Female.

[a] A death is considered Treatment-Emergent if occurred after Ulixertinib administration.

Study day is calculated as Death date - First treatment date + 1.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

# PROGRAMMING NOTES:

· Specify primary cause of death if not PD.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.8-1 - Hematology Full Analysis Set Page 1 of Y

Filename: (Specify file name.rtf)

Basket: Basket 1

| Patient<br>ID | Age/<br>Gender | Study<br>Visit | Sample Date and Time<br>(Day) | Parameter (Unit) | Result /<br>Reference Range<br>Indicator / CS?<br>[a] | LLN - ULN | CTC<br>Grade | Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| жж-жж | xx/M | Screening | DDMMYYYY / hh:mm (xx) | RBC (xxx) | жж / L / CS | хх - хх | xx | |
| | | C1D1 | DDMMYYYY / hh:mm (xx) | RBC (xxx) | жж / L / CS | xx - xx | xx | xx |
| xx-xx | xx/F | Screening | DDMMMYYYY / hh:mm (xx) | RBC (xxx) | Not Done | | | |
| | | C1D1<br> | | *** | | | | |

Note: M=Male, F=Female, L=Low, H=High, ULN=Upper Limit of Normal, LLN=Lower Limit of Normal, CS=Clinically Significant, NCS=Non Clinically Significant.

CTCAE v5.0.

Baseline is the last available assessment prior to first dose of study treatment.

Study day is calculated as (Sample Date - Study treatment start date) for dates before Study treatment start date and (Sample date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- Sort by Basket, patient ID, ascending Sample Date and Time and Parameter.
- Include all hematology parameters.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

Listing 16.2.8-2 - Biochemistry Full Analysis Set

#### PROGRAMMING NOTES:

· Repeat Listing 16.2-8.1 for all biochemistry parameters.

Listing 16.2.8-3 - Coagulation Full Analysis Set

## PROGRAMMING NOTES:

· Repeat Listing 16.2-8.1 for all coagulation parameters.

Listing 16.2.8-4 - Urinalysis Full Analysis Set

## PROGRAMMING NOTES:

Repeat Listing 16.2-8.1 for all urinalysis parameters.

Listing 16.2.8-5 - Tumor Markers Full Analysis Set

## PROGRAMMING NOTES:

· Repeat Listing 16.2-8.1 for all tumor marker parameters.



Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.8-6 - Pregnancy Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Sample<br>Type | Assessment<br>Performed? /Reason | Sample Date (Day) | Result |
|---|---|---|---|---|---|---|
| xx-xx | xx/F | Screening<br>Baseline | Serum | Yes | DDMMYYYY (xx) | Positive |
| | xx/F | | | | | |

Note: F=Female.

Baseline is the last available assessment prior to first dose of study treatment.

Study day is calculated as (Sample Date - Study treatment start date) for dates before Study treatment start date and (Sample date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, visit.


BMSOP111/F2



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-1 - Vital Signs Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment Date<br>and Time (Day) | Parameter<br>(Unit) | Result/ Reference Range<br>Indicator / CS? [a] | Position | Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMMYYYY hh:mm (xx) | Systolic Blood<br>Pressure (xxx) | жж / H / CS | Sitting | |
| | | Baseline<br> | Yes | DDMMYYYYY hh:mm (xx) | Systolic Blood Pressure (xxx) | жж / Н / CS | Supine | |
| xxx-xx | xx/F | Screening<br> | No / xxxxxx | | | Not Done | | |

Note: M=Male, F=Female, L=Low, H=High, VH=Very High, ND=Not Done, CS=Clinically Significant, NCS=Non Clinically Significant.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, ascending Assessment Date and Time and Parameter.


<sup>[</sup>a] If status = "Not Done" populate with "Not Done".

<sup>\*</sup> Baseline is the last available assessment prior to first dose of study treatment.

For temperature, Low if < 36.4°C; high if > 37.7°C.

For pulse, Low if < 55bpm; high if 101-150bpm; very high if > 150bpm.

For systolic blood pressure, Low if < 90mmHg; high if 131-160mmHg; very high if >= 161mmHg.

For diastolic blood pressure, Low if < 60mmHg; high if 86-100mmHg; very high if >= 101mmHg.

For Pulse oximetry, Very Low: < 90 %, Low: 90-95 %, Normal: ≥ 95 %.

For Respiratory Rate, Low: < 12 breaths/min, Normal: 12-16 breaths/min, High: > 16 breaths/min.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.



Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Filename: (Specify file name.rtf)

#### Listing 16.2.9-2 - Electrocardiogram Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment Date and Time (Day) | Method/<br>Position | Parameter<br>(Unit) | Result /CS? | Change from baseline |
|---|---|---|---|---|---|---|---|---|
| xx-xx | жж/М | Screening | Yes | DDMMYYYYY hh:mm<br>(xx) | 12 Lead<br>Standard/<br>Supine | Heart Rate<br>(xxx) | xx /No | |
| xx-xx | xx/F | Screening | Yes | DDMMYYYY hh:mm | 12 Lead<br>Standard/<br>Supine | Heart Rate<br>(xxx) | xx /Yes | |

Note: M=Male, F=Female, L=Low, H=High.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

## PROGRAMMING NOTES:

Sort by Basket, patient ID, ascending Assessment Date and Time and Parameter.




Protocol: BVD-523-HCQ

Statistical Analysis Plan: 2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-3 - ECHO Full Analysis Set

Basket: Basket 1

| Patient | Age / | Assessment<br>Performed? / | | | | |
|---|---|---|---|---|---|---|
| ID | Gender | Reason | Method | Assessment Date (Day) | Parameter (Unit) | Result /CS? |
| VVV-VV | xx/M | Yes | Echocardiography | DDMMYYYY (xx) | LVEF (xx) | xx /No |
| XXX-XX | XX/II | ies | Echocardrography | DDMMIIII (XX) | TAFE (XX) | XX /NO |

Note: M=Male, F=Female, LVEF=Left Ventricular Ejection Fraction.

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Sort by Basket, patient ID, ascending Assessment Date and Time.




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMYYYY

Listing 16.2.9-4 - Physical Examination


Full Analysis Set
Basket: Basket 1

| | | | Assessment | | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Performed? /<br>Reason | Assessment<br>Date | Region /Body<br>System | Result /CS? [a] | Abnormal<br>Findings |
| xx-xx | xx/M | Screening | Yes | DDMMYYYY | HEENT | Abnormal/ CS | xxxxxxx |
| xx-xx | xx/F | Screening | Yes | DDMMYYYYY | Thorax | Not Done | |

Note: M=Male, F=Female, CS=Clinically Significant, NCS=Non Clinically Significant.

[a] If status = "Not Done" populate with "Not Done".

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

## PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, Region/body system.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY


Listing 16.2.9-5 - Ophthalmology Exam Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Assessment<br>Date | Examination Test | Any Abnormal<br>Clinically<br>Significant<br>Result? | Eyes<br>Affecte<br>d | Abnormal Finding |
|---|---|---|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY | Best-corrected visual acuity | Yes | Left | XXXXXXXXXX |
| xx-xx | xx/F | Screening | Yes | DDMMYYYY | *** | Yes | Both | |

Note: M=Male, F=Female, CS=Clinically Significant, NCS=Non Clinically Significant.

Program: (Program name.sas) (run on: DDMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, examination test name




Protocol: BVD-523-HCQ Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.9-6 - ECOG Performance Status Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Assessment<br>Performed? /<br>Reason | Date of Assessment (Day) | ECOG Performance Status [a] |
|---|---|---|---|---|---|
| xx-xx | xx/M | Screening | Yes | DDMMYYYY (xx) | (0) Fully Active |
| | | Baseline<br> | Yes | DDMMMYYYY (xx) | (0) Fully Active |
| xxx-xx | xx/F | Screening | Yes | DDMMYYYYY (xx) | (1) Restricted |
| | | Baseline<br> | No, xxxx | | |

Note: M=Male, F=Female.

Baseline is the last available assessment prior to first dose of study treatment.

- [a] (0) Fully active, able to carry on all pre-disease performance without restriction
  - (1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  - (2) Ambulatory and capable of all self-care but unable to carry out any work activities
  - (3) Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  - (4) Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  - (5) Death

Study day is calculated as (Assessment Date - Study treatment start date) for dates before Study treatment start date and (Assessment date - First treatment date + 1) for dates after Study treatment start date.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


#### PROGRAMMING NOTES:

Sort by Basket, patient ID, visit, assessment date.




Protocol: BVD-523-HCQ
Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.11-1 - Pharmacokinetic Concentration Data Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Collection Date/Time (Day) / Timepoint | Analyte | Concentration (Unit) |
|---|---|---|---|---|---|
| | | | | | xxxx (ng/mL) |
| xx-xx | xx/M | C1D15 | ddmmmyyyy hh:mm (xx) / Pre-dose | BVD-523 | |

---

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM)

Filename: (Specify file name.rtf)


## PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit, assessment date and time.




Protocol: BVD-523-HCQ

Statistical Analysis Plan:

2.0 / 02-Sep-2024

BioMed Valley Discoveries

Protocol: BVD-523-HCQ ('Delivery' / 'Type')

Data extraction date: DDMMMYYYY

Listing 16.2.11-2 - Pharmacokinetic Parameters Data Full Analysis Set

Basket: Basket 1

| Patient<br>ID | Age /<br>Gender | Study<br>Visit | Visit | Analyte | PK Parameter | Result |
|---|---|---|---|---|---|---|
| xx-xx | xx/M | C1D15 | C1D15 | BVD-523 | AUC | xxxx |

---

Note: M=Male, F=Female.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)


## PROGRAMMING NOTES:

· Sort by Basket, patient ID, visit and analyte.


## Certificate Of Completion

Envelope Id: 9D451F5DDB6A406CBCF295C356DEEC6D

Subject: Complete with Docusign: BVD-523-HCQ\_SAP\_v2.0\_02Sep2024.pdf

Source Envelope:

Document Pages: 185 Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Status: Completed

Envelope Originator:

Julien Lucas julien.lucas@aixial.com

IP Address: 77.66.37.185

# Record Tracking

Status: Original

02-Sep-2024 | 16:21

Holder: Julien Lucas

julien.lucas@aixial.com

Location: DocuSign

# Signer Events

Anna Groover

agroover@biomed-valley.com

Senior Scientist

Security Level: Email, Account Authentication

(Required)

# Signature

Signatures: 6

Initials: 0

Signed by: anne Breeze

D Signer Name: Anna Groover Signing Reason: I approve this document Signing Time: 03-Sep-2024 | 08:40 CDT

Signature Adoption: Pre-selected Style

71380BDD08BC4D289E63FA3831CD4243

Signature ID:

71380BDD-08BC-4D28-9E63-FA3831CD4243

Using IP Address: 136.37.127.159

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 03-Sep-2024 | 14:39

ID: 94d5e37d-2fb2-42f9-ab4e-2e7b997de2ae

Brent Kreider

bkreider@biomed-vallev.com

President

Security Level: Email, Account Authentication

(Required)

Signed by:

Brent Kreider Signer Name: Brent Kreider

Signing Reason: I approve this document Signing Time: 04-Sep-2024 | 08:58 PDT 9FC8BD6421864A9788CCD264914F8A6C

Signature Adoption: Pre-selected Style

Signature ID:

9FC8BD64-2186-4A97-88CC-D264914F8A6C

Using IP Address: 173.197.22.10

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

I approve this document

Electronic Record and Signature Disclosure: Accepted: 04-Sep-2024 | 16:58

ID: e1a5bfa5-34ac-47ef-af7d-11b59f1cd6cc

# Timestamp

Sent: 02-Sep-2024 | 16:33 Viewed: 03-Sep-2024 | 14:39 Signed: 03-Sep-2024 | 14:40

Sent: 02-Sep-2024 | 16:33

Viewed: 04-Sep-2024 | 16:58

Signed: 04-Sep-2024 | 16:58